# Statistical Analysis Plan



| Sponsor | Arcutis Biotherapeutics, Inc. |
|---|---|
| Protocol Title: | A Phase 2a, 8-Week, Parallel Group, Double Blind, Vehicle-Controlled Study of the Safety and Efficacy of ARQ-154 Foam 0.3% Administered QD in Subjects with Seborrheic Dermatitis |
| Protocol Number: | ARQ-154-203 |
| Premier Research PCN: | ARCU210100 |
| Document Version: | Final 1.0 |
| Document Date: | 08-Sep-2020 |

# Approvals

| Role | Signatures | Date (dd-Mmm-yyyy) | |
|---|---|---|---|
| | Print Name: | 08-Sep-2020 18:05:40 | EDT |
| | Sign Name: | | |
| Biostatistician | | | |
| | Print Name: | 08-Sep-2020 18:27:44 | EDT |
| | Sign Name: | | |
| Premier Senior<br>Reviewer | | | |
| | Print Name: | 09-Sep-2020 09:41:48 | PDT |
| Arcutis Biotherapeutics, Inc. Representative | Sign Name: | | |





# **Document History**

Not applicable.





## **Table of Contents**

| Ap | provals | | 1 |
|-----|-----------|--------------------------------------------------|------|
| Do | cument | History | 2 |
| Ta | ble of C | Contents | 3 |
| Lis | st of Tal | oles | 5 |
| Lis | st of Fig | ures | 5 |
| 1. | Ov | rerview | 6 |
| 2. | Stu | ndy Objectives and Endpoints | 6 |
| | 2.1. | Study Objectives | 6 |
| | 2.1.1. | Primary Objective | 6 |
| | 2.2. | Study Endpoints | 6 |
| | 2.2.1. | Safety Endpoints | 6 |
| | 2.2.2. | Efficacy Endpoints | 7 |
| 3. | Ov | rerall Study Design and Plan | 8 |
| | 3.1. | Overall Design | 8 |
| | 3.2. | Sample Size and Power. | 8 |
| | 3.3. | Study Population | 8 |
| | 3.4. | Treatments Administered | |
| | 3.5. | Method of Assigning Subjects to Treatment Groups | 9 |
| | 3.6. | Blinding and Unblinding. | 9 |
| | 3.7. | Schedule of Events | 9 |
| 4. | Sta | tistical Analysis and Reporting | . 12 |
| | 4.1. | Introduction | . 12 |
| | 4.2. | Interim Analysis and Data Monitoring | . 12 |
| 5. | | alysis Populations | |
| 6. | Ge | neral Issues for Statistical Analysis | |
| | 6.1. | Statistical Definitions and Algorithms | . 13 |
| | 6.1.1. | Baseline | . 13 |
| | 6.1.2. | Adjustments for Covariates | . 13 |
| | | Multiple Comparisons | |
| | 6.1.4. | Handling of Dropouts or Missing Data | . 14 |
| | | Analysis Visit Windows | |
| | 6.1.6. | Pooling of Sites | . 16 |
| | | Derived Variables | |
| | 6.1.8. | Data Adjustments/Handling/Conventions | |
| | 6.2. | Special Handling for COVID-19 Disruptions | |
| 7. | Stu | ndy Patients/Subjects and Demographics | 20 |





| | 7.1. | Disposition of Subjects and Withdrawals | 20 |
|-----|--------|-------------------------------------------------------|----|
| | 7.2. | Protocol Deviations | 20 |
| | 7.3. | Demographics and Other Baseline Characteristics | 20 |
| | 7.4. | Exposure and Compliance | 21 |
| 8. | Ef | ficacy Analysis | 21 |
| | 8.1. | Primary Efficacy Analysis | 21 |
| | 8.2. | Secondary Efficacy Analysis | 23 |
| | 8.2.1. | IGA | 23 |
| | 8.2.2. | Overall Assessment of Erythema | 23 |
| | 8.2.3. | Overall Assessment of Scaling | 24 |
| | | WI-NRS | |
| | 8.3. | Exploratory Efficacy Analysis | 25 |
| 9. | Sa | fety and Tolerability Analysis | |
| | 9.1. | Adverse Event | |
| | 9.1.1. | Adverse Events Leading to Withdrawal | 26 |
| | | Deaths and Serious Adverse Events | |
| | 9.2. | Local Tolerability Assessments | 27 |
| | 9.3. | Clinical Laboratory Evaluations | |
| | 9.4. | Vital Signs | |
| | 9.5. | PHQ-8 | |
| | 9.6. | C-SSRS | 28 |
| | 9.7. | Physical Examination | 28 |
| | 9.8. | Concomitant Medication | |
| 10. | Ch | nanges from Planned Analysis | 29 |
| 11. | Ot | her Planned Analysis | 30 |
| | 11.1. | Pharmacokinetic Analysis | 30 |
| 12. | Re | eferences | 30 |
| 13. | | bles, Listings, and Figures | |
| | 13.1. | Planned Table Descriptions | |
| | 13.1.1 | . Demographic Data | 31 |
| | | . Efficacy Data | |
| | | . Safety Data | |
| | 13.2. | | |
| 14. | | bles, Listings, and Listing Shells | |
| | 14.1. | Standard Layout for all Tables, Listings, and Figures | |
| | 14.2. | Planned Table Shells | |
| | 14.3. | Planned Listing Shells | |





| Appendix 1: Premier Research Library of Abbreviations | 149 |
|-------------------------------------------------------|-----|
| List of Tables | |
| Table 1: Schedule of Events | 10 |
| Table 2: Analysis Visit Windows | |
| Table 3: IGA | 21 |
| Table 4: Erythema Grades | 23 |
| Table 5: Scaling Grades | 24 |
| Table 6: Demographic Data Summary Tables | 31 |
| Table 7: Efficacy Data Summary Tables | 31 |
| Table 8: Safety Data Summary Tables | 35 |
| Table 9: Planned Listings | 38 |
| List of Figures | |
| Figure 1: Standardized Layout | 41 |
| Figure 2: Planned Table Shells | 43 |





#### Overview 1.

This statistical analysis plan (SAP) describes the planned analysis and reporting for Arcutis Biotherapeutics, Inc. protocol number ARQ-154-203 (A Phase 2a, 8-Week, Parallel Group, Double Blind, Vehicle-Controlled Study of the Safety and Efficacy of ARQ-154 Foam 0.3% Administered QD in Subjects with Seborrheic Dermatitis), dated 07-Jan-2020 Amendment Version 1.0. Reference materials for this statistical plan include the protocol and the accompanying sample data collection documents. Operational aspects related to collection and timing of planned clinical assessments are not repeated in this SAP unless relevant to the planned analysis.

The structure and content of this SAP provides sufficient detail to meet the requirements identified by the Food and Drug Administration (FDA), European Medicines Agency (EMA), and International Conference on Harmonization (ICH) of Technical Requirements for Registration of Pharmaceuticals for Human Use: Guidance on Statistical Principles in Clinical Trials<sup>1</sup>. All work planned and reported for this SAP will follow internationally accepted guidelines, published by the American Statistical Association<sup>2</sup> and the Royal Statistical Society<sup>3</sup>, for statistical practice.

The planned analyses identified in this SAP may be included in clinical study reports (CSRs), regulatory submissions, or future manuscripts. Also, post-hoc exploratory analyses not necessarily identified in this SAP may be performed to further examine study data. Any post-hoc or unplanned, exploratory analysis performed and included in the CSR will be clearly identified as such in the final CSR.

The statistical plan described hereafter is an *a priori* plan. It will be submitted to file prior to any unblinded inferential or descriptive analysis of data pertaining to Arcutis Biotherapeutics, Inc.'s study ARQ-154-203.

#### 2. **Study Objectives and Endpoints**

#### 2.1. **Study Objectives**

#### 2.1.1. Primary Objective

The primary objective is to assess the safety and efficacy of ARQ-154 foam 0.3% (Roflumilast Foam 0.3%) administered once daily (QD) vs vehicle foam x 8 weeks in adult subjects with seborrheic dermatitis

#### 2.2. **Study Endpoints**

#### 2.2.1. Safety Endpoints

The safety endpoints of this study include the following:

- Local tolerability assessments
- Clinical laboratory parameters
- Adverse events (AEs)
- Columbia-Suicide Severity Rating Scale (C-SSRS)



- Patient Health Questionnaire depression scale (PHQ-8)
- Vital signs
- Physical examinations

### 2.2.2. Efficacy Endpoints

### 2.2.2.1. Primary Efficacy Endpoint

The primary efficacy endpoint of this study is achievement of an Investigator Global Assessment (IGA) score of "clear" or "almost clear" PLUS a 2-grade improvement from baseline at Week 8.

### 2.2.2.2. Secondary Efficacy Endpoints

The secondary efficacy endpoints of this study include the following:

- Achievement of an IGA score of "clear" or "almost clear" PLUS a 2-grade improvement from baseline at weeks 2 and 4.
- Change from baseline in Overall Assessment of Erythema score at weeks 2, 4, and 8.
- Change from baseline in Overall Assessment of Scaling score at weeks 2, 4, and 8.
- Achievement of an Overall Assessment of Erythema (0-3 scale) score of 0 or 1 PLUS a 2-grade improvement from baseline at weeks 2, 4, and 8.
- Achievement of an Overall Assessment of Scaling (0-3 scale) score of 0 or 1 PLUS a 2-grade improvement from baseline at weeks 2, 4, and 8.
- Change and percent change in Worst Itch Numeric Rating Scale (WI-NRS) pruritus score at weeks 2, 4, and 8, as compared to baseline.
- In subjects with a baseline WI-NRS pruritus score of  $\geq 4$ , achievement of a  $\geq 4$ -point improvement from baseline in WI-NRS pruritus score at weeks 2, 4, and 8.

### 2.2.2.3. Exploratory Efficacy Endpoints

The exploratory efficacy endpoints of this study include the following:

- Change and percent change in Scalpdex total score from baseline at weeks 2, 4, and 8.
- Achievement of an Overall Assessment of Erythema (0-3 scale) score of 0 or 1 at weeks 2, 4, and 8.
- Achievement of an Overall Assessment of Scaling (0-3 scale) score of 0 or 1 at weeks 2, 4, and 8.
- Achievement of an Overall Assessment of Erythema (0-3 scale) score of 0 at weeks 2, 4, and 8.
- Achievement of an Overall Assessment of Scaling (0-3 scale) score of 0 at weeks 2, 4, and 8.
- Change and percent change from baseline in Dermatology Life Quality Index (DLQI) at weeks 2, 4, and 8.
- Change and percent change from baseline in body surface area (BSA) affected at week 8.
- A 2-grade improvement in IGA from Baseline.
- Incidence of a 2 point reduction from baseline in the WI-NRS (among subjects with WI-NRS ≥2 at baseline).
- Achievement of an IGA score of "clear" or "almost clear" PLUS a 2-grade improvement from Baseline at week 9.



- Change from baseline in Overall Assessment of Erythema score at week 9.
- Change from baseline in Overall Assessment of Scaling score at week 9.
- Achievement of an Overall Assessment of Erythema (0-3 scale) score of 0 or 1 PLUS a 2-grade improvement from baseline at week 9.
- Achievement of an Overall Assessment of Scaling (0-3 scale) score of 0 or 1 PLUS a 2-grade improvement from Baseline at week 9.

### 3. Overall Study Design and Plan

### 3.1. Overall Design

This is an 8-week, parallel group, double blind, vehicle-controlled study for the treatment of subjects with seborrheic dermatitis. This study will include both male and female adults having an IGA score of at least "Moderate" (3), and approximately 184 subjects will be enrolled. After having met all inclusion criteria, and none of the exclusion criteria, subjects will be randomized in a 2:1 ratio to ARQ-154 foam 0.3% QD (Roflumilast foam 0.3%) or Vehicle foam QD which will be applied to areas of lesions of seborrheic dermatitis. There will be screening for up to 4 weeks followed by 8 weeks of treatment phase. Subjects will have to apply the study drug once a day in the evening, except for on Day 0 and Week 2, the study drug is applied at the study site. Subjects have to record the date and time each dose has been applied, any missed doses, and any additional comments. There will be a follow-up visit approximately 1 week after treatment has been completed.

### 3.2. Sample Size and Power

A sample size of approximately 184 subjects is planned for the study. Subjects will be randomized in a 2:1 ratio to ARQ-154 foam 0.3% (Roflumilast Foam 0.3%): vehicle foam QD, stratified by study site and baseline disease severity. Approximately 121 subjects will receive ARQ-154 foam 0.3% QD (Roflumilast Foam 0.3%); approximately 63 subjects will receive vehicle foam QD. A sample size of 184 subjects will provide approximately 90% power to detect an active response of at least 58.5%, assuming 159 subjects complete the study and a vehicle response of 30%, based on two-group Chi-squared test of equal proportions (without continuity correction), using a 2-sided alpha of 0.10.

#### 3.3. Study Population

Study population consists of male and female subjects of age 18 years or older with no more than 20% BSA of seborrheic dermatitis. Subjects should have a minimum IGA of 'Moderate' (3) at baseline.

#### 3.4. Treatments Administered

Subjects who meet the eligibility criteria will be randomized to 1 of the 2 following treatment groups in a 2:1 ratio (active:vehicle):

- ARQ-154 foam 0.3% QD (Roflumilast Foam 0.3%)
- Matching vehicle foam QD.





### 3.5. Method of Assigning Subjects to Treatment Groups

Subjects will be randomized and assigned to active drug or vehicle in a 2:1 ratio according to a computer-generated randomization list. Randomization will be stratified by study site and baseline disease severity (IGA = 3 or IGA = 4).

### 3.6. Blinding and Unblinding

This is a double-blind study, therefore neither the subjects nor the Investigator, clinical personnel, or sponsor will be aware of which treatment an individual has received. Emergency unblinding will be done using the study internet-based randomization system (IWRS) system in consultation with the Medical Monitor and the sponsor's Chief Medical Officer (CMO).

#### 3.7. Schedule of Events

A detailed schedule of events for the study is provided in Table 1.





#### **Table 1: Schedule of Events**

| Study Procedure | Screen | Baseline<br>Day 0 | Wk 2<br>Day 14 | Wk 4<br>Day 28 | Wk 8<br>Day 56 | Wk 9<br>Day 63 |
|---|---|---|---|---|---|---|
| Visit | 1 | 2 | 3 | 4 | 5 | 6 |
| Visit Window | -4 weeks | | +/- 3 day | +/- 5 days | +/- 5 days | +/-5 days |
| Informed consent/assent | X | | | | | |
| Medical history | X | | | | | |
| Physical examination <sup>a</sup> | X | X | | | X | |
| I/E criteria | X | X | | | | |
| Randomization | | X | | | | |
| Hematology, Serum | | | | | | |
| Chemistries, and Urine | X | X | | | X | |
| Analysis | | | | | | |
| Vital signs, height, weight <sup>b</sup> | X | X | X | X | X | X |
| IGAc, Overall Assessment of | | | | | | |
| Erythema <sup>c</sup> , Overall Assessment | X | X | X | X | X | X |
| of Scaling <sup>c</sup> | | | | | | |
| WI-NRS, DLQI, Scalpdex | X | X | X | X | X | |
| BSA | X | X | | | X | |
| Application Site Reaction | | X | | X | X | |
| Assessment/Local Tolerability <sup>d</sup> | | Λ | | Λ | Λ | |
| Pigmentation Assessment <sup>e</sup> | X | X | X | X | X | X |
| C-SSRS, PHQ-8 | X | X | | X | X | |
| Medical Photography <sup>f</sup> | | X | X | X | X | |
| Pregnancy test <sup>g</sup> | X | X | | X | X | |
| PK draws <sup>h</sup> | | X | | X | X | |
| IP/vehicle application at the | | X | X | | | |
| study site <sup>i</sup> | | Λ | Λ | | | |
| Dispense study medication kit <sup>j</sup> | | X | X | X | | |
| Dispense/review diary | | X | X | X | X | |
| Weigh study medication kitk | | X | X | X | X | |
| Compliance calculation <sup>1</sup> | | X | X | X | X | |
| Adverse event assessment | X | X | X | X | X | X |
| Concomitant medications | X | X | X | X | X | X |

<sup>&</sup>lt;sup>a</sup> Limited physical examination: skin, lungs, and heart only

being taken. Remove any jackets, outerwear, and shoes. Remove any objects of significant weight (i.e., cell phones, wallet, key chains). A 5% weight loss from Baseline should be reported to the medical monitor.

<sup>&</sup>lt;sup>c</sup> IGA will be a 5-point scale ranging from clear (0) to severe (4). IGA should be completed prior to other physician assessments. Overall assessment of erythema (0-3 scale) and overall assessment of scaling (0-3 scale) will be completed.

d Local tolerability Assessments: The Investigator local tolerability assessment of skin irritation (Berger and Bowman skin irritation score) should be performed prior to the investigational product application at Baseline, and at Weeks 4 and 8. Reactions at the site of product application, which may occur post-Baseline, should be differentiated from the preexisting inflammation associated with the subject's seborrheic dermatitis. Subjects will perform the local tolerability

Statistical Analysis Plan, Sponsor Arcutis Biotherapeutics, Inc. Protocol Number ARQ-154-203 PCN Number ARCU210100



assessment 10-15 minutes post-drug application at Baseline, and recall assessments at Weeks 4 and 8 for the subject's '0-3' burning/stinging assessment.

- <sup>e</sup> An assessment for hypopigmentation and hyperpigmentation will be performed by the investigator at all clinic visits.
- f At selected sites, medical photography will be obtained for target lesions. All efforts will be made to de-identify the subjects. Subjects who are unwilling to participate in the medical photography will be allowed to opt out of this procedure.
- <sup>g</sup> A pregnancy test will be administered to all females of child-bearing potential. A serum pregnancy test will be performed at the Screening visit only. A urine pregnancy test will be performed at Baseline, Week 4, and Week 8. A negative result is required for continued participation in the study, and results must be available prior to dispensing of investigational product at each visit.
- <sup>h</sup> PK draws (trough / pre-dose) will be collected at Days 0, 28 and 56. At baseline, this draw will be pre-dose relative to drug application in the clinic. Ensure study medication is not applied in the area where PK will be drawn.
- <sup>i</sup> Subjects to apply assigned IP at the study site at every designated visit, to confirm understanding of instruction on how to apply initially.
- <sup>j</sup> Kits will be dispensed based on %BSA affected. See IP Handling Manual for details.
- <sup>k</sup> The entire kit should be weighed and recorded at every visit. See IP Handling Manual for details.
- <sup>1</sup> Compliance calculation is described in the IP Handling Manual.





### 4. Statistical Analysis and Reporting

#### 4.1. Introduction

Data processing, tabulation of descriptive statistics, calculation of inferential statistics, and graphical representations, will be performed primarily using SAS (release 9.4 or higher). If the use of other software is warranted for analyses conducted by Premier Research, the final statistical methodology report will detail what software was used for what purposes.

Continuous (quantitative) variable summaries will include the number of subjects (n) with non-missing values, mean, standard deviation (SD), median, minimum, and maximum.

Categorical (qualitative) variable summaries will include the frequency and percentage of subjects who are in the particular category or each possible value. In general, the denominator for the percentage calculation will be based upon the total number of subjects in the study population for the treatment group, unless otherwise specified.

Unless otherwise indicated, all statistical tests will be conducted at the 0.10 significance level using 2-tailed tests, and P values will be reported. Corresponding 90% confidence intervals (CIs) will be presented for statistical tests. In addition, 95% CIs have been added for the efficacy table summaries as requested by sponsor. Wilson confidence intervals for binomial proportions will be computed.

Statistical testing will be performed at the 0.10 level using two-tailed tests.

ARQ-154 0.3% foam will be described as "Roflumilast Foam 0.3%" throughout the tables, figures, and listings.

### 4.2. Interim Analysis and Data Monitoring

Based on protocol section 6.1.3, one interim futility analysis was planned when the first 60 subjects randomized and have had the opportunity to complete the 8 week disease assessment. This futility analysis will be nonbinding and will be used for decision making on further expansion of the clinical development program in seborrheic dermatitis. The sponsor considered that the analysis is no longer needed for decision making and interim analysis was not carried out upon their request. This interim analysis was not meant to change the accrual to or conduct of this trial.

### 5. Analysis Populations

The following analysis populations are planned for this study:

- Safety Population (SAF): The Safety population includes all subjects who are enrolled and received at least 1 confirmed dose of investigational product (IP). This population will be used for all safety analyses.
- Intent-To-Treat Population (ITT): The ITT population includes all randomized subjects. This population will be used as sensitivity analysis of primary and secondary endpoints along with disposition.



- Modified Intent-To-Treat Population (mITT): The mITT population includes all randomized subjects with the exception of subjects who missed the week 8 IGA assessment specifically due to the novel coronavirus disease (COVID-19) disruption. This population will be the primary analysis population for the analysis of efficacy endpoints.
- Pruritus Population (PRU4): The PRU population is a subset of the ITT population and includes subjects with WI-NRS pruritus score ≥4 at Baseline. This population will be used for the analysis of achievement of a 4-point reduction in WI-NRS pruritus score as compared to Baseline.
- **Pruritus Population (PRU2):** The PRU population is a subset of the ITT population and includes subjects with WI-NRS pruritus score ≥2 at Baseline. This population will be used for the analysis of achievement of a 2-point reduction in WI-NRS pruritus score as compared to Baseline.
- Pharmacokinetic Population (PK): The PK population will include all subjects receiving the active drug with sufficient plasma concentrations of roflumilast to define a profile, as determined by the pharmacokineticist. This population will be used for analyses of PK parameters. Analyses using the PK Population will be presented in a separate PK report, provided by the pharmacokineticist.

### 6. General Issues for Statistical Analysis

### 6.1. Statistical Definitions and Algorithms

#### 6.1.1. Baseline

The last observation recorded on or before the day of first dose of IP will be used as the baseline observation for all calculations of change from baseline for all the efficacy and vital signs data. For the laboratory and PHQ data, the last observation recorded before the first dose of IP will be used as the baseline observation for all calculations of change from baseline.

For subject tolerability assessments, baseline is derived as the last non-missing measurement taken on the day of first application of study drug.

### **6.1.2.** Adjustments for Covariates

If there is a statistical difference among treatment groups with respect to baseline characteristics, that variable may be added to the statistical models as a blocking factor or covariate to determine the effect on treatment.

Subgroup analyses may be generated for the baseline covariates.

### **6.1.3.** Multiple Comparisons

No adjustments will be made for multiple comparisons; all analyses will be conducted at the  $\alpha = 0.10$  level.



### 6.1.4. Handling of Dropouts or Missing Data

Any subject who prematurely withdraws from the study will have their last available data assigned to an analysis window as described in Section 6.1.5.

For the primary efficacy endpoint of IGA score, the primary analysis will impute missing values using a regression-based multiple imputation model. This is a three step process.

- 1. The first step is to understand the pattern of missingness. In order to perform the multiple imputation, a monotone missing pattern has to be achieved. For example, if there exists values for baseline and Week 8 visits, but missing values for the Week 2 or 4 visits, Markov-Chain Monte-Carlo (MCMC) method will be used to impute the small amount of missing data that may be missing at the intermediate visits that is required to make the missing data pattern monotone before applying the multiple imputation algorithm. This method uses a non-informative Jeffreys prior to derive the posterior mode from the expectation-maximization (EM) algorithm as the starting values for the MCMC method. MCMC method will use seed of 878508. The IGA score will be treated as a continuous variable for this step. To avoid values that could not be observed in practice, imputed values will be constrained to be integers in the range of 0 to 4.
  - a. The table below will determine the number of datasets to be imputed in this step. Determine the proportion of datapoints with non-monotone pattern across all visits and subjects which could be derived as a percentage of number of nonmonotone data points/total number of expected data points.

This can be determined as  $\frac{number\ of\ non\ montone\ visits}{total\ number\ of\ visits\ across\ all\ subjects}*100$ 

| Non-monotone<br>Missing Data | Number of Imputed Datasets |
|------------------------------|----------------------------|
| ≤ 2% | 1 |
| $> 2\%$ to $\le 5\%$ | 3 |
| > 5% | 10 |

2. Once the monotone pattern is achieved, the next step is to implement the imputation algorithm. For this, the Predictive Mean Matching method (PMM) will be used. This method is particularly helpful if the normality assumption is violated. For subjects with complete data up to a particular visit, a PMM model will be fit that includes the outcome at that visit as the dependent variable and as independent variables, baseline IGA score, treatment group, and investigational site at baseline using a seed of 633621. This process will be repeated 25 times, resulting in a total of 25 to 250 complete analysis datasets, depending on the number of imputed monotone datasets that are required. The seed may





be changed after unblinding in case of any issues with the imputation process, and it will be documented in the CSR if any change is required.

3. For each completed dataset, compute the necessary derived variables. The dichotomous success rate (clear or almost clear with at least a 2-point change from baseline) will be derived. The results obtained will be analyzed using the Cochran-Mantel-Haenszel (CMH) analysis for each of the complete analysis data sets stratified by baseline IGA score and site. The results will be combined into one multiple imputation inference (odds ratio, associated confidence interval and *P* value) using PROC MIANALYZE as illustrated<sup>4</sup>.

This approach to imputation should be superior to other strategies such as carrying forward the last available observation, which may yield unrealistic imputed values. Also, the use of multiple imputation avoids the problem of artificially increasing power through data imputation associated with single-imputation methods because it accounts for the uncertainty associated with the imputation. Other missing data will not be imputed, with the exception of incomplete dates as described in Section 6.1.8. For responder analysis, only observed data will be used. Only observed data will be summarized using descriptive statistics.

The SAS pseudo code for the multiple imputation process is listed below:

### Step 1:

```
proc mi data=example seed=878508 nimpute=XX round=1 out=example_1;
    mcmc impute=monotone;
    var <baseline score> ........... <visit8 score>;

run;

Step 2:

proc mi data=example_1 seed=633621 nimpute=XX out=example_2;
    class <treatment> <site>;
    monotone regpmm(<baseline score> ........... <visit8 score>);
    var <treatment> <site> <baseline score> ........... <visit8 score>;

run;

XX will be the determined based on the proportion of missing data across visits.
```

Step 3: This step involves running CMH test stratified by pooled site and baseline iga score on each completed dataset and combining the results using proc mianalyze.

```
proc freq data=example noprint;
by <imputationnumber> <visit> ;
tables <site>*<baseline score>*<treatment>*<outcome>/ cmh alpha=0.1;
output out=example_stat cmh;
run;
```

In order to apply PROC MIANALYZE, normalizing transformations have to be applied to odds ratio. *P* values are obtained using Wilson Hilferty transformation as illustrated<sup>4</sup>.





### 6.1.5. Analysis Visit Windows

Visits will be analyzed as scheduled. Unscheduled, early termination visits, and/or repeated measurements will only be included if a scheduled measurement is not available and the early termination or unscheduled/repeated measurement falls within the analysis visit windows as described in Table 2. The windows follow the Schedule of Events in Table 1. Unscheduled/repeated measurements will be listed.

**Table 2: Analysis Visit Windows** 

For Week 9 visit, only lower limit will be used and if the study day falls on or after the lower limit, the unscheduled or early termination visit would be set to week 9 as appropriately.

| Visit Name | Visit Number | Target Start Day | Lower Limit | Upper Limit |
|------------|--------------|------------------|-------------|-------------|
| Week 2 | 3 | 14 | 2 | 22 |
| Week 4 | 4 | 28 | 23 | 42 |
| Week 8 | 5 | 56 | 43 | 61 |
| Week 9 | 6 | 63 | 62 | |

### **6.1.6.** Pooling of Sites

Sites will be pooled for statistical analysis as follows. For analysis, sites should have a minimum of 10 randomized subjects. The smallest sites will be grouped sequentially in order of smallest to largest, restricting to those sites that did not meet the minimum enrollment of 10, until each pooled site has a minimum of 10 subjects with at least 1 subject in each treatment group.

### 6.1.7. Derived Variables

- **IGA success** = IGA of "Clear" or "Almost Clear" plus a 2-grade improvement from Baseline.
- **Compliance** = number of applications divided by the expected number of IP applications for each subject. Compliance will be calculated using drug accountability data over the entire treatment period for each subject, up to treatment completion or discontinuation.
  - **Number of expected IP applications** = calculated as last treatment date first treatment date + 1.
  - Treatment end date = for subjects that completed the study it is calculated as week 8 date obtained from COMP CRF. If subjects are missing week 8 date, the last available date from SV will be used. If subject discontinued from study, the last available COMP date will be used. In the absence of date in COMP page, the last available date from SV with visit performed will be used.
  - **Number of IP applications** = number of expected IP applications missed IP applications as collected in the CRF.



- Weight of IP (g) = dispensed can weight returned can weight.
- **BMI** (kg/m²) = (weight in kg)/[(height in cm/100)²]. For Week 2, and 4, baseline height will be used to derive BMI. For Week 8, and 9, Week 8 height will be used to derive BMI since height is not collected at all visits.
- BMI Categories;

• Underweight - BMI < 18.5

• Normal - 18.5 <= BMI <= 24.9

• Overweight  $-25.0 \le BMI \le 29.9$ 

• Obese - BMI >= 30.0

- WI-NRS 4-point reduction = achievement of a 4-point reduction in WI-NRS pruritus score at Weeks 2, 4, and 8 compared to baseline, calculated only for subjects with a pruritus score of  $\geq 4$  at baseline.
- WI-NRS 2-point reduction = achievement of a 2-point reduction in WI-NRS pruritus score at Weeks 2, 4, and 8 compared to baseline, calculated only for subjects with a pruritus score of ≥ 2 at baseline.
- **DLQI Score** = sum of the 10 questions (individual questions scored as Very much=3, A lot=2, A little=1, Not at all=0, Not relevant=0, Question 7: Yes=3, No=0, with Not relevant recorded to 0; range for score 0 to 30). If 1 item is missing, it is scored as 0 for that item. If 2 or more items are missing, the score should not be calculated.
- **PHQ-8** = sum of the 8 questions (individual questions scored as Not at all=0, Several days=1, More than half the days=2, and Nearly every day=3; range for score 0 to 24). If more than 1 item is missing the score should not be calculated. If 1 item is missing the score is calculated as (sum of answered items\*8)/number of answered items.
- Scalpdex score transformation = Scalpdex is rated on a 1 to 5 scale which will be transformed to 0 to 100 Scale where 1=0; 2=25; 3=50; 4=75; 5=100. This transformed score is used to calculate scale scores.
  - Emotions Scale = average of (Q2, Q4, Q5, Q6, Q7, Q9, Q10, Q11, Q12, Q14, Q16, Q17, Q19, Q20, Q22) after transforming to 0 to 100 scale as mentioned above.

Q refers to question number. Q19 will be reverse scored i.e., 1=100; 2=75; 3=50; 4=25; 5=0.

• Symptoms Scale = average of (Q1, Q3, Q8) after transforming to 0 to 100 scale as mentioned above. Q refers to question number.



- Functioning Scale = average of (Q13, Q15, Q18, Q21, Q23) after transforming to 0 to 100 scale as mentioned above. Q refers to question number.
- Scalpdex Total Score = calculated as mean of all the 23 scalpdex questions using the transformed scale of 0 to 100. Q19 will be reverse scored i.e., 1=100; 2=75; 3=50; 4=25; 5=0 while calculating the mean. Q refers to question number.
- Change from baseline = value at current time point value at baseline.
- TEAE = any AE with an onset date/time after the first application of IP.
- C-SSRS Suicidal Ideation = A "yes" answer at any time during treatment to any one of the five suicidal ideation questions (Categories 1-5: Wish to be Dead, Non-specific Active Suicidal Thoughts, Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act, Active Suicidal Ideation with Some Intent to Act, without Specific Plan Active Suicidal Ideation with Specific Plan and Intent).
- C-SSRS Suicidal Behavior = A "yes" answer at any time during treatment to any one of the five suicidal behavior questions (Categories 6-10: Preparatory Acts or Behavior, Aborted Attempt, Interrupted Attempt, Actual Attempt (non-fatal), Completed Suicide).

### 6.1.8. Data Adjustments/Handling/Conventions

All collected data will be presented in CDISC datasets. Data not subject to analysis according to this plan will not appear in any tables or graphs but will be included only in the CDISC datasets.

All P values will be displayed in four decimals and rounded using standard scientific notation (eg, 0.XXXX). If a P value less than 0.0001 occurs it will be shown in tables as <0.0001; similarly, if a P value greater than 0.9999 occurs it will be shown in tables as >0.9999.

Adverse events will be coded using the MedDRA version 23.0 thesaurus.

A treatment-related AE is any AE with a relationship to the study drug of possibly, probably, likely, or missing.

For partial AE and medication start dates:

- If the year is unknown, then do not impute the date but assign a missing value.
- If the year is known, but the month or month and day is unknown, then:
  - o If the year matches the year of first dose date and the end date (if present) is after first dose date, then impute as the month and day of the first dose date.
  - o Otherwise, assign 01 January.
- If the year and month are known, but the day is unknown, then:



- o If the month and year match the month and year of the first dose date, then impute as the day of the first dose date.
- o Otherwise, assign 01.

### For partial AE and medication end dates:

- If the year is unknown, then do not impute the date but assign as missing value.
- If the year is known, but the month or month and day is unknown, then:
  - o If the year matches the year of the last date of the study (date of last contact if subject lost to follow-up; date of completion or early termination otherwise), then impute as the month and day of the last date of the study.
  - Otherwise, assign 31 December.
- If the year and month are known, but the day is unknown, then:
  - o If the month and year match the month and year of the last date of the study, then impute as the day of the last date of the study.
  - Otherwise, assign the last day of the month.

### 6.2. Special Handling for COVID-19 Disruptions

In some cases, study visits will have to be delayed/not performed as a result of COVID-19 disruptions (e.g., sites were closed or subjects were under stay-at-home orders). Where possible, study sites may collect post-baseline data from subjects remotely by telemedicine; this will be clearly documented in the source. If possible, sites should adhere to the protocol visit window for remote data collection.

Investigator assessments and subject questionnaires normally completed directly in the tablet during on-site visits should be completed on the appropriate paper source documents. The following assessments/questionnaires are approved to be collected via telemedicine/remotely:

- WI-NRS
- DLQI
- Scalpdex
- C-SSRS
- PHO-8
- Subject Local Tolerability

The following assessments cannot be completed via telemedicine/remotely:

- IGA
- BSA
- Investigator Local Tolerability
- Overall Assessment of Erythema
- Overall Assessment of Scaling
- Pigmentation Assessment





### • Subject Weight

Study visits and procedures must be followed per protocol whenever possible. Any specific changes in study conduct that deviate from the protocol should be communicated to the institutional review board and Sponsor. All protocol deviations which occurred as a result of COVID-19 disruptions (e.g., visits out of window, missed assessments, etc.) will be differentiated from other protocol deviations.

Subjects who were affected by COVID-19 disruptions by either missing their Week 8 visit or being discontinued before having a Week 8 visit due to COVID-19 related disruptions will be excluded from the mITT population, as described in Section 

### 7. Study Patients/Subjects and Demographics

### 7.1. Disposition of Subjects and Withdrawals

Disposition will include tabulations of the number of subjects randomized into each treatment group, the number of subjects who received treatment, subjects completing the study, tabulated reasons for discontinuation from the study overall and due to COVID-19 disruption, and number of subjects in each analysis population. Disposition will be summarized for all subjects who were entered into database by treatment group and overall.

#### 7.2. Protocol Deviations

The number of subjects with major protocol deviations and/or eligibility deviations will be summarized in categories by treatment group and overall for subjects in Safety population.

### 7.3. Demographics and Other Baseline Characteristics

Summary statistics for age, gender (including child-bearing potential), race, ethnicity, height, weight, baseline disease characteristics (IGA, Overall Assessment of Erythema, Overall Assessment of Scaling, Scalpdex, WI-NRS), percent BSA, and BMI will be presented by treatment group and overall.

A summary of treatment history, including history of response, intolerance, or contraindication to topical corticosteroids and/or topical antifungals will be provided.

For the continuous variables, the number of non-missing values and the mean, standard deviation, minimum, median and maximum will be tabulated.

For ordinal variables such as the IGA, and WI-NRS, summary statistics including the mean, median, and range of the ordinal variable will be presented as well as frequency counts of each level of the ordinal variable.

For the categorical variables, the counts and proportions of each value will be tabulated.

These analyses will be conducted for the mITT and Safety populations.





### 7.4. Exposure and Compliance

The number of IP applications by each subject based on diary data will be summarized using descriptive statistics appropriate for continuous variables.

The amount of IP used by each subject based on can weight will be summarized descriptively by treatment group using continuous methods.

A subject will be considered compliant with the dosing regimen if the subject applies at least 80% of the expected applications during the IP application period and does not miss more than 3 consecutive doses.

Investigational product application compliance will be calculated based on number of applications divided by the expected number of IP applications. Compliance will be summarized descriptively by treatment group using the following categories:

- > 100%
- $\geq 80\% \leq 100\%$
- < 80%

### 8. Efficacy Analysis

### 8.1. Primary Efficacy Analysis

The IGA is an ordinal scale with five severity grades which is reported only in integers.

Table 3 illustrates the description of each severity grade.

Table 3: IGA

| Score | Description |
|---|---|
| 0 | <b>Completely clear:</b> No erythema, no scaling (hypo-hyperpigmentation can be present) |
| 1 | Almost clear: Residual slight erythema and/or trace amounts of scaling |
| 2 | Mild: Pink to red color and/or slight scaling |
| 3 | Moderate: Distinct redness and/or clearly visible scaling |
| 4 | <b>Severe:</b> Severe erythema (intense, fiery red) and/or severe scaling (coarse, thick scales with flaking onto clothes or skin) |





For this study, the primary estimand is the odds ratio of achieving IGA success at 8 weeks; that is, the ratio of the odds of achieving IGA success at 8 weeks ARQ-154 (Roflumilast Foam 0.3%) relative to the odds of success at 8 weeks of using a matching vehicle cream. In the course of the 8-week randomized treatment period, subjects may be exposed to possible known or unknown inter-current events that could possibly impact the estimand, such as treatment discontinuation due to a specific adverse effect or perhaps a lack of effect. However, the COVID-19 pandemic related issues may impact the integrity of the interpretation of the primary endpoint analysis; thus the "Principle Stratum Strategy" has been adopted to handle subjects impacted by COVID-19 related issues by removing them from the analysis entirely; thus the stratum of subjects included in this analysis are those who either have a Week 8 visit or were discontinued for a reason other than COVID-19 related issues. Discontinuations for any other reasons or other known or unknown intercurrent events will be handled using the "Treatment Policy Strategy" where the ITT principle will serve as the analytical basis for interpreting the estimand. In other words, the odds ratio of achieving IGA success for ARQ-154 (Roflumilast Foam 0.3%) relative to vehicle at 8 weeks will be evaluated regardless of the occurrence of any such intercurrent event, with the exception of subjects who are unable to attend the week 8 visit due to COVID-19 disruption. The study database will collect whether or not subjects missed a visit specifically due to COVID-19 disruption. It is the sponsor's assumption that data missing due to COVID-19 disruption are MCAR, and therefore, the mITT population will be no different than the ITT population for the purpose of generating this result. Under this assumption, the use of the mITT population will provide an unbiased estimate and facilitate the interpretation of the study in the presence of COVID-19 disruption. This estimand shall be estimated using the CMH approach. This approach produces an estimate which is the combined odds ratio resulting from adjusting for the possible effects of two classification factors – investigative site and baseline disease severity.

The primary efficacy endpoint is success in IGA of disease severity, defined as an IGA of "Clear" or "Almost Clear" plus a 2-grade improvement from Baseline at Week 8.

The primary endpoint will be analyzed using a CMH test stratified by site (throughout all analyses that use stratification, it will be based on the pooling algorithm described in Section 6.1.6) and baseline IGA. Statistical significance will be concluded at the 10% significance level (2-sided). Additionally, both 90% and 95% Wilson CIs for proportion of successes in each treatment group will be presented.

For the primary analysis, missing IGA scores will be imputed using multiple imputation as described in Section 6.1.4. These imputations will result in a minimum of 25 to a maximum of 250 complete analysis datasets, depending on the number of imputed monotone datasets that are required.

The CMH analyses will be performed separately for each of the complete analysis data sets, and the results will be combined into one multiple imputation inference (estimated treatment effect and associated CI and *P* value).

Sensitivity analyses of the primary endpoint will also be performed using the original (non-imputed) dataset. These will include a repeated measures logistic regression model (GEE) with IGA success as the dependent variable and treatment, site, baseline IGA score, and visit as the independent variables, as well as the above described CMH test on the non-imputed data.

All other missing data for all other analyses and summaries will remain missing and will not be





imputed. Only observed data will be included in the summaries showing descriptive statistics.

The primary efficacy analysis will be based on mITT population and these analyses will be repeated for the ITT population.

If subjects were unable to attend the week 8 visit due to COVID-19 related issues they will be excluded from the primary analyses for efficacy, which is handled by the mITT population.

### 8.2. Secondary Efficacy Analysis

All secondary efficacy analyses will be performed using the mITT and ITT populations.

#### 8.2.1. IGA

Achievement of an IGA score of "clear" or "almost clear" PLUS a 2-grade improvement from Baseline at weeks 2 and 4 will be analyzed similar to the primary efficacy endpoint using CMH test stratified by site, and baseline IGA with the exception that missing data will not be imputed. In addition, the number and percentage of subjects in each category will be summarized by treatment and visit. Additionally, both 90% and 95% Wilson CIs for proportion of successes in each treatment group will be presented.

### 8.2.2. Overall Assessment of Erythema

The assessment is performed at Screening, Baseline, and Weeks 2, 4, 8, and 9. The score is reported in ordinal scale with severity grades ranging from 0-3.

- Analysis of change and percent change from baseline in Overall Assessment of Erythema at Weeks 2, 4, and 8 will be performed using descriptive summaries (mean, median, inter quartile range) by treatment group and study visit. The treatment groups will be compared using an exact Wilcoxon rank-sum test as continuous variable. In addition, the number and percentage of subjects in each category will be summarized by treatment and study visit.
- Achievement of an Overall Assessment of Erythema (0-3 scale) score of 0 or 1 PLUS a 2-grade improvement from Baseline at Weeks 2, 4, and 8 will be analyzed using CMH tests stratified by site, and baseline IGA similar to the primary analysis above, with the exception that missing data will not be imputed. Additionally, both 90% and 95% Wilson CIs for proportion of successes in each treatment group will be presented.

Table 4 illustrates description of erythema grades.

**Table 4: Erythema Grades** 

| Score | Description |
|-------|------------------------------------------------------------|
| 0 | None: No evidence of erythema |
| 1 | Mild: Barely perceptible erythema which is faint or patchy |
| 2 | Moderate: Distinct erythema, |
| 3 | Severe: Intense (fiery red) erythema |





### 8.2.3. Overall Assessment of Scaling

This assessment is performed at Screening, Baseline, and Weeks 2, 4, 8, and 9. The score is reported in ordinal scale with severity grades ranging from 0-3.

- Analysis of change and percent change from baseline in Overall Assessment of Scaling score at weeks 2, 4, and 8 will be performed using descriptive summaries (median, inter quartile range) by treatment group and study visit. The treatment groups will be compared using an exact Wilcoxon rank-sum test as continuous variable.
- In addition, the number and percentage of subjects in each category will be summarized by treatment and visit. Achievement of an Overall Assessment of Scaling (0-3 scale) score of 0 or 1 PLUS a 2-grade improvement from Baseline at weeks 2, 4, and 8 will be analyzed using CMH tests stratified by site, and baseline IGA similar to the primary analysis above, with the exception that missing data will not be replaced. Additionally, both 90% and 95% Wilson CIs for proportion of successes in each treatment group will be presented.

Table 5 illustrates description of scaling grades.

**Table 5: Scaling Grades** 

| Score | Description |
|---|---|
| 0 | None: No scaling evident on lesions |
| 1 | Mild: Barely detectable, scattered, small flaking scales |
| 2 | Moderate: Scales clearly visible and prominent |
| 3 | <b>Severe:</b> Coarse, thick scales, with flaking into clothes or skin |

#### 8.2.4. WI-NRS

WI-NRS scale ranges from 0 to 10 with 0 being "no itch" and 10 equaling "worst imaginable itch". This will be determined by asking the subject's assessment of worst itch over the past 24 hours.

- Analysis of change from baseline in WI-NRS pruritus score at Weeks 2, 4, and 8 will be performed using descriptive summaries (mean, median, inter quartile range) by treatment group and study visit. In addition, the number and percentage of subjects for each scale score will be summarized by treatment and visit.
- Analysis of change from baseline in WI-NRS pruritus score at Weeks 2, 4, and 8 will be analyzed using an analysis of covariance with the factors treatment, study site (grouped as specified in Section 6.1.6), baseline IGA, and baseline value of the respective scale as independent variables. The LS Means, standard errors, 90% CIs, 95% CIs, and P values for change from baseline and testing difference in treatments will be presented.
- In subjects with a baseline WI-NRS pruritus score of ≥4, achievement of a ≥4-point improvement from baseline in WI-NRS pruritus score at Weeks 2, 4, and 8 will be analyzed using CMH tests stratified by site and baseline IGA similar to the primary analysis above, with the exception that missing data will not be replaced. This will be summarized using PRU4 population. Additionally, both 90% and 95% Wilson CIs for





proportion of successes in each treatment group will be presented.

### 8.3. Exploratory Efficacy Analysis

Exploratory efficacy analysis will be performed for subjects belonging to mITT and ITT populations.

The exploratory endpoints include:

- Change and percent change in Scalpdex total score from baseline at Weeks 2, 4, and 8
- Achievement of an Overall Assessment of Erythema (0-3 scale) score of 0 or 1 at Weeks 2, 4, and 8
- Achievement of an Overall Assessment of Scaling (0-3 scale) score of 0 or 1 at Weeks 2, 4, and 8
- Achievement of an Overall Assessment of Erythema (0-3 scale) score of 0 at Weeks 2, 4, and 8
- Achievement of an Overall Assessment of Scaling (0-3 scale) score of 0 at Weeks
   2, 4, and 8
- Change and percent change from baseline in DLQI at Weeks 2, 4, and 8
- Change and percent change from baseline in BSA affected at Week 8
- A 2-grade improvement in IGA from Baseline.
- Incidence of a 2 point reduction from baseline in the WI-NRS (among subjects with WI-NRS ≥ 2 at baseline
- Achievement of an IGA score of "clear" or "almost clear" PLUS a 2-grade improvement from Baseline at week 9.
- Change from baseline in Overall Assessment of Erythema score at week 9.
- Change from baseline in Overall Assessment of Scaling score at week 9.
- Achievement of an Overall Assessment of Erythema (0-3 scale) score of 0 or 1 PLUS a 2-grade improvement from baseline at week 9.
- Achievement of an Overall Assessment of Scaling (0-3 scale) score of 0 or 1 PLUS a 2-grade improvement from Baseline at week 9.

Scalpdex questionnaire consists of 23 questions which are categorized into emotions, symptoms and functioning scales. The scale scores and total score are calculated as described in the Section 6.1.7. Change and percent change from baseline for Scalpdex scale scores along with total score are summarized descriptively. In addition, number and percentages for each Scalpdex question is summarized by study visit and treatment group.

Change and percent change from baseline for DLQI, and BSA will be summarized descriptively. In addition change from baseline values for Scalpdex scale scores and total score, DLQI, and BSA will be analyzed using an analysis of covariance with the factors treatment, study site (grouped as specified in Section 6.1.6), baseline IGA, and baseline value of the respective scale as independent variables. Statistical comparisons between the treatment groups will be obtained using contrasts. The LS Means, standard errors, 90% CIs, 95% CIs, and P values for change from baseline and testing difference in treatments will be presented.





Analysis of 2 point reduction from baseline in the WI-NRS (among subjects with WI-NRS  $\geq$  2 at baseline) will be conducted similarly as described in Section 8.2.4; i.e., CMH test stratified by site and baseline IGA will be presented for Weeks 2, 4, and 8 for PRU2 population.

For efficacy analysis purposes, the data that is collected by ERT will be used for BSA summarization.

### 9. Safety and Tolerability Analysis

Safety will be evaluated from reported AEs, physical examinations, local tolerability assessments, changes in clinical laboratory values, changes in vital signs/weight, C-SSRS, and PHQ-8 results.

All safety analyses will be performed on the Safety population.

#### 9.1. Adverse Event

All AEs, TEAEs, and SAEs will be coded using the MedDRA dictionary version 23.0.

A treatment emergent AE (TEAE) is defined as an AE that started post application of IP at the Baseline visit through study completion. An overall summary of TEAEs will be provided; this will present number and percent of subjects who reported at least 1: TEAE (including all TEAEs, TEAEs by maximum severity, and TEAEs by greatest relationship), SAE, discontinued the study due to a TEAE, or had a TEAE resulting in death.

The number and percent of subjects reporting TEAEs, grouped by MedDRA system organ class and preferred term, will be tabulated by severity or greatest relationship to study IP and treatment group. In the case of multiple occurrences of the same TEAE within the same subject, each subject will only be counted once for each preferred term.

In the summaries showing severity and relationship to study medication the event with the maximum severity (mild < moderate < severe) or strongest relationship (not related < related) will be reported. If a particular event is missing the severity and/or relationship, then the strongest possible severity or relationship will be assumed for analysis (severity = severe, relationship = likely).

In the AE data listings, all AEs will be displayed. AEs that are treatment emergent will be flagged.

### 9.1.1. Adverse Events Leading to Withdrawal

A summary of incidence rates (frequencies and percentages) of TEAEs leading to withdrawal of study drug, by treatment group, SOC, and preferred term will be prepared for the Safety Population. No inferential statistical tests will be performed.

A data listing of AEs leading to withdrawal of study drug will also be provided, displaying details of the event(s) captured on the CRF.

#### 9.1.2. Deaths and Serious Adverse Events

Any deaths that occur during the study will be listed.





Serious adverse events (SAEs) will be listed and tabulated by system organ class and preferred term and presented by treatment group, severity, and relationship to study treatment.

### 9.2. Local Tolerability Assessments

The investigator's assessment of the application site reaction will be summarized by study visit using both categorical methods (number and percentage of subject with each score) as well as continuous methods (e.g., mean, median, etc.). Categorical summaries will be provided for dermal response as well as other effects. No inferential statistical tests will be performed.

The subject's assessment of the application site reaction will be summarized similarly.

### 9.3. Clinical Laboratory Evaluations

Laboratory test results will be summarized descriptively by treatment and study visit as both observed values and change from baseline values for continuous hematology, chemistry, and urinalysis results. Categorical urinalysis results will be summarized using frequencies by study visit and treatment.

The number of subjects with clinical laboratory values below, within, or above the normal range by study visit and in relation to baseline will be tabulated for each clinical laboratory analyte by treatment group (shift table).

Abnormal results will be flagged in the listings. In addition, pregnancy test results and hormonal laboratory results will be listed.

#### 9.4. Vital Signs

Descriptive summaries of observed values and changes from baseline will be calculated for systolic blood pressure, diastolic blood pressure, heart rate, height, weight, body mass index and oral body temperature by treatment group and visit.

Changes in weight by treatment group will summarize the number of subjects who gain or lose >=5% of their baseline body weight during the course of the study, as well as subjects who gain or lose >=10% of their baseline body weight over the course of the study by treatment group and visit.

BMI is derived as specified in Section 6.1.7. Shift tables by treatment group for subjects who shift from their baseline BMI category (underweight, normal, overweight, obese) to a different BMI category throughout the course of the study will be provided by treatment group and visit.

Upon sponsor's request, shift in BMI, and changes in weight are summarized by intentional and unintentional or missing weight loss question captured in the CRF.





### 9.5. PHQ-8

Data for PHQ-8 will be classified using each subject's total score at a time point into a category based on the following scoring system:

- None Minimal depression (0 to 4)
- Mild depression (5 to 9)
- Moderate depression (10 to 14)
- Moderately severe depression (15 to 19)
- Severe depression (20 to 24)

Shift tables showing the category of severity at each visit by treatment group will be presented.

### 9.6. **C-SSRS**

The C-SSRS is a questionnaire that prospectively assesses Suicidal Ideation and Suicidal Behavior. At the Screening study visit, "Baseline/Screening" version of the C-SSRS will be used. This version assesses Suicidal Ideation and Suicidal Behavior during the subject's lifetime and during the past 6 months. For the Screening visit, "lifetime" experience of the subject with Suicidal Ideation and Suicidal Behavior will be summarized. From Baseline visit, the "Since Last Visit" version will be used.

Suicidality data collected on the C-SSRS will be listed for all subjects. Tables will include results from the Suicidal Ideation and Suicidal Behavior sections of the C-SSRS. Frequencies and percentages of subjects with a response of "Yes" at any point on the Suicidal Ideation and Suicidal Behavior items will be summarized by study visit and treatment group.

### 9.7. Physical Examination

The number and percentage of subjects with normal and abnormal findings in the physical examination will be displayed at each study visit and treatment group.

#### 9.8. Concomitant Medication

Prior and concomitant medications will be summarized descriptively by treatment group, ATC level 4, and preferred term using counts and percentages.

Prior medications will be presented separately from concomitant medications. Medications that started before the first application of IP will be considered prior medications whether or not they were stopped prior to the first application of study drug. Any medications continuing or starting after the first application of study drug will be considered to be concomitant. If a medication starts before the first application of study drug and continues after the first application of study drug it will be considered both prior and concomitant.

Medications will be coded using WHODrug Global B3, version September 2019.





### 10. Changes from Planned Analysis

Based on protocol amendment, the significance level has been changed from 0.05 to 0.10. However, protocol Section 6.3.1 indicates alpha = 0.05 but section 6.1 indicates significance level to be 0.10. The alpha level of 0.10 is the intended level, and this SAP uses 0.10 as significance level as documented throughout. The PRU4 and PRU2 populations have been added to facilitate WI-NRS analysis. These populations are not included in the protocol. Additional exploratory endpoints have been added in the SAP which are not specified in the protocol. They are:

- Incidence of a 2 point reduction from baseline in the WI-NRS (among subjects with WI-NRS > 2 at baseline
- Achievement of an IGA score of "clear" or "almost clear" PLUS a 2-grade improvement from Baseline at week 9
- Change from baseline in Overall Assessment of Erythema score at week 9
- Change from baseline in Overall Assessment of Scaling score at week 9
- Achievement of an Overall Assessment of Erythema (0-3 scale) score of 0 or 1 PLUS a 2-grade improvement from baseline at week 9
- Achievement of an Overall Assessment of Scaling (0-3 scale) score of 0 or 1 PLUS a 2-grade improvement from Baseline at week 9.
- In addition, percentage change from baseline summaries have been added for Scalpdex, DLQI, BSA and WI-NRS.

Based on the sponsor's request the following changes have been made:

- 95% CIs have been added in the efficacy table summaries along with 90% CIs as the alpha level is 0.1.
- If a subject is unable to attend the week 8 visit due to COVID-19, they will be excluded from the primary analyses for efficacy. To facilitate this, mITT population has been added to replace the ITT population.
- The ITT population will be used as a sensitivity analysis of the primary, secondary, and exploratory efficacy analysis along with disposition.
- ANCOVA analysis has been added for change in baseline scores of Erythema, Scaling and WI-NRS.
- A new BMI shift table has been added.
- Shift from baseline in Weight and BMI tables are repeated based on the intentional/nonintentional or missing weight loss question captured in the CRF.
- For efficacy analysis purposes, data collected from ERT will be used for BSA summarization.
- Per Protocol population and associated analyses have been removed as they were considered to be uninformative.
- ANCOVA analysis have been added for change from baseline scores for WI-NRS and BSA.
- Wilcoxon rank sum test has been added to summarize the continuous data associated with Overall Assessment of Erythema and Scaling.





An interim analysis was planned to make a decision on further expansion of the clinical development program for seborrheic dermatitis. The sponsor considered the interim analysis as no longer needed for decision making and therefore no interim analysis was conducted. The interim analysis was not meant to change enrollment or conduct of this trial.

### 11. Other Planned Analysis

### 11.1. Pharmacokinetic Analysis

All PK collection information from the eCRF will be presented in a listing.

Concentration data and pk parameters will be summarized by timepoint (concentrations data) and treatment group using summary statistics. In addition, PK concentration and parameter listings will be presented as well.

#### 12. References

- 1. US Federal Register. (1998) International Conference on Harmonization; Guidance on Statistical Principles for Clinical Trials. Department of Health and Human Services: Food and Drug Administration [Docket No. 97D-0174]. Federal Register Volume 63, Number 179, pages 49583-49598. September 16, 1998.
- 2. ASA. (2016) Ethical Guidelines for Statistical Practice. Prepared by the Committee on Professional Ethics, April 2016. http://www.amstat.org/about/ethicalguidelines.cfm
- 3. RSS. (2014) The Royal Statistical Society: Code of Conduct, 2014. http://www.rss.org.uk/Images/PDF/join-us/RSS-Code-of-Conduct-2014.pdf.
- 4. Ratitch, B., Lipkovich, I., & O'Kelly, M. (2013). *Combining Analysis Results from Multiply Imputed Categorical Data*. PharmaSUG. <a href="https://www.pharmasug.org/proceedings/2013/SP/PharmaSUG-2013-SP03.pdf">https://www.pharmasug.org/proceedings/2013/SP/PharmaSUG-2013-SP03.pdf</a>

### 13. Tables, Listings, and Figures

All TLFs will have a header showing the sponsor company name and protocol and a footer showing the version of SAS, the file name and path, and the source of the data (e.g., listing number).

### 13.1. Planned Table Descriptions

The following are planned summary tables for protocol number ARQ-154-203. The table numbers and page numbers are place holders only and will be determined when the tables are produced.





## 13.1.1. Demographic Data

**Table 6: Demographic Data Summary Tables** 

| Number | Population | Title | Topline |
|---|---|---|---|
| Table 14.1.1 | All<br>Randomized | Summary of Subject Disposition | X |
| Table 14.1.2.1 | Safety | Summary of Demographics and Baseline<br>Characteristics | X |
| Table 14.1.2.2 | mITT | Summary of Demographics and Baseline<br>Characteristics | |
| Table 14.1.3 | Safety | Previous Treatment History of Seborrheic<br>Dermatitis | X |
| Table 14.1.4 | Safety | Summary of Protocol Deviations | |
| Table 14.1.5 | Safety | Summary of Prior Medications by ATC<br>Class Level 4 and Preferred Term | |
| Table 14.1.6 | Safety | Summary of Study Drug Exposure and Compliance | |

## 13.1.2. Efficacy Data

**Table 7: Efficacy Data Summary Tables** 

| Number | Population | Title | Topline |
|---|---|---|---|
| Table 14.2.1.1 | mITT | Summary and Change from Baseline in<br>Investigator Global Assessment (IGA)<br>Grades by Study Visit – Observed Data | |
| Table 14.2.1.2 | ITT | Summary and Change from Baseline in<br>Investigator Global Assessment (IGA)<br>Grades by Study Visit – Observed Data | |
| Table 14.2.1.3 | mITT | Summary and Change from Baseline in<br>Investigator Global Assessment (IGA)<br>Grades by Study Visit – Multiple Imputation | X |
| Table 14.2.1.4 | ITT | Summary and Change from Baseline in<br>Investigator Global Assessment (IGA)<br>Grades by Study Visit – Multiple Imputation | |
| Table 14.2.1.6 | mITT | Summary of Investigator Global Assessment (IGA) Grades and Success by Study Visit Categorical Results – Observed Data | |



| Number | Population | Title | Topline |
|---|---|---|---|
| Table 14.2.1.7 | ITT | Summary of Investigator Global Assessment (IGA) Grades and Success by Study Visit Categorical Results – Observed Data | |
| Table 14.2.1.9 | mITT | Summary of Investigator Global Assessment (IGA) Grades and Success by Study Visit – Multiple Imputation Categorical Results | X |
| Table 14.2.1.10 | ITT | Summary of Investigator Global Assessment (IGA) Grades and Success by Study Visit – Multiple Imputation Categorical Results | |
| Table 14.2.1.11 | mITT | Summary of Investigator Global Assessment (IGA) Grades and Success by Study Visit Tabulation of Fitted Point Estimates from Generalized Estimating Equations for Binary Response – Observed Data | |
| Table 14.2.1.12 | ITT | Summary of Investigator Global Assessment (IGA) Grades and Success by Study Visit Tabulation of Fitted Point Estimates from Generalized Estimating Equations for Binary Response – Observed Data | |
| Table 14.2.1.13 | mITT | Summary of Investigator Global Assessment (IGA) – 2-grade Improvement from Baseline – Observed Data | |
| Table 14.2.2.1 | mITT | Summary and Change from Baseline in<br>Overall Assessment of Erythema – Severity<br>Grades by Study Visit – Wilcoxon Test | |
| Table 14.2.2.2 | mITT | Summary of Overall Assessment of Erythema – Severity Grades and Success by Study Visit Categorical Results | X |
| Table 14.2.2.3 | ITT | Summary and Change from Baseline in<br>Overall Assessment of Erythema – Severity<br>Grades by Study Visit | |
| Table 14.2.2.4 | ITT | Summary of Overall Assessment of<br>Erythema – Severity Grades and Success by<br>Study Visit<br>Categorical Results | |



| Number | Population | Title | Topline |
|---|---|---|---|
| Table 14.2.2.5 | mITT | Summary of Overall Assessment of Erythema – Success Score of 0 or 1 and Success Score of 0 by Study Visit | |
| Table 14.2.2.6 | ITT | Summary of Overall Assessment of Erythema – Success Score of 0 or 1 and Success Score of 0 by Study Visit | |
| Table 14.2.2.7 | mITT | Summary and Change from Baseline in<br>Overall Assessment of Erythema – Severity<br>Grades by Study Visit – Wilcoxon Test | |
| Table 14.2.2.8 | ITT | Summary and Change from Baseline in<br>Overall Assessment of Erythema – Severity<br>Grades by Study Visit – Wilcoxon Test | |
| Table 14.2.3.1 | mITT | Summary and Change from Baseline in<br>Overall Assessment of Scaling – Severity<br>Grades by Study Visit | |
| Table 14.2.3.2 | mITT | Summary of Overall Assessment of Scaling –<br>Severity Grades and Success by Study Visit<br>Categorical Results | X |
| Table 14.2.3.3 | ITT | Summary and Change from Baseline in<br>Overall Assessment of Scaling – Severity<br>Grades by Study Visit | |
| Table 14.2.3.4 | ITT | Summary of Overall Assessment of Scaling –<br>Severity Grades and Success by Study Visit<br>Categorical Results | |
| Table 14.2.3.5 | mITT | Summary of Overall Assessment of Scaling – Success Score of 0 or 1 and Success Score of 0 by Study Visit | |
| Table 14.2.3.6 | ITT | Summary of Overall Assessment of Scaling – Success Score of 0 or 1 and Success Score of 0 by Study Visit | |
| Table 14.2.3.7 | mITT | Summary and Change from Baseline in<br>Overall Assessment of Scaling – Severity<br>Grades by Study Visit – Wilcoxon Test | |
| Table 14.2.3.8 | ITT | Summary and Change from Baseline in<br>Overall Assessment of Scaling – Severity<br>Grades by Study Visit – Wilcoxon Test | |
| Table 14.2.4.1 | mITT | Summary and Change from Baseline in<br>Worst Itch – Numeric Rating Scale (WI-<br>NRS) Pruritus Score by Study Visit | X |
| Table 14.2.4.2 | ITT | Summary and Change from Baseline in<br>Worst Itch – Numeric Rating Scale (WI-<br>NRS) Pruritus Score by Study Visit | |



| Number | Population | Title | Topline |
|---|---|---|---|
| Table 14.2.4.3 | PRU4-mITT | Worst Itch – Numeric Rating Scale (WI-NRS) Pruritus Score Success by Study Visit | X |
| Table 14.2.4.4 | PRU2-mITT | Worst Itch – Numeric Rating Scale (WI-NRS) Pruritus Score Success by Study Visit | |
| Table 14.2.4.5 | PRU4-ITT | Worst Itch – Numeric Rating Scale (WI-NRS) Pruritus Score Success by Study Visit | |
| Table 14.2.4.6 | PRU2-ITT | Worst Itch – Numeric Rating Scale (WI-NRS) Pruritus Score Success by Study Visit | |
| Table 14.2.4.7 | mITT | Summary of Worst Itch – Numeric Rating<br>Scale (WI-NRS) by Study Visit - ANCOVA | |
| Table 14.2.4.8 | ITT | Summary of Worst Itch – Numeric Rating<br>Scale (WI-NRS) by Study Visit - ANCOVA | |
| Table 14.2.4.9 | mITT | Summary of Worst Itch - Numeric Rating<br>Scale (WI-NRS) by Study Visit - Categorical<br>Scale | |
| Table 14.2.4.10 | ITT | Summary of Worst Itch - Numeric Rating<br>Scale (WI-NRS) by Study Visit - Categorical<br>Scale | |
| Table 14.2.5.1 | mITT | Change from Baseline in Scalpdex by Study<br>Visit | |
| Table 14.2.5.2 | mITT | Summary of Scalpdex by Study Visit -<br>ANCOVA | |
| Table 14.2.5.3 | ITT | Change from Baseline in Scalpdex by Study<br>Visit | |
| Table 14.2.5.4 | ITT | Summary of Scalpdex by Study Visit -<br>ANCOVA | |
| Table 14.2.5.5 | mITT | Categorical Summary of Individual<br>Responses by Study Visit – Scalpdex<br>Questionnaire | |
| Table 14.2.5.6 | ITT | Categorical Summary of Individual<br>Responses by Study Visit – Scalpdex<br>Questionnaire | |
| Table 14.2.6.1 | mITT | Change from Baseline in Dermatology Life<br>Quality Index (DLQI) by Study Visit | |
| Table 14.2.6.2 | mITT | Summary of Dermatology Life Quality Index (DLQI) by Study Visit – ANCOVA | |
| Table 14.2.6.3 | ITT | Change from Baseline in Dermatology Life<br>Quality Index (DLQI) by Study Visit | |
| Table 14.2.6.4 | ITT | Summary of Dermatology Life Quality Index (DLQI) by Study Visit – ANCOVA | |



| Number | Population | Title | Topline |
|---|---|---|---|
| Table 14.2.7.1 | mITT | Change from Baseline in Body Surface Area (BSA) by Study Visit | |
| Table 14.2.7.2 | mITT | Summary of Body Surface Area (BSA) by<br>Study Visit – ANCOVA | |
| Table 14.2.7.3 | ITT | Change from Baseline in Body Surface Area (BSA) by Study Visit | |
| Table 14.2.7.4 | ITT | Summary of Body Surface Area (BSA) by<br>Study Visit – ANCOVA | |

# 13.1.3. Safety Data

## **Table 8: Safety Data Summary Tables**

| Number | Population | Title | Topline |
|---|---|---|---|
| 14.3.1 Displays of Adverse Events | | | |
| Table 14.3.1.1 | Safety | Summary of Treatment Emergent Adverse Events | X |
| Table 14.3.1.2 | Safety | Incidence of Treatment Emergent Adverse Events by System Organ Class and Preferred Term | |
| Table 14.3.1.3 | Safety | Incidence of Treatment Emergent Adverse Events by System Organ Class, Preferred Term, and Maximum Severity | |
| Table 14.3.1.4 | Safety | Incidence of Treatment Emergent Adverse Events by System Organ Class,<br>Preferred Term, and Relationship to Study Drug | |
| Table 14.3.1.5 | Safety | Incidence of Treatment Emergent Adverse Events Leading to Study Drug<br>Discontinuation by System Organ Class and Preferred Term | |
| 14.3.2 Summai | ry of Deaths, | Other Serious and Significant Adverse Events | |
| Table 14.3.2.1 | Safety | Incidence of Serious Adverse Events by System Organ Class and Preferred Term | |
| Table 14.3.2.2 | Safety | Incidence of Serious Adverse Events by System Organ Class, Preferred Term, and Relationship to Study Drug | |
| Table 14.3.2.3 | Safety | Incidence of Serious Adverse Events by System Organ Class, Preferred Term, and Maximum Severity | |
| 14.3.3 Narrativ | es of Deaths, | Other Serious and Certain Other Significant Adverse Events | |
| Table 14.3.3.1 | Safety | Listing of Adverse Events Leading to Study Drug Discontinuation | |
| Table 14.3.3.2 | Safety | Listing of Serious Adverse Events | |
| Table 14.3.3.3 | Safety | Listing of Deaths | |
| 14.3.4 Abnormal Laboratory Value | | | |
| NA | | | |



| Number | Population | Title | Topline |
|---|---|---|---|
| 14.3.5 Laborat | tory Data Sur | nmary Tables | |
| Table 14.3.5.1.1 | Safety | Summary of Serum Chemistry Laboratory Results by Study Visit | |
| Table 14.3.5.1.2 | Safety | Shift from Baseline in Clinical Chemistry Laboratory Results by Study<br>Visit | |
| Table 14.3.5.2.1 | Safety | Summary of Hematology Laboratory Results by Study Visit | |
| Table 14.3.5.2.2 | Safety | Shift from Baseline in Hematology Laboratory Results by Study Visit | |
| Table 14.3.5.3.1 | Safety | Summary of Quantitative Urinalysis Laboratory Results by Study Visit | |
| Table 14.3.5.3.2 | Safety | Shift from Baseline in Quantitative Urinalysis Laboratory Results by Study Visit | |
| Table 14.3.5.3.3 | Safety | Summary of Qualitative Urinalysis Laboratory Results by Study Visit | |
| 14.3.6 Other S | afety Data Su | ımmary Tables | |
| Table 14.3.6.1 | Safety | Shift from Baseline in Patient Health Questionnaire (PHQ-8) by Study Visit | |
| Table 14.3.6.2.1 | Safety | Summary of Investigator Local Tolerability Assessment by Study Visit | |
| Table 14.3.6.2.2 | Safety | Summary of Investigator Local Tolerability Assessment (Dermal Response) by Study Visit Categorical Results | |
| Table 14.3.6.2.3 | Safety | Summary of Investigator Local Tolerability Assessment (Other Effects) by Study Visit Categorical Results | |
| Table 14.3.6.3.1 | Safety | Summary of Subject Local Tolerability Assessment by Study Visit | |
| Table 14.3.6.3.2 | Safety | Summary of Subject Local Tolerability Assessment by Study Visit<br>Categorical Results | X |
| Table 14.3.6.4.1 | Safety | Summary of Vital Signs by Study Visit | |
| Table 14.3.6.4.2 | Safety | Shift from Baseline in Weight by Study Visit | |
| Table 14.3.6.4.3 | Safety | Shift from Baseline in BMI by Study Visit | |
| Table 14.3.6.4.4 | Safety | Shift from Baseline in Weight by Study Visit – by Weight Loss Intentional/Non-Intentional | |




| Number | Population | Title | Topline |
|---|---|---|---|
| Table 14.3.6.4.5 | Safety | Shift from Baseline in BMI by Study Visit – by Weight Loss Intentional/Non-Intentional | |
| Table 14.3.6.5 | Safety | Summary of Columbia-Suicide Severity Rating Scale (C-SSRS) Suicidal Ideation and Suicidal Behavior by Study Visit | |
| Table 14.3.6.6 | Safety | Summary of Physical Examination by Study Visit | |
| Table 14.3.6.7 | Safety | Summary of Concomitant Medications by ATC Class Level 4 and Preferred Term | |
| 14.4 Pharmaco | kinetic and I | Pharmacodynamic Summary Tables | |
| 14.4.1.1 | PK | Summary of Pharmacokinetic Results by Study Visit | |
| 14.4.1.2 | PK | Summary of Pharmacokinetic Parameters by Study Visit | |





### 13.2. Planned Listing Descriptions

The following are planned data and patient/subject data listings for protocol number ARQ-154-203.

In general, one listing will be produced per CRF domain. All listings will be sorted by site, and subject number. All calculated variables will be included in the listings. Screen failures will only be presented in Listing 16.2.2.1.

In all listings a blank line will be placed between each subject. Within a data listing, if an item appears line after line (e.g., repetition of subject number), then only the first occurrence will be displayed.

In data listings, the information for one subject will be kept on one page if at all possible, rather than splitting a subject's information across pages.

**Table 9: Planned Listings** 

| Number | Population | Title |
|---|---|---|
| 16.2.1 Subject Disco | ontinuations/Comp | letions |
| Listing 16.2.1.1 | All Subjects | Subject Disposition |
| Listing 16.2.1.2 | All Subjects | Subject Visits |
| 16.2.2 Protocol Dev | iations | |
| Listing 16.2.2.1 | All Subjects | Inclusion and Exclusion Criteria Not Met |
| Listing 16.2.2.2 | All Subjects | Protocol Deviations |
| 16.2.3 Subjects Excl | luded from the Effi | cacy Analyses |
| Listing 16.2.3 | All Subjects | Analysis Populations |
| 16.2.4 Demographic | Data and Other B | aseline Characteristics |
| Listing 16.2.4.1 | All Subjects | Subject Demographics |
| Listing 16.2.4.2 | All Subjects | Medical History |
| 16.2.5 Compliance a | and/or Drug Conce | ntration Data |
| Listing 16.2.5.1 | All Subjects | Study Drug Application at the Study Site |
| Listing 16.2.5.2 | All Subjects | Cans |
| Listing 16.2.5.3 | All Subjects | Diary Dispensation |
| Listing 16.2.5.4 | All Subjects | Compliance (CRF) |
| Listing 16.2.5.5 | All Subjects | Missed Doses |
| Listing 16.2.5.6 | PK | Pharmacokinetic Blood Collection |
| Listing 16.2.5.7 | PK | Pharmacokinetic Calculated Parameters |
| 16.2.6 Individual Ef | fficacy Response Da | nta |
| Listing 16.2.6.1 | All Subjects | Investigator Global Assessment (IGA) |



| Number | Population | Title |
|---|---|---|
| Listing 16.2.6.2 | All Subjects | Overall Assessment of Erythema |
| Listing 16.2.6.3 | All Subjects | Overall Assessment of Scaling |
| Listing 16.2.6.4 | All Subjects | Worst Itch Numerical Rating Scale (WI-NRS) |
| Listing 16.2.6.5 | All Subjects | Scalpdex |
| Listing 16.2.6.6 | All Subjects | Dermatology Life Quality Index (DLQI) |
| Listing 16.2.6.7 | All Subjects | Body Surface Area (BSA) including Scalp |
| 16.2.7 Adverse Eve | nt Listings (by Subj | ect) |
| Listing 16.2.7.1 | All Subjects | Adverse Events |
| 16.2.8 Laboratory V | Values (by Subject) | |
| Listing 16.2.8.1.1 | All Subjects | Clinical Laboratory Data: Clinical Chemistry |
| Listing 16.2.8.1.2 | All Subjects | Clinical Laboratory Data: Hematology |
| Listing 16.2.8.1.3 | All Subjects | Clinical Laboratory Data: Urinalysis |
| Listing 16.2.8.1.4 | Female Subjects | Clinical Laboratory Data: Serum and Urine Pregnancy Test |
| 16.2.9 Other Clinic | al Observations and | Measurements (by Subject) |
| Listing 16.2.9.1 | All Subjects | Investigator Local Tolerability Assessments |
| Listing 16.2.9.2 | All Subjects | Subject Local Tolerability Assessments |
| Listing 16.2.9.3 | All Subjects | Pigmentation Assessment |
| Listing 16.2.9.4.1 | All Subjects | Vital Signs |
| Listing 16.2.9.4.2 | All Subjects | Vital Signs - Weight |
| Listing 16.2.9.5 | All Subjects | Physical Examination |
| Listing 16.2.9.6 | All Subjects | Medical Photography |
| Listing 16.2.9.7 | All Subjects | Prior and Concomitant Medications |
| Listing 16.2.9.8 | All Subjects | Patient Health Questionnaire (PHQ-8) |
| Listing 16.2.9.9 | All Subjects | Columbia-Suicide Severity Rating Scale (C-SSRS) |





## 14. Tables, Listings, and Listing Shells

## 14.1. Standard Layout for all Tables, Listings, and Figures

The following standard layout will be applied to all TLFs in support of this study. Note that programming notes may be added if appropriate after each TLF shell.



**premier** research

# Figure 1: Standardized Layout

| Arcutis Biotherapeutics, Inc.<br>Protocol: ARQ-154-203 | Page X of Y |
|---|---|
| <table, figure="" listing,=""> xx.x.x<br/><title figure="" listing="" of="" or="" table="">&lt;br&gt;&lt;Study Population and if applicable subgroup Description&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;Body of Table, Listing or Figure&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;&lt;Note: If directly Applicable&gt; Footnote 1 &lt;if applicable&gt; Footnote 2 &lt;if applicable&gt; Footnote n &lt;if applicable&gt; Footnote n &lt;if applicable&gt; Footnote n &lt;if applicable&gt; Footnote n+1 pgm path and name&gt;, &lt;date&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;/tbody&gt;&lt;/table&gt;</title></table,> | |



**premier** research



See Figure 2 below.



**premier** research



## Summary of Subject Disposition All Randomized Subjects Table 14.1.1

| | Roflumilast Foam 0.3% | Vehicle | Overall | ı |
|---|---|---|---|---|
| Status | (XX=N) | (N=XX) | (N=XX) | 1 |
| Study Populations: | | | | |
| ITŤ Population [1] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | |
| Safety Population [2] | XX (XX.X%) | (%X:X%) XX | XX (XX.X%) | |
| mITT Population [3] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | |
| PRU4 Population [4] | XX (XX.X%) | XX (XX.X%) | XX (XX:X%) | |
| PRU2 Population [5] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | |
| PK Population [6] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | |
| Completed Study | XX (XX.X%) | XX (XX.X%) | (%X:X%) | |
| Ongoing in Study | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | |
| Prematurely Discontinued from Study | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | |
| Reason for Discontinuation: | | | | |
| Withdrawal by Subject | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | |
| Sponsor's Decision | XX (XX.X%) | (%X:X%) XX | XX (XX.X%) | |
| Pl's Decision | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | |
| Non-Compliance | XX (XX.X%) | (%X:X%) XX | XX (XX.X%) | |
| Protocol Violation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | |
| Lost to Follow-up | XX (XX.X%) | (%X:X%) | XX (XX.X%) | |
| Adverse Event | XX (XX.X%) | XX (XX.X%) | XX (XX:X%) | |
| Death | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | |
| Pregnancy | XX (XX.X%) | (%X:X%) XX | (%X:X%) | |
| Other | XX (XX:X%) | XX (XX.X%) | (%X:XX) XX | |

Abbreviations: COVID-19 = novel coronavirus disease; IGA = investigator global assessment; ITT = Intent-to-treat; mITT = modified intent-to-treat; PI = principal investigator; PK = Pharmacokinetic; PRU2 = Subjects with WI-NRS Pruritus Score ≥2 at Baseline; PRU4 = Subjects with WI-NRS Pruritus Score ≥4 at Baseline; WI-NRS = Worst Itch - Numeric Rating Scale.

Note: Percentages are n/Number of subjects randomized within planned treatment and overall\*100.

The ITT population includes all randomized subjects.

[2] The Safety population includes all subjects who are enrolled and received at least 1 confirmed dose of IP.
[3] The mITT population includes all randomized subjects with the exception of subjects who missed the week 8 IGA assessment specifically due to COVID-19. disruption.

[4] The PRU4 population is a subset of the ITT population and includes subjects with WI-NRS pruritus score ≥ 4 at Baseline. This population will be used for the analysis of achievement of a 4-point reduction in WI-NRS pruritus score as compared to Baseline.

[5] The PRU2 population is a subset of the ITT population and includes subjects with WI-NRS pruritus score ≥ 2 at Baseline. This population will be used for the

analysis of achievement of a 2-point reduction in WI-NRS pruritus score as compared to Baseline.

[6] The PK population includes all subjects receiving the active drug with sufficient plasma concentrations of roflumilast to define a profile, as determined by the pharmacokineticist. This population will be used for analyses of PK parameters.

Reference Listings: 16.2.1, 16.2.3

Table 14.1.1 (cont.)





## Summary of Subject Disposition All Randomized Subjects

| Status | Roflumilast Foam 0.3%<br>(N=XX) | Vehicle<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|
| Prematurely Discontinued from the Study Due to COVID-19 Disruption Reason for Discontinuation: | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| XXXXXXXXX | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| XXXXXXXXX | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Abbreviations: COVID-19 = novel coronavirus disease; ITT = Intent-to-treat; IP = investigational product; PI = principal investigator; PK Pharmacokinetic.

Note: Percentages are n/Number of subjects randomized within planned treatment and overall\*100

The ITT population includes all randomized subjects.

[2] The Safety population includes all subjects who are enrolled and received at least 1 confirmed dose of IP. [3] The mITT population includes all randomized subjects with the exception of subjects who missed the week 8 disease assessment specifically due to COVID-19 disruption.

[4] The PRU2 population is a subset of the ITT population and includes subjects with WI-NRS pruritus score ≥ 4 at Baseline. This population will be used for the analysis of achievement of a 4-point reduction in WI-NRS pruritus score as compared to Baseline.

[5] The PRU2 population is a subset of the ITT population and includes subjects with WI-NRS pruritus score ≥ 2 at Baseline. This population will be used for the analysis of achievement of a 2-point reduction in WI-NRS pruritus score as compared to Baseline.

[6] The PK population will include all subjects receiving the active drug with sufficient plasma concentrations of roflumilast to define a profile, as determined by the pharmacokineticist. This population will be used for analyses of PK parameters.

Reference Listings: 16.2.1, 16.2.3

Programming note: "Ongoing in Study" row will be removed once the database has hardlocked and all subjects have completed the study; For COVID Disruption, list only the reasons for discontinuation as populated in the database.

Table 14.1.2.1 Summary of Demographics and Baseline Characteristics Safety Population

**premier** research

| Variable<br>Statistic or Category | Roflumilast Foam 0.3% (N=XX) | Vehicle<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|
| Age (years)<br>n<br>Mean (SD)<br>Median<br>Min, Max | XX | ()<br>XX XX XX<br>XX XX XX | XX |
| Gender<br>Male<br>Female | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) |
| Child-Bearing Potential? [1]<br>Yes<br>No | (%XXX)<br>XX (XXXX)<br>XX (XXXX) | (%X:XX)<br>XX (XX:X%)<br>XX (XX:X%) | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) |
| Ethnicity<br>Hispanic or Latino<br>Not Hispanic or Latino | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) |
| Race<br>American-Indian or Alaska Native<br>Asian<br>Black or African-American<br>Native Hawaiian or Other Pacific Islander<br>White<br>Other<br>More than One Race | (((((((((((((((((((((((((((((((((((((( | | |

Abbreviations: BSA = body surface area; IGA = investigator global assessment; WI-NRS = Worst Itch – Numeric Rating Scale. Note: Percentages are n/Number of subjects in the Safety population within treatment received and overall\*100. [1] Only captured for female subjects; percentages are based on the number of female subjects in the Safety population.

<sup>[2]</sup> The % BSA affected by seborrheic dermatitis.
[3] The WI-NRS will be determined by asking the subject's assessment of worst itch over the past 24 hours. The scale is from 0 to 10, which ranges from "no itch" to "worst imaginable itch".
Reference Listings: 16.2.4.1, 16.2.6.1, 16.2.6.1, 16.2.6.3, 16.2.6.5, 16.2.6.5, 16.2.6.7, 16.2.9.4.1, 16.2.9.4.2



Table 14.1.2 (cont.)
Demographics and Baseline Characteristics
Safety Population

| Variable<br>Statistic or Category | Roflumilast Foam 0.3% (N=XX) | Vehicle<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|
| Height (cm)<br>n<br>Mean (SD)<br>Median<br>Min, Max | ×××<br>×××<br>××××<br>×××× | (X<br>XX)<br>XX<br>XX<br>XX<br>XX<br>XX | ××××<br>××××<br>××××× |
| Weight (kg)<br>n<br>Mean (SD)<br>Median<br>Min, Max | XX XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX<br>XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XX XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| Body Mass Index (kg/m²)<br>n<br>Mean (SD)<br>Median<br>Min, Max | XX XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XX | XX |
| Body Surface Area (%) [2]<br>n<br>Mean (SD)<br>Median<br>Min, Max | XX.X(XX.XX)<br>XX.X.XX<br>XX.XX | XXX<br>XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XX |
| Baseline IGA<br>Completely Clear<br>Almost Clear<br>Mild<br>Moderate<br>Severe | (%%<br>%%<br>XXXXX<br>XXXX<br>XXX<br>XXXX<br>XXX<br>XXXX | (% % | (%XXX)<br>(%XXX)<br>(%XXX)<br>(%XXX)<br>(XXX)<br>(X |

Abbreviations: BSA = body surface area; IGA = investigator global assessment; WI-NRS = Worst Itch – Numeric Rating Scale. Note: Percentages are n/Number of subjects in the Safety population within treatment received and overall\*100. [1] Only captured for female subjects; percentages are based on the number of female subjects in the Safety population.

<sup>[2]</sup> The % BSA affected by seborrheic dematitis.
[3] The WI-NRS will be determined by asking the subject's assessment of worst itch over the past 24 hours. The scale is from 0 to 10, which ranges from "no itch" to "worst imaginable itch".
Reference Listings: 16.2.4.1, 16.2.6.1, 16.2.6.1, 16.2.6.3, 16.2.6.4, 16.2.6.5, 16.2.6.7, 16.2.9.4.1, 16.2.9.4.2



Table 14.1.2.1 (cont.)
Demographics and Baseline Characteristics
Safety Population

| Variable<br>Statistic or Category | Roflumilast Foam 0.3% (N=XX) | Vehicle<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|
| Baseline IGA - Numeric<br>n<br>Mean (SD)<br>Median<br>Min, Max | (X X X X X X X X X X X X X X X X X X X | XX | (X, X, X |
| Baseline Erythema<br>None<br>Mild<br>Moderate<br>Severe | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) |
| Baseline Scaling<br>None<br>Mild<br>Moderate<br>Severe | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) |
| Baseline Scalpdex<br>n<br>Mean (SD)<br>Median<br>Min, Max | (XX XX | ×× | XX |
| Baseline WI-NRS - Numeric [3]<br>n<br>Mean (SD)<br>Median<br>Min, Max | ×××<br>×××<br>×××<br>××× | ××××<br>××××<br>××××× | ×××<br>×××<br>××× |

Abbreviations: BSA = body surface area; IGA = investigator global assessment; WI-NRS = Worst Itch – Numeric Rating Scale. Note: Percentages are n/Number of subjects in the Safety population within treatment received and overall\*100. [1] Only captured for female subjects; percentages are based on the number of female subjects in the Safety population.

<sup>[2]</sup> The % BSA affected by seborrheic dermatitis.
[3] The WI-NRS will be determined by asking the subject's assessment of worst itch over the past 24 hours. The scale is from 0 to 10, which ranges from "no itch" to "worst imaginable itch".
Reference Listings: 16.2.4.1, 16.2.6.1, 16.2.6.2, 16.2.6.3, 16.2.6.5, 16.2.6.7, 16.2.9.4.1, 16.2.9.4.2

**premier** research



| Variable<br>Statistic or Category | Roflumilast Foam 0.3% (N=XX) | Vehicle<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|
| Baseline WI-NRS [3] | | | |
| 0 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| _ | XX (XX X%) | (%X:X%) XX | (%X:X%) XX |
| 2 | XX (XX.X%) | XX (XX.X%) | XX (XX:X%) |
| က | XX (XX: X%) | XX (XX.X%) | XX (XX.X%) |
| 4 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 2 | XX (XX: X%) | (%X:X%) XX | (%X:X%)<br>XX |
| 9 | XX (XX.X%) | (%X:X%) XX | (%X:X%) XX |
| 7 | XX (XX.X%) | XX (XX.X%) | XX (XX:X%) |
| 8 | XX (XX.X%) | (%X:X%) XX | (%X:X%)<br>XX |
| თ | XX (XX: X%) | (%X:X%) XX | (%X:X%) |
| 10 | (%X:X%) | XX (XX.X%) | XX (XX.X%) |

Abbreviations: BSA = body surface area; IGA = investigator global assessment; WI-NRS = Worst Itch – Numeric Rating Scale. Note: Percentages are n/Number of subjects in the Safety population within treatment received and overall\*100. [1] Only captured for female subjects; percentages are based on the number of female subjects in the Safety population. [2] The % BSA affected by seborrheic dermaitiis. [3] The WI-NRS will be determined by asking the subject's assessment of worst itch over the past 24 hours. The scale is from 0 to 10, which ranges from "no itch" to "worst imaginable itch". Reference Listings: 16.2.6.1, 16.2.6.1, 16.2.6.2, 16.2.6.5, 16.2.6.7, 16.2.9.1, 16.2.9.4.2.

Statistical Analysis Plan, Sponsor Arcutis Biotherapeutics, Inc. Protocol Number ARQ-154-203 PCN Number ARCU210100



Table 14.1.2.2 Summary of Demographics and Baseline Characteristics mITT Population

(Same shell as Table 14.1.2.1; subjects are summarized by planned treatment, not treatment received; Update Note: footnote as Percentages are n/Number of subjects in the mITT population within planned treatment and overall\*100.)





Table 14.1.3
Previous Treatment History of Seborrheic Dermatitis
Safety Population

| Category | Roflumilast Foam 0.3% | Vehicle<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|
| Inadequate Response. Intolerance or | (,,,,,,) | | (,,,,,) |
| Contraindication to | | | |
| Topical Corticosteroids | XX (XX:X%) | XX (XX.X%) | XX (XX: X%) |
| Topical Antifungals | (%X:XX) XX | XX (XX.X%) | (%X:X%) XX |
| Subjects have Facial Involvement | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Note: Percentages are n/Number of subjects in the Safety population within treatment received and overall\*100. Subjects with a response of "Yes" are summarized. Reference Listing: 16.2.4.2



Table 14.1.4 Summary of Protocol Deviations Safety Population

**premier** research

| Category | Roflumilast Foam 0.3% (N=XX) | Vehicle<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|
| Subjects with Any Protocol Deviations | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Subjects with Major Protocol Deviations XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) |

Note: Percentages are n/Number of subjects in the Safety population within treatment received and overall\*100. Only major protocol deviations are presented. Subjects with any protocol deviations row can include counts from major and minor deviations. Subjects with one or more deviations within a type of protocol deviation were counted only once. Protocol Deviations were collected throughout the

Reference Listing: 16.2.2.2

Programming note: the structure of this table may change depending on the information in the protocol deviations file.



Table 14.1.5 Summary of Prior Medications by ATC Class Level 4 and Preferred Term Safety Population

| | Roflumilast Foam | | |
|---|---|---|---|
| ATC Class Level 4 | 0.3% | Vehicle | Overall |
| Preferred Term | (N=XX) | (N=XX) | (N=XX) |
| Subjects with at least 1 Prior Medication | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| ATC Class 1 | (%X:X%) | (%X:X%) | (XX.X%) |
| Preferred Term 1 | XX (XX: X%) | (%X:XX) XX | (XX.X%) |
| Preferred Term 2 | XX (XX: X%) | (%X:X%) | XX (XX.X%) |
| Preferred Term 3 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| ATC Class 2 | (%X:X%) | (XX:X%) | (%X:X%) |
| Preferred Term 1 | XX (XX: X%) | (%X:XX) XX | (%X:X%) |
| Preferred Term 2 | (%X:X%) XX | (%X:XX) XX | (%X:X%) XX |
| Preferred Term 3 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Abbreviations: ATC = Anatomic Therapeutic Chemical; PT = preferred term; WHO-DDE = World Health Organization-Drug Dictionary

Note: Percentages are n/Number of subjects in the Safety population within treatment received and overall\*100. Medications were coded using WHO-DDE Global B3 version September 2019. Prior medications are all medications that were started before the application of study drug. Medications are displayed by alphabetical order of ATC Level 4 classification, then descending frequency of PT within ATC, and then alphabetically by PT. Subjects were counted only once for each ATC and PT.

Reference Listing: 16.2.9.7

Programming note: ATC & PT text should be presented as is from the dataset.

**premier** research

Table 14.1.6 Summary of Study Drug Exposure Safety Population

| Variable<br>Statistic / Category | Roflumilast Foam<br>0.3%<br>(N=XX) | Vehicle<br>(N=XX) |
|---|---|---|
| Total Number of IP Applications | | ; |
| n<br>Mean (SD) | XX | (XX.XX)<br>XX.XX |
| wedan<br>Min, Max | XX,XX | X, XX |
| Total Weight (g)of IP Applied [1]<br>n | × | × |
| Mean (SD)<br>Median | XX.X (XX.XX)<br>XX.X | XX.X (XX.XX)<br>XX.X |
| Min, Max | XX, XX | X, X |
| Compliance [2] >100% | XX (XX.X%) | (%X:XX) XX |
| ≥ 80% - ≤100% | (%X:X%) | (%X:XX) XX |
| > 80% | XX (XX.X%) | XX (XX.X%) |
| > 3 Consecutive Missed Doses | XX (XX.X%) | (%X:XX) XX |
| Compliant [3] | XX (XX.X%) | XX (XX.X%) |

Abbreviation: IP = investigational product. Note: n is the number of subjects in the Note: n is the number of subjects in the Safety Population. Percentages are n/Number of subjects in the

Safety Population within treatment received\*100. [1] Total weight from the dispensed can weight. [2] Compliance is calculated based on number of applications divided by the expected number of IP

applications for each subject\*100.
[3] A subject is considered compliant if the subject applies at least 80% of the expected applications during the IP application period and does not miss more than 3 consecutive doses.

Reference Listings: 16.2.5.1, 16.2.5.2, 16.2.5.4



Table 14.2.1.1 Summary and Change from Baseline in Investigator Global Assessment (IGA) Grades by Study Visit – Observed Data mITT Population

| Study Visit | Roflumilast Foam 0.3% (N=XX) | Foam 0.3%<br>XX) | Vehicle (N=XX) | icle<br>XX) |
|---|---|---|---|---|
| Statistic | Observed | Change | Observed | Change |
| Baseline | | | | |
| L | × | | × | |
| Mean (SD) | XX.X (X.XX) | | XX.X (X.XX) | |
| Median | ××× | | ××× | |
| Min, Max | ××× | | ××× | |
| Q1, Q3 | XXX | | XXX | |
| Week 2 | | | | |
| _ | × | × | × | × |
| Mean (SD) | XX.X (X.XX) | XX.X (X.XX) | XX.X (X.XX) | XX:X (X:XX) |
| Median | ××× | ××× | ××× | ××× |
| Min, Max | ××× | ×××× | ××× | ××× |
| Q1, Q3 | XXX | XXX | XX.X | XXX |

## Repeat for Week 4, Week 8, Week 9.

Note: Subjects are summarized by planned treatment. IGA is a static qualitative evaluation of overall seborrheic dermatitis severity involving an ordinal scale with 5 severity grades (reported only in integers of 0 to 4) where 0 = Clear; 1 = Almost Clear; 2 = Mild; 3 = Moderate; 4 = Severe. Baseline is the last non-missing measurement taken on or before the day of first application of study drug. Change from baseline is calculated as result - baseline result. Week 9 summaries are provided only for the subjects that didn't rollover to the extension study.

Reference Listing: 16.2.6.1



Table 14.2.1.2

Summary and Change from Baseline in Investigator Global Assessment (IGA) Grades by Study Visit - Observed Data ITT Population

(Same shell as Table 14.2.1.1)

Summary and Change from Baseline in Investigator Global Assessment (IGA) Grades by Study Visit - Multiple Imputation

Table 14.2.1.3

mITT Population

(Same shell as Table 14.2.1.1; Programming note: update "Note:" portion of footnote to add in the following text just after "Note:": Separate multiple imputation steps were used for monotone and non-monotone missing data. For monotone missing pattern, predictive mean matching model will be used to impute missing value for a subject at particular visit having baseline IGA score, treatment group and investigational site as independent variables and study visit as dependent variable. For non-monotone missing IGA values, Markov-Chain Monte Carlo (MCMC) method will be used to impute the data at intermediate visits to make the missing data pattern into monotone before applying predictive mean matching multiple imputation algorithm. Subjects are summarized by planned treatment.)

Summary and Change from Baseline in Investigator Global Assessment (IGA) Grades by Study Visit – Multiple Imputation ITT Population Table 14.2.1.4

(Same shell as Table 14.2.1.1; Programming note: update "Note:" portion of footnote to add in the following text just after "Note:": Separate multiple imputation steps were used for monotone and non-monotone missing data. For monotone missing pattern, predictive mean matching model will be used to impute missing value for a subject at particular visit having baseline IGA score, treatment group and investigational site as independent variables and study visit as dependent variable. For non-monotone missing IGA values, Markov-Chain Monte Carlo (MCMC) method will be used to impute the data at intermediate visits to make the missing data pattern into monotone before applying predictive mean matching multiple imputation algorithm. Subjects are summarized by planned treatment.)

Summary of Investigator Global Assessment (IGA) Grades and Success by Study Visit - Observed Data Categorical Results mITT Population Table 14.2.1.5

| Study Visit<br>Category/Statistic | Roflumilast Foam 0.3%<br>(N=XX) | Vehicle<br>(N=XX) |
|---|---|---|
| Baseline | | |
| 0 = Clear | XX (XX.X%) | XX (XX.X%) |
| 1 = Almost Clear | XX (XX.X%) | XX (XX.X%) |
| 2 = Mild | XX (XX.X%) | XX (XX.X%) |
| 3 = Moderate | XX (XX.X%) | XX (XX.X%) |
| 4 = Severe | XX (XX.X%) | XX (XX.X%) |
| Week 2 | | |
| 0 = Clear | XX (XX.X%) | XX (XX.X%) |
| 1 = Almost Clear | XX (XX.X%) | (%X:X%) |
| 2 = Mild | (%X:X%) | (%X:X%) |
| 3 = Moderate | XX (XX.X%) | (%X:X%)<br>XX |
| 4 = Severe | XX (XX.X%) | XX (XX.X%) |
| IGA Success [1] | | |
| Yes | XX (XX.X%) | XX (XX.X%) |
| 90% CI [2] | (X.XX, X.XX) | (XXX, XXX) |
| 95% CI [2] | (X.XX, X.XX) | (XXX, XXX) |
| No | XX (XX.X%) | XX (XX.X%) |
| Odds Ratio (90% CI) [3]<br>Odds Ratio (95% CI) [3]<br>P value [3] | XXX (XXX, XXX)<br>XXX (XXX, XXX)<br>XXXXX | |

Repeat for all Week 4, Week 8, and Week 9.

Abbreviations: CI = confidence interval; IGA = investigator global assessment.

Note: Percentages are n/Number of subjects in the mITT population within planned treatment at each visit\*100. Baseline is the last non-missing measurement taken on or before the day of first application of study drug. Week 9 summaries are provided only for the subjects that didn't rollover to the extension study. [1] IGA success ("Yes") is defined as an IGA score of "Clear" or "Almost Clear" plus a ≥2-grade improvement

from baseline; "No" otherwise.
[2] 90% and 95% CI for "Yes" are obtained using Wilson method.
[3] The odds ratio, 90% CI, 95% CI, and P value are obtained from Cochran Mantel Haenszel test (stratified by study site and baseline IGA) comparing Roflumilast Foam 0.3% to Vehicle.

Reference Listing: 16.2.6.1



Table 14.2.1.6
Summary of Investigator Global Assessment (IGA) Grades and Success by Study Visit – Observed Data
Categorical Results
ITT Population

(Same shell as Table 14.2.1.5; update the first line in "Note:" as "Percentages are n/Number of subjects in the ITT population within planned treatment\*100.")

Table 14.2.1.7
Summary of Investigator Global Assessment (IGA) Grades and Success by Study Visit – Multiple Imputation
Categorical Results
mITT Population

subject at particular visit having baseline IGA score, treatment group and investigational site as independent variables and study visit as dependent variable. For non-monotone missing IGA values, Markov-Chain Monte Carlo (MCMC) method will be used to impute the data at intermediate visits to make the missing data pattern into monotone before applying imputation steps were used for monotone and non-monotone missing data. For monotone missing pattern, predictive mean matching model will be used to impute missing value for a "Note:". The grades and success scores were obtained from observed dataset. The odds ratio and p values were summarized using multiple imputation dataset. Separate multiple (Same shell as Table 14.2.1.5; The grades and success scores will be based on observed data; update "Note:" portion of footnote to add in the following text just after predictive mean matching multiple imputation algorithm.)



Summary of Investigator Global Assessment (IGA) Grades and Success by Study Visit – Multiple Imputation Categorical Results ITT Population Table 14.2.1.8

subject at particular visit having baseline IGA score, treatment group and investigational site as independent variables and study visit as dependent variable. For non-monotone missing IGA values, Markov-Chain Monte Carlo (MCMC) method will be used to impute the data at intermediate visits to make the missing data pattern into monotone before applying predictive mean matching multiple imputation algorithm. Percentages are n/Number of subjects in the ITT population within planned treatment at each visit\*100.) "Note:": The grades and success scores were obtained from observed dataset. The odds ratio and p values were summarized using multiple imputation dataset. Separate multiple imputation steps were used for monotone and non-monotone missing data. For monotone missing pattern, predictive mean matching model will be used to impute missing value for a (Same shell as Table 14.2.1.5; The grades and success scores will be based on observed data; update "Note:" portion of footnote to add in the following text just after



Summary of Investigator Global Assessment (IGA) Grades and Success by Study Visit - Observed Data Tabulation of Fitted Point Estimates from Generalized Estimating Equations for Binary Response mITT Population Table 14.2.1.9

| Study Visit | Roflumila | Roflumilast Foam 0.3% (N=XX) | | Vehicle<br>(N=XX) | Treatment | Treatment Difference (Roflumilast Foam 0.3% vs Vehicle) [3] | st Foam 0.3% vs Veh | licle) [3] |
|---|---|---|---|---|---|---|---|---|
| Category/Statistic | n [1] | Responder [2] | n [1] | Responder [2] | Odds Ratio | 90% CI for OR | 95% CI for OR | P value |
| Week 2 | × | %X:XX | × | %X:XX | XXX | (XX.XX, XX.XX) | (XX.XX, XX.XX) | XXXXX |
| Week 4 | × | %X:XX | × | %X:XX | × | (XX.XX, XX.XX) | (XX.XX, XX.XX) | X.XXX |
| Week 8 | × | %X:XX | × | %X:XX | × | (XX.XX, XX.XX) | (XX.XX, XX.XX) | X.XXX |
| Week 9 | × | %X:XX | × | %X:XX | × | (XX.XX, XX.XX) | (XX.XX, XX.XX) | X.XXX |

Abbreviations: CI = Confidence interval; IGA = investigator global assessment; OR = odds ratio.

Note: Percentages are n/Number of subjects in the mITT population within planned treatment at each visit\*100. Baseline is the last non-missing measurement taken on or before the day of first application of study drug. Week 9 summaries are provided only for the subjects that didn't rollover to the extension study.

[1] Number of subjects at each visit.

success as the dependent variable and treatment, site, baseline IGA score, and visit as the independent variables. An unstructured correlation matrix was used to model [2] Number of subjects with an IGA score of "Clear" or "Almost Clear" plus a ≥2-grade improvement from baseline. [3] Estimates for odds ratio, 90% CI for odds ratio, 95% CI for odds ratio, and P value are from a generalized estimating equations for binary response model, with IGA the within subject correlation. In case of convergence issues, other covariance structures will be used including Toeplitz, compound symmetry or Autoregressive (1) (AR[1]) covariance structure will be used, following this sequence until convergence is achieved. The odds ratio is the estimate of the odds of having IGA response for subjects treated with Roflumilast Foam 0.3% relative to that for subjects treated with vehicle. Reference Listing: 16.2.6.1 



Table 14.2.1.10
Summary of Investigator Global Assessment (IGA) Grades and Success by Study Visit – Observed Data
Tabulation of Fitted Point Estimates from Generalized Estimating Equations for Binary Response
ITT Population

(Programming note: Same as table shell 14.2.1.9; update first line of note footnote to "Percentages are n/Number of subjects in the ITT population within planned treatment at each visit\*100.")



Summary of Investigator Global Assessment (IGA) – 2-grade Improvement from Baseline – Observed Data mITT Population Table 14.2.1.11

| Study Visit | Roflumilast Foam 0.3% | Vehicle |
|---|---|---|
| Category/Statistic | (X=X) | (XX=N) |
| Week 2 | | |
| IGA Success [1] | | |
| Yes | XX (XX: X%) | XX (XX: X%) |
| 90% CI [2] | (X.XX, X.XX) | (X, XX, X, XX) |
| 95% CI [2] | (X.XX, X.XX) | (X, X, X, X, X) |
| No | XX (XX.X%) | (%X.XX) XX |
| Odds Ratio (90% CI) [3]<br>Odds Ratio (95% CI) [3]<br>P value [3] | XXX (X.XX, X.XX)<br>XXX (X.XX, X.XX)<br>X.XXXX | |

# Repeat for all Week 4, Week 8, and Week 9.

Abbreviations: CI = confidence interval; IGA = investigator global assessment.

Note: Percentages are n/Number of subjects in the mTT population within planned treatment\*100. Baseline is the last non-missing measurement taken on or before the day of first application of study drug. Week 9

summaries are provided only for the subjects that didn't rollover to the extension study.

[1] IGA success ("Yes") is defined as a 2-grade improvement from baseline; "No" otherwise.

[2] 90% and 95% CI for "Yes" are obtained using Wilson method.

[3] The odds ratio, 90% CI, 95% CI, and P value are obtained from Cochran Mantel Haenszel test (stratified by study site and baseline IGA) comparing Roflumilast Foam 0.3% to Vehicle.

Reference Listing: 16.2.6.1

Statistical Analysis Plan, Sponsor Arcutis, Inc. Protocol Number ARQ-154-203 PCN Number ARCU0100



Summary of Investigator Global Assessment (IGA) – 2-grade Improvement from Baseline ITT Population Table 14.2.1.12

(Programming note: Same as table shell 14.2.1.11; update first line of note footnote to "Percentages are n/Number of subjects in the ITT population within planned treatment at each visit\*100.")



| | | % Change | | | | | | | | | × | XX.X (X.XX) | ××× | ××× | ××× | XXXXX | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Vehicle<br>(N=XX) | i | Change | | | | | | | | | × | XX.X (X.XX) | ××× | ×××× | ××× | XXXXX | |
| | | Observed | | × | XX.X (X.XX) | ××× | ××× | ××× | X.XXXX | | × | XX.X (X.XX) | XX.Xs | ××× | ××× | X.XXXX | k 8, Week 9. |
| | | % Change | | | | | | | | | × | XX.X (X.XX) | ××× | ××× | ××× | X.XXXX | Repeat for Week 4, Wee |
| Roflumilast Foam 0.3% | (XX=N) | Change | | | | | | | | | | | | | | XXXXXX | |
| | | Observed | | × | XX.X (X.XX) | ××× | ×,× | ××× | X.XXXX | | × | XX.X (X.XX) | ××× | ×××× | ××× | X.XXX.X | |
| Table 14.2.2.1 Summary and Change from Baseline in Overall Assessment of Erythema – Severity Grades by Study Visit Wilcoxon Test mITT Population | Study Visit | Statistic | Baseline | _ | Mean (SD) | Median | Min, Max | Q1, Q3 | P value [1] | Week 2 | ٦ | Mean (SD) | Median | Min, Max | Q1. Q3 | P value [1] | |

Note: Subjects are summarized by planned treatment. Overall Assessment of Erythema is a static qualitative evaluation involving an ordinal scale with 4 severity grades (reported only in integers of 0 to 3) where 0 = None; 1 = Mild; 2 = Moderate; 3 = Severe. Baseline is the last non-missing measurement taken on or before the day of first application of study drug. Change from baseline is calculated as result - baseline result. Percent change from baseline is calculated as (change from baseline)\*100.
[1] P value was obtained from an exact Wilcoxon rank sum test, comparing Roflumilast Foam 0.3% with Vehicle.
Reference Listing: 16.2.6.2



Summary of Overall Assessment of Erythema – Severity Grades and Success by Study Visit Categorical Results mITT Population Table 14.2.2.2

| 3% Vehicle (N=XX) | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | XX (XX. X%)<br>(X.XX, X.XX)<br>(X.XX, X.XX)<br>XX (XX. X%) | |
|---|---|---|---|---|
| Roflumilast Foam 0.3% (N=XX) | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>(X.XX, X.XX)<br>(X.XX, X.XX)<br>XX (XX.XX) | XXX (XXX, XXX)<br>XXX (XXX, XXX)<br>XXXXX |
| Study Visit<br>Category/Statistic | Baseline<br>0 = None<br>1 = Mild<br>2 = Moderate<br>3 = Severe | Week 2<br>0 = None<br>1 = Mild<br>2 = Moderate<br>3 = Severe | Erythema Success [1] Yes 90% CI [2] 95% CI [2] No | Odds Ratio (90% CI) [3]<br>Odds Ratio (95% CI) [3]<br>P value [3] |

Repeat for Week 4, Week 8, and Week 9.

Abbreviations: CI = confidence interval; IGA = investigator global assessment.

Note: Percentages are n/Number of subjects in the mITT population within planned treatment\*100. Baseline is the last non-missing measurement taken on or before the day of first application of study drug. Week 9 summaries are provided only for the subjects that didn't rollover to the extension study. [1] Erythema success ("Yes") is defined as an Erythema score of "0" or "1" plus a ≥2-grade improvement

from baseline; "No" otherwise.
[2] 90% and 95% CI for "Yes" are obtained using Wilson method.
[3] The odds ratio, 90% CI, 95% CI, and P value are obtained from Cochran Mantel Haenszel test (stratified by study site and baseline IGA) comparing Roflumilast Foam 0.3% to Vehicle.
Reference Listing: 16.2.6.2



Table 14.2.2.3

Summary and Change from Baseline in Overall Assessment of Erythema – Severity Grades by Study Visit Wilcoxon Test ITT Population

(Programming note: Same as table 14.2.2.1; Update any instances of mITT to ITT in the footnotes.)

Table 14.2.2.4
Summary of Overall Assessment of Erythema – Severity Grades and Success by Study Visit
Categorical Results
ITT Population

(Programming note: Same as table 14.2.2.2. Update the first line of footnotes to "Note: Percentages are n/Number of subjects in the ITT population within planned treatment" 100.")



Summary of Overall Assessment of Erythema – Score of 0 or 1 and Score of 0 by Study Visit Categorical Results mITT Population Table 14.2.2.5

| #5077777 | | |
|---|---|---|
| Study Visit<br>Category/Statistic | Roflumilast Foam 0.3%<br>(N=XX) | Vehicle<br>(N=XX) |
| Week 2 | | |
| Erythema Score of 0 or 1 [1] | | |
| Yes | (%X:X%)<br>XX | XX (XX:X%) |
| 90% CI [2] | (X.XX, X.XX) | |
| 95% CI [2] | (XXX, XXX) | |
| No. | XX (XX.X%) | XX (XX.X%) |
| Odds Ratio (90% CI) [3]<br>Odds Ratio (95% CI) [3] | X.XX (X.XX, X.XX)<br>X.XX (X.XX, X.XX) | |
| P value [3] | X.XXXX | |
| Erythema Success Score of 0 [4] | | |
| Yes | XX (XX.X%) | (%X:XX) XX |
| 90% CI [2] | (X.XX, X.XX) | (X.XX, X.XX) |
| 95% CI [2] | (X.XX, X.XX) | (X.XX, X.XX) |
| OZ. | XX (XX.X%) | XX (XX.X%) |
| Odds Ratio (90% CI) [3] | X.XX (X.XX, X.XX) | |
| Odds Ratio (95% CI) [3] | X.XX (X.XX, X.XX) | |
| r value [3] | V.VVV. | |

Repeat for Week 4, Week 8, and Week 9.

Abbreviations: CI = confidence interval; IGA = investigator global assessment.

Note: Percentages are n/Number of subjects in the mTT population within planned treatment\*100. Baseline is the last non-missing measurement taken on or before the day of first application of study drug. Week 9

summaries are provided only for the subjects that didn't rollover to the extension study.

[1] Erythema ("Yes") is defined as an Erythema score of "O" or "1"; "No" otherwise.

[2] 90% and 95% CI for "Yes" are obtained using Wilson method for each Success test separately.

[3] The odds ratio, 90% CI, 95% CI, and P value are obtained from Cochran Mantel Haenszel test (stratified by study site and baseline IGA) comparing Roflumilast Foam 0.3% to Vehicle.

[4] Erythema success ("Yes") is defined as an Erythema score of "O"; "No" otherwise.





Table 14.2.2.6
Summary of Overall Assessment of Erythema – Success Score of 0 or 1 and Success Score of 0 by Study Visit
Categorical Results
ITT Population

(Programming note: Same as table 14.2.2.5. Replace any instances of mITT with ITT)



Table 14.2.3.1 Summary and Change from Baseline in Overall Assessment of Scaling – Severity Grades by Study Visit mITT Population

qualitative evaluation involving an ordinal scale with 4 severity grades (reported only in integers of 0 to 3) where 0 = None; 1 = Mild; 2 = Moderate; 3 = Severe. Baseline is the last non-missing measurement taken on or before the day of first application of study drug. Change from baseline is calculated as result - baseline result. Percent change from baseline is calculated as (change from baseline)\*100."; update reference listing to 16.2.6.3) (Programming note: Same as table 14.2.2.1. Update the footnotes to "Note: Subjects are summarized by planned treatment. Overall Assessment of Scaling is a static

Table 14.2.3.2
Summary of Overall Assessment of Scaling – Severity Grades and Success by Study Visit
Categorical Results
mITT Population

(Programming note: Same as table 14.2.2.2. Change Reference Listing to 16.2.6.3. Update any instances of Erythema to Scaling)

Table 14.2.3.3 Summary and Change from Baseline in Overall Assessment of Scaling – Severity Grades by Study Visit ITT Population

qualitative evaluation involving an ordinal scale with 4 severity grades (reported only in integers of 0 to 3) where 0 = None; 1 = Mild; 2 = Moderate; 3 = Severe. Baseline is the last non-missing measurement taken before the first application of study drug. Change from baseline is calculated as result - baseline result. Percent change from (Programming note: Same as table 14.2.2.1. Update the footnotes to "Note: Subjects are summarized by planned treatment. Overall Assessment of Scaling is a static baseline is calculated as (change from baseline/baseline)\*100."; update reference listing to 16.2.6.3)

Table 14.2.3.4
Summary of Overall Assessment of Scaling – Severity Grades and Success by Study Visit
Categorical Results
ITT Population

(Programming note: Same as table 14.2.2.2. Update the first line of footnotes to "Note: Percentages are n/Number of subjects in the ITT population within planned treatment\*100". Change Reference Listing to 16.2.6.3. Update any instances of Erythema to Scaling)



Summary of Overall Assessment of Scaling – Success Score of 0 or 1 by Study Visit Categorical Results mITT Population Table 14.2.3.5

(Programming note: Same as 14.2.2.5. Update reference listing to 16.2.6.3; Change any instance of Erythema to Scaling)

Summary of Overall Assessment of Scaling – Success Score of 0 or 1 by Study Visit Categorical Results ITT Population Table 14.2.3.6

(Programming note: Same as 14.2.2.5. Update reference listing to 16.2.6.3; Change any instance of Erythema to Scaling and replace mITT with ITT in the footnotes)




Summary and Change from Baseline in Worst Itch – Numeric Rating Scale (WI-NRS) Pruritus Score by Study Visit mITT Population Table 14.2.4.1

| | % Change | | | | | | | | × | XX.X (X.XX) | ×× | X, X | XXX |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Vehicle<br>(N=XX) | Change | | | | | | | | × | XX.X (X.XX) | ××× | ×××× | ××× |
| | Observed | | × | (XX:X) X:XX | ××× | ××× | XX.X | | × | XX.X (X.XX) | XX.Xs | ×××× | XX.X |
| | % Change | | | | | | | | × | XX.X (X.XX) | ×× | ××× | ×:× |
| Roflumilast Foam 0.3% (N=XX) | Change | | | | | | | | × | XX.X (X.XX) | ××× | ××× | ×:× |
| | Observed | | × | XX.X (X.XX) | ××× | ×××× | X.X | | × | XX.X (X.XX) | ××× | ×××× | X.XX |
| Study Visit | Statistic | Baseline | Ц | Mean (SD) | Median | Min, Max | Q1, Q3 | Week 2 | Г | Mean (SD) | Median | Min, Max | Q1, Q3 |

Repeat for Week 4, Week 8, Week 9.

Note: Subjects are summarized by planned treatment. The WI-NRS will be determined by asking the subject's assessment of worst itch over the past 24 hours. The scale is from 0 to 10, which ranges from "no itch" to "worst imaginable itch". Baseline is the last non-missing measurement taken on or before the day of first application of study drug. Change from baseline is calculated as result - baseline result. Percent change from baseline is calculated as result - baseline result. Reference Listing: 16.2.6.4



Summary and Change from Baseline in Worst Itch – Numeric Rating Scale (WI-NRS) Pruritus Score by Study Visit ITT Population Table 14.2.4.2

(Programming note: Same as table 14.2.4.1. Change Reference Listing to 16.2.6.4. Update the footnotes as "Note: Subjects are summarized by planned treatment. The WI-NRS will be determined by asking the subject's assessment of worst itch over the past 24 hours. The scale is from 0 to 10, which ranges from "no itch" to "worst imaginable itch". Baseline is the last non-missing measurement taken on or before the day of first application of study drug. Change from baseline is calculated as result - baseline result. Percent change from baseline is calculated as (change from baseline)\*100.




Worst ltch – Numeric Rating Scale (WI-NRS) Pruritus Score Success by Study Visit mITT Population, Subjects with WI-NRS Pruritus Score ≥4 at Baseline (PRU4 Population) Table 14.2.4.3

| Study Visit | Roflumilast Foam 0.3% | Vehicle |
|---|---|---|
| Category/statistic | (N=XX) | (N=XX) |
| Week 2 | | |
| WI-NRS Success [1] | | |
| Yes | (%X:X%) | (%X:X%) |
| 90% CI [2] | (X.XX, X.XX) | (X, XX, X, XX) |
| 95% CI [2] | (X.XX, X.XX) | (XXX, XXX) |
| No | XX (XX.X%) | (%X.X%) XX |
| Odds Ratio (90% CI) [3]<br>Odds Ratio (95% CI) [3] | X.XX (X.XX, X.XX)<br>X.XX (X.XX, X.XX) | |
| P value [3] | XXXXX | |

Repeat for all Week 4, and Week 8.

Abbreviations: CI = confidence interval; IGA = investigator global assessment.

Note: Percentages are n/Number of subjects in the mITT PRU4 population within planned treatment\*100.

Baseline is the last non-missing measurement taken on or before the day of first application of study drug.

[1] WI-NRS success ("Yes") is defined as an achievement of a ≥4-point improvement from baseline score of ≥4; "No" otherwise.
[2] 90% and 95% CI for "Yes" are obtained using Wilson method.
[3] The odds ratio, 90% CI, 95% CI, and P value are obtained from Cochran Mantel Haenszel test (stratified by study site and baseline IGA) comparing ARQ-154 to Vehicle.
Reference Listing: 16.2.6.4


Table 14.2.4.4
Worst Itch – Numeric Rating Scale (WI-NRS) Pruritus Score Success by Study Visit mITT Population, Subjects with WI-NRS Pruritus Score ≥2 at Baseline (PRU2 Population)

(Programming note: Same as table 14.2.4.3. Update any instances of PRU4 to PRU2. Update footnotes to "Percentages are n/Number of subjects in the mITT PRU2 population within planned treatment\*100." Update footnote [1] as "WI-NRS success ("Yes") is defined as an achievement of a ≥2-point improvement from baseline score of ≥2; "No" otherwise.)

Table 14.2.4.5
Worst Itch – Numeric Rating Scale (WI-NRS) Pruritus Score Success by Study Visit ITT Population, Subjects with WI-NRS Pruritus Score ≥4 at Baseline (PRU4 Population)

(Programming note: Same as table 14.2.4.3. Update any instances of mITT with ITT)

Table 14.2.4.6
Worst Itch – Numeric Rating Scale (WI-NRS) Pruritus Score Success by Study Visit ITT Population, Subjects with WI-NRS Pruritus Score ≥2 at Baseline (PRU2 Population)

(Programming note: Same as table 14.2.4.3. Update any instances of PRU4 to PRU2. Update footnotes to "Percentages are n/Number of subjects in the ITT PRU2 population within planned treatment"100." Update footnote [1] as "WI-NRS success ("Yes") is defined as an achievement of a ≥2-point improvement from baseline score of ≥2; "No" otherwise.)



Summary of Worst Itch – Numeric Rating Scale (WI-NRS) by Study Visit - ANCOVA mITT Population Table 14.2.4.7

| Study Visit<br>Statistic [1] | ARQ-154 0.3%<br>(N=XX) | Vehicle<br>(N=XX) |
|---|---|---|
| Week 2 | × | × |
| LS Mean Change from Baseline (SE) | (X:XX (X:XXX) | X.XX (X.XXX)<br>X. X. X. X.X) |
| (95% CI for LS Mean Change from Baseline) P value for LS Mean Change from Baseline) [2] | (XXX, XXX)<br>XXXXX<br>XXXXX | (X.XX, X.XX) |
| LS Mean Difference from Vehicle (SE) (90% CI for Difference from Vehicle) (95% CI for Difference from Vehicle) P value for Difference from Vehicle [3] | (XXX, XXX)<br>XXX (XXXX)<br>XXXX XXXX | |

Repeat for Week 4, Week 8, and Week 9.

Abbreviations: CI = confidence interval; IGA = investigator global assessment; LS = least-squares; SE = standard error.

Note: Subjects are summarized by planned treatment. Baseline is the last non-missing measurement taken on or before the day of first application of study drug. The WI-NRS will be determined by asking the subject's assessment of worst itch over the past 24 hours. The scale is from 0 to 10, which ranges from "no itch" to "worst imaginable itch.

[1] Estimates for LS means (change from baseline and difference from vehicle [i.e., change from baseline for Roflumilast Foam 0.3% minus change from baseline for vehicle]) and accompanying 90%, 95% CIs, and P values are from an analysis of covariance (ANCOVA) with treatment, study site, baseline IGA, and baseline WI-NRS score as independent variables.
[2] P value for testing change from baseline is zero.
[3] P value for testing difference (Roflumilast Foam 0.3% minus Vehicle) in change from baseline from is zero.
Reference Listings: 16.2.6.1, 16.2.6.4





Table 14.2.4.8 Summary of Worst Itch – Numeric Rating Scale (WI-NRS) by Study Visit - ANCOVA ITT Population

(Programming note: Same as table 14.2.4.7; Update any instances of mITT into ITT)



Table 14.2.4.9 Summary of Worst Itch - Numeric Rating Scale (WI-NRS) by Study Visit - Categorical Scale mITT Population

| Study Visit | Roflumilast Foam 0.3% | Vehicle |
|-------------|-----------------------|------------|
| Category | (N=XX) | (N=XX) |
| Baseline | | |
| 0 | XX (XX.X%) | XX (XX.X%) |
| _ | XX (XX. X%) | (%X:XX) XX |
| 2 | XX (XX.X%) | (%X:X%) |
| က | XX (XX. X%) | (%X:XX) XX |
| 4 | XX (XX.X%) | (%X:X%) |
| 5 | (%X:X%) | (%X:XX) XX |
| 9 | (%X:X%) | (%X:XX) XX |
| 7 | (%X:X%) | (%X:XX) XX |
| 8 | (%X:X%) | (%X:XX) XX |
| 0 | (%X:X%) | (%X:XX) XX |
| 10 | (%X:X%) | (%X:X%) XX |

Repeat for Week 2, Week 4, and Week 8.

Note: Percentages are n/Number of subjects in the mITT population within planned treatment\*100. The WINS will be determined by asking the subject's assessment of worst itch over the past 24 hours. The scale is from 0 to 10, which ranges from "no itch" to "worst imaginable itch. Baseline is the last non-missing measurement taken on or before the day of first application of study drug.

Reference Listing: 16.2.6.4





Table 14.2.4.10 Summary of Worst Itch - Numeric Rating Scale (WI-NRS) by Study Visit - Categorical Scale ITT Population

(Programming note: Same as table 14.2.4.9; Update any instances of mITT into ITT)



Change from Baseline in Scalpdex by Study Visit mITT Population Table 14.2.5.1

| Study Visit<br>Scale | | Roflumilast Foam 0.3% (N=XX) | | | Vehicle<br>(N=XX) | | 1 |
|---|---|---|---|---|---|---|---|
| Statistic | Observed | Change | % Change | Observed | Change | % Change | 1 |
| Baseline | | | | | | | |
| Emotions [1] | | | | | | | |
| u | × | | | × | | | |
| Mean (SD) | XX.X (X.XX) | | | XX.X (X.XX) | | | |
| Median | ××× | | | ××× | | | |
| Min, Max | ××× | | | ××× | | | |
| 01, 03 | ××× | | | X.XX | | | |
| Symptoms [2] | | | | | | | |
| | × | | | × | | | |
| Mean (SD) | XX.X (X.XX) | | | XX:X (X:XX) | | | |
| Median | XXX | | | XXX | | | |
| Min, Max | ××× | | | ××× | | | |
| Q1, Q3 | XXX | | | XXX | | | |
| Functioning [3] | | | | | | | |
| L | × | | | × | | | |
| Mean (SD) | XX.X (X.XX) | | | XX.X (X.XX) | | | |
| Median | XXX | | | ××× | | | |
| Min, Max | ××× | | | ×,× | | | |
| Q1, Q3 | ××× | | | ×:× | | | |
| | | Repeat for Total Score | [4] and continue the sar | Repeat for Total Score [4] and continue the same for Week 2, Week 4 and Week 8. | Week 8. | | |

Note: Subjects are summarized by planned treatment. Baseline is the last non-missing measurement taken before the first application of study drug. Change from baseline is calculated as result - baseline result. Percent change from baseline is calculated as result - baseline result. Percent change from baseline is calculated as result as calculated as result. Percent change from baseline is calculated as average of the (QZ, Q4, Q5, Q6, Q7, Q9, Q10, Q11, Q12, Q14, Q16, Q17, Q19, Q20, and Q22; Q19 will be reverse scored i.e., 1 = 100; 2 = 75; 3 = 50; 4 = 25; 5 = 0) after scale transformation as noted above.

[2] Symptoms scale is calculated as average of the (Q1, Q3, and Q8) after scale transformation as noted above.
[3] Functioning scale is calculated as average of the (Q1, Q3, and Q8) after scale transformation as noted above.
[4] Total score is calculated as mean of all 23 questions. Q19 will be reverse scored as mentioned in [1].

Protocol Number ARQ-154-203 PCN Number ARCU0100 Statistical Analysis Plan, Sponsor Arcutis, Inc.



Summary of Scalpdex by Study Visit - ANCOVA mITT Population Table 14.2.5.2

| Study Visit<br>Scale [1]<br>Statistic [2] | Roflumilast Foam 0.3%<br>(N=XX) | Vehicle<br>(N=XX) |
|---|---|---|
| Week 2<br>Emotions | | |
| n<br>I S Maca Change from Bootling (SE) | ×× >> > | ×××× |
| LS Mearl Criarige IIOII Basellire (SE)<br>(90% Cl for LS Mean Change from Baseline) | (X,XX, X,XX) | (X,XX, X,XX)<br>(X,XX, X,XX) |
| (95% CI for LS Mean Change from Baseline) | (X.XX, X.XX) | (X.XX, X.XX) |
| P value for LS Mean Change from Baseline) [3] | XXXXX | |
| LS Mean Difference from Vehicle (SE) | (X.XX, X.XX) | |
| (90% CI for Difference from Vehicle) | X.XX (X.XXX) | |
| (95% CI for Difference from Vehicle) P value for Difference from Vehicle [4] | X.XXXX)<br>X.XXXXX | |

# Continue for Symptoms, Functioning, Total Score; Repeat for Week 4, and Week 8.

Abbreviations: CI = confidence interval; IGA = investigator global assessment; LS = least-squares; SE = standard error.

Note: Subjects are summarized by planned treatment. Baseline is the last non-missing measurement taken on or before the day of first application of study drug. Scalpdex questionnaire consists of 23 questions which is divided into 3 scales. Scalpdex is rated on a 1 to 5 scale which is transformed into 0 to 100 scale as follows; 1 = 0; 2 = 25; 3 = 50; 4 = 75; 5 = 100

[1] Emotions scale is calculated as average of the (Q2, Q4, Q5, Q6, Q7, Q9, Q10, Q11, Q12, Q14, Q16, Q17, Q19, Q20, and Q22; Q19 will be reverse scored i.e., 1 = 100; 2 = 75; 3 = 50, 4 = 25; 5 = 0) after scale transformation as noted above.

Symptoms scale is calculated as average of the (Q1, Q3, and Q8) after scale transformation as noted above. Functioning scale is calculated as average of (Q13, Q15, Q18, Q21, and Q23) after scale transformation as noted above. Total score is calculated as mean of all the 23 questions. Q18 will be reverse scored as mentioned above.

baseline for vehicle]) and accompanying 90%, 95% Cls, and P values are from an analysis of covariance (ANCOVA) with treatment, study site, [2] Estimates for LS means (change from baseline and difference from vehicle [i.e., change from baseline for ARQ-154 minus change from baseline IGA, and baseline Scalpdex scale score as independent variables.

[3] P value for testing change from baseline is zero.

[4] P value for testing difference (ARQ-154 minus Vehicle) in change from baseline from is zero. Reference Listings: 16.2.6.1, 16.2.6.5



Table 14.2.5.3 Change from Baseline in Scalpdex by Study Visit ITT Population

(Programming note: Same as table 14.2.5.1; Replace any instances of mITT with ITT)

Table 14.2.5.4 Summary of Scalpdex by Study Visit - ANCOVA ITT Population

(Programming note: Same as table 14.2.5.2; Replace any instances of mITT with ITT)



Table 14.2.5.5 Categorical Summary of Individual Responses by Study Visit – Scalpdex Questionnaire mITT Population

| | | Roflumik | Roflumilast Foam 0.3% (N=XX | N=XX) | | | | Vehicle (N=XX) | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Question [1]<br>Study Visit | Never | Rarely | Sometimes | Often | All the time | Never | Rarely | Sometimes | Often | All the time |
| 1. My scalp hurts | | | | | | | | | | |
| Baseline | (%X:X%) XX | | (%X:X%) | XX (XX.X%) | X(XX.X%) | XX (XX:X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | (%X:X%) XX |
| Week 2 | (%X:X%) XX | | (%X:XX) XX | (%X:X%) | X(XX.X%) | (%X:X%) XX | XX (XX.X%) | (%X:X%) | (%X:XX) XX | (%X:XX) XX |
| Week 4 | (%X:X%) XX | | XX (XX:X%) | (%X:X%) | X(XX.X%) | XX (XX:X%) | XX (XX.X%) | XX (XX.X%) | (%X:XX) XX | XX (XX.X%) |
| Week 8 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | X(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | (%X:X%) XX | XX (XX.X%) |
| 2. My scalp itches | | | | | | | | | | |
| Baseline | XX (XX:X%) | XX (XX.X%) | XX (XX:X%) | XX (XX.X%) | X(XX:X%) | (%X:X%) | XX (XX.X%) | XX (XX:X%) | XX (XX.X%) | XX (XX.X%) |
| Week 2 | (%X:X%) XX | (%X:X%) | XX (XX:X%) | XX (XX.X%) | X(XX.X%) | (%X:X%) XX | XX (XX.X%) | XX (XX.X%) | (%X:XX) XX | XX (XX.X%) |
| Week 4 | XX (XX.X%) | (%X:X%) | XX (XX.X%) | (%X:X%) | X(XX.X%) | XX (XX:X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Week 8 | (%X:X%) | XX (XX.X%) | (%X:XX) XX | XX (XX.X%) | (%X:XX)X | XX (XX.X%) | XX (XX.X%) | (%X:X%) XX | XX (XX.X%) | XX (XX.X%) |

### Continue for all the 23 questions

Note: Percentages are n/Number of subjects in the mITT Population within planned treatment\*100. Baseline is the last non-missing measurement taken on or before the day of first

application of study drug.
[1] These questions are based on the "How often during the past 4 weeks do these statements describe you?" prompt. Reference Listing: 16.2.6.5



Table 14.2.5.6 Categorical Summary of Individual Responses by Study Visit – Scalpdex Questionnaire ITT Population

Change from Baseline in Dermatology Life Quality Index (DLQI) by Study Visit mITT Population Table 14.2.6.1

(Programming note: Same as table 14.2.4.1; Update footnotes as "Note: Subjects are summarized by planned treatment. Baseline is the last non-missing measurement taken before the first application of study drug. The DLQI total score is calculated as sum of all the 10 questions at each visit and ranges between 0-30. The individual questions are scored as 'Very much' or 'Yes'= 3, 'A Little' = 1, 'Not at all' or 'Not Relevant' = 0. If 1 item is missing, it is scored as 0 for that item. If 2 or more items are missing, the score should not be calculated. Percent change from baseline is calculated as (result – baseline result)\*100."; Change reference listing to 16.2.6.6)



Summary of Dermatology Life Quality Index (DLQI) by Study Visit – ANCOVA mITT Population Table 14.2.6.2

measurement taken on or before the day of first application of study drug. The DLQI total score is calculated as sum of all the 10 questions at each visit and ranges between 0-30. The individual questions are scored as 'Very much' or 'Yes'= 3, 'A lot' = 2, 'A Little' = 1, 'Not at all' or 'Not Relevant' = 0. If 1 item is missing, it is scored as 0 for that item. If 2 or more items (Programming note: Same as table 14.2.4.7; Update Note part of the footnotes as "Note: Subjects are summarized by planned treatment. Baseline is the last non-missing are missing, the score should not be calculated."; Change reference listing to 16.2.6.1, 16.2.6.6)

Change from Baseline in Dermatology Life Quality Index (DLQI) by Study Visit Table 14.2.6.3

before the first application of study drug. The DLQI total score is calculated as sum of all the 10 questions at each visit and ranges between 0-30. The individual questions are scored as 'Very much' or 'Yes'= 3, 'A lot' = 2, 'A Little' = 1, 'Not at all' or 'Not Relevant' = 0. If 1 item is missing, it is scored as 0 for that item. If 2 or more items are missing, the score should (Programming note: Same as table 14.2.4.1; Update footnotes as "Note: Subjects are summarized by planned treatment. Baseline is the last non-missing measurement taken not be calculated. Percent change from baseline is calculated as (result – baseline result)\*100°.; Change reference listing to 16.2.6.6)

Summary of Dermatology Life Quality Index (DLQI) by Study Visit - ANCOVA ITT Population Table 14.2.6.4

(Programming note: Same as table 14.2.4.7; Update Note part of the footnotes as "Note: Subjects are summarized by planned treatment. Baseline is the last non-missing measurement taken on or before the day of first application of study drug. The DLQI total score is calculated as sum of all the 10 questions at each visit and ranges between 0-30. The individual questions are scored as 'Very much' or 'Yes'= 3, 'A lot' = 2, 'A Little' = 1, 'Not at all' or 'Not Relevant' = 0. If 1 item is missing, it is scored as 0 for that item. If 2 or more items are missing, the score should not be calculated."; Change reference listing to 16.2.6.1, 16.2.6.5; Update any instances of mITT with ITT)



Table 14.2.7.1 Change from Baseline in Body Surface Area (BSA) by Study Visit mITT Population (Programming note: Same as table 14.2.4.1; Update footnotes as "Note: Subjects are summarized by planned treatment. Baseline is the last non-missing measurement taken on or before the day of first application of study drug. Change from baseline is calculated as result - baseline result. Percent change from baseline is calculated as (change from baseline)\*100." Change reference listing to 16.2.6.7)

Table 14.2.7.2 Summary of Body Surface Area (BSA) by Study Visit - ANCOVA mITT Population

measurement taken on or before the day of first application of study drug. The BSA affected by seborrheic dermatitis will be calculated as sum of coverage areas of heard, upper and lower limbs, and trunk." Change reference listings to 16.2.6.1, 16.2.6.7) (Programming note: Same as table 14.2.4.7; Update note part of the footnotes as "Note: Subjects are summarized by planned treatment. Baseline is the last non-missing

Table 14.2.7.3
Change from Baseline in Body Surface Area (BSA) by Study Visit ITT Population

(Programming note: Same as table 14.2.4.1; Update footnotes as "Note: Subjects are summarized by planned treatment. Baseline is the last non-missing measurement taken on or before the day of first application of study drug. Change from baseline is calculated as result - baseline result. Percent change from baseline is calculated as (change from baseline)\*100." Change reference listing to 16.2.6.7; Update mITT with ITT)

Table 14.2.7.4 Summary of Body Surface Area (BSA) by Study Visit - ANCOVA mITT Population

measurement taken on or before the day of first application of study drug. The BSA affected by seborrheic dermatitis will be calculated as sum of coverage areas of heard, upper and lower limbs, and trunk." Change reference listings to 16.2.6.7; Update mITT with ITT) (Programming note: Same as table 14.2.4.7; Update note part of the footnotes as "Note: Subjects are summarized by planned treatment. Baseline is the last non-missing



Table 14.3.1.1 Summary of Treatment Emergent Adverse Events Safety Population

| Category | Roflumilast Foam<br>0.3%<br>(N=XX) | Vehicle<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|
| Subjects with at least 1 TEAE | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Maximum Severity of TEAE [1]<br>Grade 1 (Mild) | XX (XX. X%) | XX (XX.X%) | XX (XX.X%) |
| Grade 2 (Moderate) | XX (XX: X%) | XX (XX: X%) | XX (XX: X%) |
| Grade 4 (Life-threatening consequences) | XX (XX. X%) | XX (XX: X%)<br>XX (XX: X%) | (%X:X%)<br>XX (XX:X%) |
| Grade 5 (Death related to AE) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Subjects with a Related TEAE [2] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Subjects with a TEAE Leading to Discontinuation of Study Drug | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Subjects with an SAE | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Subjects with a Grade 5 TEAE [3] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Abbreviations: CTCAE = Common Terminology Criteria for Adverse Events; IP = investigational product; SAE = serious adverse event;

TEAE = treatment emergent adverse event.

Note: Percentages are n/Number of subjects in the Safety population within treatment received\*100. A TEAE is defined as an AE that started post application of IP at the baseline visit through study completion.

[1] Severity grades are reported according to the CTCAE version 4.0. Subjects are counted only once at the worst severity. If a severity designation is missing, it was considered as severe.
[2] AEs with a relationship of possibly, probably, likely, or missing were considered related.
[3] A Grade 5 TEAE is a TEAE leading to death.
Reference Listing: 16.2.7.1

Sponsor Arcutis, Inc. Protocol Number ARQ-154-203 PCN Number ARCU0100 Statistical Analysis Plan,



| System Organ Class | Roflumilast Foam 0.3% (N=XX) | Vehicle | Overall |
|---|---|---|---|
| Preferred Term | | (N=XX) | (N=XX) |
| Subjects with at least 1 TEAE | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| System Organ Class 1 | XX (XX.X%) | (%X:X%) | XX (XX: X%) |
| Preferred Term 1 | XX (XX.X%) | XX (XX:X%) | XX (XX: X%) |
| Preferred Term 2 | XX (XX.X%) | XX (XX. X%) | (%X XX) XX |
| Preferred Term 3 | XX (XX.X%) | XX (XX. X%) | XX (XX X%) |
| System Organ Class 2<br>Preferred Term 1<br>Preferred Term 2 | (%X XX)<br>(%X XX)<br>XX<br>XX<br>XX | XX (XX. X%)<br>XX (XX. X%)<br>XX (XX. X%) | XX (XX. X%)<br>XX (XX. X%)<br>XX (XX. X%) |
| Preferred Term 3 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Abbreviations: AE = adverse event; IP = investigational product; MedDRA = Medical Dictionary for Regulatory Activities; TEAE =

treatment emergent adverse event.

Note: Percentages are n/Number of subjects in the Safety population within treatment received and overall\*100. AEs were coded using MedDRA version 23.0. A TEAE is defined as an AE that started post application of IP at the baseline visit through study completion. Subjects are counted once for each system organ class (SOC) and once for each preferred term (PT). AEs are displayed by descending frequency of SOC, then PT within SOC, and then alphabetically by PT.

Reference Listing: 16.2.7.1

Programming note: SOC & PT text should be presented as is from the dataset.



Incidence of Treatment Emergent Adverse Events by System Organ Class, Preferred Term, and Maximum Severity Safety Population Table 14.3.1.3

| System Organ Class<br>Preferred Term<br>Maximum Severity [1] | Roflumilast Foam 0.3%<br>(N=XX) | Vehicle<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|
| Subjects with at least 1 TEAE Grade 1 (Mild) Grade 2 (Moderate) Grade 3 (Severe) Grade 4 (Life-threatening consequences) Grade 5 (Death related to AE) | X (XX X%)<br>XX (XX X%) | (%X XX)<br>(XX)<br>(XX)<br>(XX)<br>(XX)<br>(XX)<br>(XX)<br>(XX) | (%X:XX)<br>(%X:XX)<br>(%X:XX)<br>(%X:XX)<br>(X:XX)<br>(X:XX |
| System Organ Class 1 Grade 1 (Mild) Grade 2 (Moderate) Grade 3 (Severe) Grade 4 (Life-threatening consequences) Grade 5 (Death related to AE | X (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | (%X.XX)<br>(XX)<br>(XX)<br>(XX)<br>(XX)<br>(XX)<br>(XX)<br>(XX) | (%::X) |
| Preferred Term 1<br>Grade 1 (Mild)<br>Grade 2 (Moderate) | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) |

Abbreviations: AE = adverse event; IP = investigational product; CTCAE = Common Terminology Criteria for Adverse Events; MedDRA = Medical Dictionary for Regulatory Activities; TEAE = treatment emergent adverse event.

Note: Percentages are n/Number of subjects in the Safety population within treatment received and overall\*100. AEs were coded using MedDRA

version 23.0. A TEAE is defined as an AE that started post application of IP at the baseline visit through study completion. Subjects are counted

once for each system organ class (SOC) and once for each preferred term (PT) at the maximum severity.

[1] Severity grades are reported according to the CTCAE version 4.0. The severity shown is the greatest severity reported for a particular subject (Death related to AE > Life-threatening consequences > Severe > Moderate > Mild). AEs with a missing severity were counted as Severe. AEs are displayed by descending frequency of SOC, then PT within SOC, and then alphabetically by PT.

Reference Listing: 16.2.7.1

Programming note: SOC & PT text should be presented as is from the dataset.



Incidence of Treatment Emergent Adverse Events by System Organ Class, Preferred Term, and Relationship to Study Drug Safety Population Table 14.3.1.4

| System Organ Class | Roflumilast Foam | | |
|-------------------------------|------------------|------------|------------|
| Preferred Term | 0.3% | Vehicle | Overall |
| Relationship [1] | (N=XX) | (N=XX) | (N=XX) |
| Subjects with at least 1 TEAE | (%X:XX) XX | (%X:X%) | (XX:X%) |
| Related | (%X:XX) XX | XX (XX.X%) | (%X XX) XX |
| Not Related | (%X:XX) XX | (%X:X%) XX | (%X:XX) |
| System Organ Class 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Related | (%X:X%) XX | (%X:X%) XX | (%X:XX) XX |
| Not Related | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 1 | (%X:X%) | (%X:X%) | (%X:X%) |
| Related | (%X:XX) XX | (%X:XX) XX | (%X:XX) |
| Not Related | (%X:XX) XX | (%X:XX) XX | XX (XX:X%) |

Abbreviations: AE = adverse event; IP =investigational product; MedDRA = Medical Dictionary for Regulatory Activities; TEAE = treatment emergent adverse event.

relationship category. The relationship shown is the greatest relationship reported for a particular subject (Related > Not Related). AEs with a missing relationship were counted as Related. AEs are displayed by descending frequency of SOC, then PT within SOC, Note: Percentages are n/Number of subjects in the Safety population within treatment received and overall\*100. AEs were coded using MedDRA version 23.0. A TEAE is defined as an AE that started post application of IP at the baseline visit through study completion. Subjects are counted once for each system organ class (SOC) and once for each preferred term (PT) at the greatest

and then alphabetically by PT. [1] Related = Probably Related, Possibly Related, Likely Related, and Missing; Not Related = Unrelated and Unlikely Related. Reference Listing: 16.2.7.1

Programming note: SOC & PT text should be in proper case in table, as shown in the shell.



Incidence of Treatment Emergent Adverse Events Leading to Study Drug Discontinuation by System Organ Class and Preferred Term Safety Population Table 14.3.1.5

(Same shell as Table 14.3.1.2)

Incidence of Serious Adverse Events by System Organ Class and Preferred Term Safety Population Table 14.3.2.1

(Same shell as Table 14.3.1.2; first-row text is "Subjects with at least 1 SAE"; add SAE = serious adverse event)

Table 14.3.2.2 Incidence of Serious Adverse Events by System Organ Class, Preferred Term, and Relationship to Study Drug Safety Population

(Same shell as Table 14.3.1.4; first-row text is "Subjects with at least 1 SAE"; add SAE = serious adverse event)



Table 14.3.2.3 Incidence of Serious Adverse Events by System Organ Class, Preferred Term, and Maximum Severity Safety Population

(Same shell as Table 14.3.1.3; first-row text is "Subjects with at least 1 SAE"; add SAE = serious adverse event)



Table 14.3.3.1 Listing of Adverse Events Leading to Study Drug Discontinuation Safety Population

| Subject Treatment<br>ID Received | System Organ Class/<br>Preferred Term/<br>Verbatim Term | Outcome/ Start Date/Time (Study Day)/ CTCAE Toxicity Grade/ Study Drug Action Taken/ End Date/Time (Study Day) Relationship Other Action Taken | CTCAE Toxicity Grade.<br>Relationship | Outcome/<br>/ Study Drug Action Taken/<br>Other Action Taken | Serious?/<br>Criteria Met |
|---|---|---|---|---|---|
| XXXXXXXX XXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMONYYYY/hh:mm (X)/<br>DDMONYYYY/hh:mm (X) | XXXXXXXXXX | /XXXXXXXXXXXX/<br>/XXXXXXXXXXXXXXXXXXXXXX | × |
| XXXXXXX XXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMONYYYY/hh:mm (X)/<br>DDMONYYYY/hh:mm (X) | XXXXXXXXXX | /xxxxxxxxx<br>/xxxxxxxxxxxxxxxxxxxxxxxxxx | × |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMONYYYY/hh:mm (X)/<br>DDMONYYYY/hh:mm (X) | XXXXXXXXXX | /xxxxxxxxxx/<br>/xxxxxxxxxxxxxxxxxxxxxxxx | XXXXXXXX |

Abbreviations: CTCAE = Common Terminology Criteria for Adverse Events; MedDRA = Medical Dictionary for Regulatory Activities.

Note: Study day is calculated relative to the date of first application of study drug. AEs were coded using MedDRA version 23.0. Severity grades are reported according to the CTCAE version 4.0. Programming note: If time missing, display "- ---". "Other Action Taken" will be either None, Concomitant Medication, Non-drug Therapy, Hospitalization or Prolongation of Hospitalization, Discontinued Study or Other; if specify text is needed, concatenate "Concomitant Medication:" or "Other:" with the text. If Serious? is Yes, concatenate all serious criteria marked as Yes with a semicolon. If no events meet the criteria for display, present are reported." SOC & PT text should be presented as is from the dataset.






(Same shell as Table 14.3.3.1)

Table 14.3.3.3 Listing of Deaths Safety Population

(Same shell as Table 14.3.3.1)



Table 14.3.5.1.1 Summary of Clinical Chemistry Laboratory Results by Study Visit Safety Population

Parameter: XXXXXXX (unit)

| 21-37-1-1-10 | Roflumilast Foam 0.3% | Foam 0.3% | Vehicle | <u>ə</u> S | Overal | rall |
|---|---|---|---|---|---|---|
| Statistic | Observed | CFB | Observed | CFB | Observed | CFB |
| Baseline | | | | | | |
| | × | | × | | × | |
| Mean (SD) | XX.X (XX.XX) | | (XX:XX) | | XX.X (XX.XX) | |
| Median | XX | | ××× | | ××× | |
| Min, Max | XX, XX | | XX, XX | | ×, × | |
| Week 8 | | | | | | |
| u | × | × | × | × | × | × |
| Mean (SD) | XX.XX (XX.XX) | XX.X (XX.XX) | (XX:XX) | (XX:XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | ××× | ××× | ××× | ××× | ××× | ××× |
| Min, Max | XX, XX | XX, XX | XX XX | ×××× | ×, × | XX, XX |

## Continue for other parameters. Sort alphabetically by parameter.

Abbreviation: CFB = change from baseline.

Note: Subjects are summarized by treatment received and overall. Baseline is the last non-missing measurement taken before the first application of study drug. Reference Listing: 16.2.8.1.1



Table 14.3.5.1.2
Shift from Baseline in Clinical Chemistry Laboratory Results by Study Visit Safety Population

Parameter: XXXXXXX (unit)

| | | | | | | | Baseline Grade | rade | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Roi | Roflumilast Foam 0.3% (N=XX) | 3% | | | | Vehicle (N=XX) | icle<br>XX) | |
| Study Visit | Study Visit Post-Baseline<br>Grade | Missing | Low | Normal | High | Total | Missing | Low | Normal | High | Total |
| Week 8 | Missing | | | | | | | | | | |
| | Low | (%X:X%) | (%X:X%) | (%X:X%) | (%X:X%) | XX (XX:X%) | (%X:X%) | XX (XX:X%) | (%X:X%) | (%X:X%) | (%X:X%) XX |
| | Normal | XX (XX.X%) | (%X.X%) | XX (XX:X%) | XX (XX.X%) | XX (XX:X%) | XX (XX.X%) | XX (XX.X%) | XX (XX:X%) | XX (XX:X%) | XX (XX.X%) |
| | High | (%X:XX) XX | (%X:X%) XX | (%X:X%) | (%X:XX) XX | (%X:XX) XX | XX (XX.X%) | (%X:X%) | XX (XX:X%) | (%X:X%) | (%X:XX) XX |
| | Total | (%X:X%) XX | (%X:X%) XX | (%X:X%) | (%X.XX) XX | (%X:X%) | XX (XX.X%) | (%X:X%) | (%X:X%) XX | XX (XX: X%) | (%X:XX) XX |
| | | | | Repeat for ( | Overall and all c | t for Overall and all clinical chemistry parameters (excluding serum HCG results). | parameters (excl | uding serum HC | 3G results). | | |

Note: Percentages are n/Number of subjects in the Safety population within treatment received\*100. Baseline is the last non-missing measurement taken before the first application of study drug. Reference Listing: 16.2.8.1.1




Summary of Hematology Laboratory Results by Study Visit Safety Population Table 14.3.5.2.1

(Same shell as Table 14.3.5.1.1; Reference Listing: 16.2.8.1.2)

Shift from Baseline in Hematology Laboratory Results by Study Visit Safety Population Table 14.3.5.2.2

(Same shell as Table 14.3.5.1.2; Reference Listing: 16.2.8.1.2)

Table 14.3.5.3.1 Summary of Quantitative Urinalysis Laboratory Results by Study Visit Safety Population

(Same shell as Table 14.3.5.1.1; Reference Listing: 16.2.8.1.3)

Table 14.3.5.3.2 Shift from Baseline in Quantitative Urinalysis Laboratory Results by Study Visit Safety Population

(Same shell as Table 14.3.5.1.2; Reference Listing: 16.2.8.1.3)



Table 14.3.5.3.3 Summary of Qualitative Urinalysis Laboratory Results by Study Visit Safety Population

| | : 41 | | |
|---------------|------------------|------------|---------------|
| Study Visit | Roflumilast Foam | Vehicle | Overall |
| Category | 0.3%<br>(XX=X) | (X=X) | (N=XX) |
| oring of | , , , , , , | | |
| XXXXXXXX | (%X XX) XX | (%X XX) XX | (%X XX) XX |
| | | (0/2/20) | (0/1/20/) 10/ |
| XXXXXXXXXX | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Week 8 | | | |
| XXXXXXXX | XX (XX.X%) | XX (XX.X%) | (%X:X%) |
| XXXXXXXXXXXXX | XX (XX:X%) | (%X:XX) XX | (%X:X%) |
| XXXXXXXX | XX (XX.X%) | XX (XX.X%) | (%X:X%) |

Note: Percentages are n/Number of subjects in the Safety population within treatment received and overall\*100. Baseline is the last non-missing measurement taken before the first application of study drug. Reference Listing: 16.2.8.1.3



Table 14.3.6.1 Shift from Baseline in Patient Health Questionnaire (PHQ-8) by Study Visit Safety Population

| -oam 0.3% Vehicle (N=XX) | Moderately arate Severe Severe None Mild Moderate Severe Severe | XX XX XX XX XX | (XX.X%) (XX.X%) (XX.X%) (XX.X%) (XX.X%) (XX.X%) | × | (XX.X%) (XX.X%) | × | (XX.X%) (XX.X%) (XX.X%) (XX.X%) (XX.X%) (XX.X%) | × × × × × × × | (XX.X%) (XX.X%) (XX.X%) (XX.X%) (XX.X%) (XX.X%) | × | (XX.X%) (XX.X%) (XX.X%) (XX.X%) (XX.X%) (XX.X%) | × | (XX.X%) (XX.X%) (XX.X%) (XX.X%) (XX.X%) (XX.X%) | >> | XX XX XX XX |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | None | × | (XX.X%) | × | (XX.XX) | × | (XX.XX) | × | (XX.XX) | × | (XX:X%) | × | (XX:XX) | × | (XX.X%) |
| | Missing | × | (XX.X%) | × | (XX:X%) | × | (XX:X%) | × | (XX:X%) | × | (XX:X%) | × | (XX:X%) | × | (XX.XX) |
| | Severe | × | (XX.XX) | × | (XX:X%) | × | (XX:X%) | × | (XX:X%) | × | (XX.XX) | × | (XX:X%) | × | (XX:X%) |
| | Moderately<br>Severe | × | (XX:XX) | × | (XX:XX) | × | (XX:XX) | × | (XX:XX) | × | (XX:XX) | × | (%X:X%) | × | (XX:X%) |
| XX) | Moderate | × | (XX:XX) | × | (%X:X%) | × | (%X:X%) | × | (%X:X%) | × | (XX:XX) | × | (%X:X%) | × | (XX:X%) |
| | Mild | × | (XX:X%) | × | (XX:XX) | × | (XX:XX) | × | (XX:XX) | × | (XX:X%) | × | (XX:XX) | × | (XX:X%) |
| | None | × | (XX:X%) | × | (XX:X%) | × | (XX:X%) | × | (XX:X%) | × | (XX:X%) | × | (XX:X%) | × | (XX.X%) |
| | Missing | × | (XX.XX) | × | (XX.XX) | × | (XX.XX) | × | (XX.XX) | × | (XX.XX) | × | (XX.XX) | × | (XX.XX) |
| | Study Visit<br>Category [1] | Week 4 | | Missing | 1 | None | | Mild | | Moderate | | Moderately | Severe | Severe | |

Programming note: Add Total category for both column and row. Repeat for Overall and continue for Week 8

Abbreviation: PHQ = patient health questionnaire.

Note: Percentages are n/Number of subjects in the Safety population within treatment received\*100. Baseline is the last non-missing measurement taken on or before the day of first application of study drug. PHQ total score is calculated as sum of the 8 questions (individual questions scored as Not at all=0, Several days=1, More than half the days=2, and Nearly every day=3). The total score ranges from 0 to 24. If more than 1 item is missing the score should not be calculated. If 1 item is missing the score is calculated as (sum of answered items\*8)/number of answered items.

[1] If the total score ranges from 0 to 4, it is classified as None – Minimal Depression; 5 – 9 classified as Mild; 10 – 14 classified as Moderate; 15-19 classified as Moderately Severe; 20 – 24 classified as Severe Depression.

Reference Listing: 16.2.9.8



Summary of Investigator Local Tolerability Assessment (Dermal Response) by Study Visit Safety Population Table 14.3.6.2.1

(Same shell as Table 14.3.5.1.1; Reference Listing: 16.2.9.1; Repeat for Week 4, Week 8; Add "Abbreviation: IP = investigational product." as the first line of footnotes. Add this line at the end in note footnote – "Lower scores indicate no evidence of irritation while higher scores indicate worsening reaction. Investigator tolerability assessment should be performed prior to the IP application in the study site. Subjects not meeting this condition on baseline visit are completely removed from the table summary."; Update the baseline definition as "Baseline is the last non-missing measurement taken on or before the day of first application of study drug.") 



Summary of Investigator Local Tolerability Assessment (Dermal Response) by Study Visit Categorical Results
Safety Population Table 14.3.6.2.2

| Category | 0.3% (N=XX) | (XX=N) | (N=XX) |
|---|---|---|---|
| Baseline | | | |
| 0 = No evidence of irritation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 1 = Minimal erythema | XX (XX: X%) | XX (XX:X%) | XX (XX.X%) |
| 2 = Definite erythema | (%X:X%) | XX (XX.X%) | XX (XX.X%) |
| 3 = Erythema and papules | (%X:XX) XX | (%X:XX) XX | XX (XX:X%) |
| 4 = Definite edema | (%X:X%) | (%X:XX) XX | (%X:XX) |
| 5 = Erythema, edema and papules | (%X:XX) XX | (%X:XX) XX | XX (XX:X%) |
| 6 = Vesicular eruption | (%X:X%) | XX (XX.X%) | (%X:X%)<br>XX |
| 7 = Strong reaction spreading beyond application site | | | |
| Week 4 | | | |
| 0 = No evidence of irritation | (%X:X%) | XX (XX.X%) | (%X:X%) |
| 1 = Minimal erythema | (%X:XX) XX | XX (XX:X%) | (%X:XX) XX |
| 2 = Definite erythema | (%X:X%) | (%X:XX) | (%X:XX) |
| 3 = Erythema and papules | (%X:X%) | (%X:XX) XX | (%X:XX) |
| 4 = Definite edema | (%X:XX) XX | XX (XX.X%) | (%X:X%) |
| 5 = Erythema, edema and papules | (%X:X%) | (%X:XX) XX | (%X:XX) |
| 6 = Vesicular eruption | (%X:XX) XX | XX (XX.X%) | (%X:X%) |
| 7 = Strong reaction spreading beyond application site | (%X XX) XX | (%X XX) XX | (%X XX) XX |

#### Repeat for Week 8

Abbreviation: IP = investigational product.

Note: Percentages are n/Number of subjects in the Safety Population within treatment received and overall\*100. Baseline is the last non-missing measurement taken on or before the day of first application of study drug. Investigator tolerability assessment should be performed prior to the IP application in the study site. Subjects not meeting this condition on baseline visit are completely removed from the table summary.

Reference Listing: 16.2.9.1



Summary of Investigator Local Tolerability Assessment (Other Effects) by Study Visit Table 14.3.6.2.3

| Categorical Results | Safety Population |
|---------------------|-------------------|

| Study Visit<br>Category | Roflumilast Foam<br>0.3%<br>(N=XX) | Vehicle<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|
| Baseline | | | |
| A = Slight glazed appearance | XX (XX: X%) | XX (XX.X%) | XX (XX.X%) |
| B = Marked glazing | (%X:X%) | XX (XX.X%) | XX (XX:X%) |
| C = Glazing with peeling and cracking | (%X:X%) | (%X:XX) XX | XX (XX:X%) |
| D = Glazing with fissures | (%X:X%) | (%X:XX) XX | XX (XX:X%) |
| E = Film of dried serous exudates | XX (XX: X%) | (%X:X%) XX | XX (XX:X%) |
| F = Small petechial erosions and/or scabs | (%X:XX) | (%X:XX) XX | XX (XX:X%) |
| G = No other effects | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Week 4 | | | |
| A = Slight glazed appearance | XX (XX.X%) | XX (XX.X%) | XX (XX:X%) |
| B = Marked glazing | (%X:XX) | (%X:XX) XX | XX (XX:X%) |
| C = Glazing with peeling and cracking | (%X:X%) | XX (XX.X%) | XX (XX:X%) |
| D = Glazing with fissures | (%X:XX) | XX (XX.X%) | XX (XX:X%) |
| E = Film of dried serous exudates | (%X.XX) | (%X:XX) XX | XX (XX:X%) |
| F = Small petechial erosions and/or scabs | (%X:X%) | XX (XX.X%) | XX (XX:X%) |
| G = No other effects | XX (XX: X%) | (%X:XX) XX | (%X:XX) XX |

#### Repeat for Week 8

Abbreviation: IP = investigational product.

Note: Percentages are n/Number of subjects in the Safety Population within treatment received and overall\*100. Baseline is the last non-missing measurement taken on or before the day of first application of study drug. Investigator tolerability assessment should be performed prior to the IP application in the study site. Subjects not meeting this condition on baseline visit are completely removed from the table summary.

Reference Listing: 16.2.9.1



Summary of Subject Local Tolerability Assessment by Study Visit Safety Population Table 14.3.6.3.1

the end in note footnote – "Lower scores indicate no sensation while higher scores indicate worsening/severe reaction. This assessment should be performed 10 – 15 minutes after the application of IP in the study site. Subjects not meeting this condition on baseline visit are completely removed from the table summary.") Update Baseline definition as Baseline for subject local tolerability assessment is the last non-missing measurement taken on the day of first application of study drug. (Same shell as Table 14.3.5.1.1; Reference Listing: 16.2.9.2; Repeat for Week 4, Week 8; Add "Abbreviation: IP = investigational product." as the first line of footnotes. Add this line at


Sponsor Arcutis, Inc. Protocol Number ARQ-154-203 PCN Number ARCU210100 Statistical Analysis Plan,

Summary of Subject Local Tolerability Assessment by Study Visit Categorical Results Safety Population Table 14.3.6.3.2

| Study Visit<br>Category | Roflumilast Foam 0.3% | Vehicle<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|
| | (XX=N) | | |
| Baseline | | | |
| 0 = None (no sensation) | XX (XX.X%) | XX (XX.X%) | (%X:X%) |
| 1 = Mild (slight warm, tingling sensation) | (%X:XX) XX | (%X:XX) XX | (%X:XX) XX |
| 2 = Moderate (definite warm, tingling sensation) | (%X:X%) | (%X:X%) | (%X:X%) |
| 3 = Severe (hot, tingling/stinging sensation) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Week 4 | | | |
| 0 = None (no sensation) | XX (XX: X%) | XX (XX.X%) | XX (XX.X%) |
| 1 = Mild (slight warm, tingling sensation) | (%X:XX) XX | XX (XX:X%) | (%X:X%) XX |
| 2 = Moderate (definite warm, tingling sensation) | (%X:XX) XX | XX (XX:X%) | (%X:XX) XX |
| 3 = Severe (hot, tingling/stinging sensation) | XX (XX. X%) | XX (XX.X%) | XX (XX.X%) |

#### Repeat for Week 8

Abbreviation: IP = investigational product.

Note: Percentages are n/Number of subjects in the Safety Population within treatment received and overall\*100. Baseline for subject local tolerability assessment is the last non-missing measurement taken on the day of first application of study drug. This assessment should be performed 10 – 15 minutes after the application of IP in the study site. Subjects not meeting this condition on baseline visit are completely removed from the table summary.

Reference Listing: 16.2.9.2





Summary of Vital Signs by Study Visit Safety Population Table 14.3.6.4.1

(Same shell as Table 14.3.5.1.1; visits include Baseline, Week 2, Week 8, Week 9; parameters include Temperature (°C), Heart Rate (bpm), Sitting Systolic Blood Pressure (mmHg), Height (cm), Weight (kg), BMI (kg/m²) [1]; Update Baseline definition as "Baseline is the last non-missing measurement taken on or before the first application of study drug." [1] Body Mass Index (BMI) = weight (kg) / [height (m)]².

Reference Listings: 16.2.9.4.1, 16.2.9.4.2)



Table 14.3.6.4.2 Shift from Baseline in Weight by Study Visit Safety Population

| Study Visit<br>Category | Roflumilast Foam 0.3% (N=XX) | Vehicle<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|
| Week 2 | | | |
| Change from Baseline ≤-10% | XX (XX.X%) | (%X:XX) | (%X:X%) |
| Change from Baseline ≤-5% | XX (XX.X%) | (%X:X%) | (%X:XX) XX |
| Change from Baseline ≥5% | (%X.XX) | (%X:XX) XX | (%X:XX) XX |
| Change from Baseline ≥10% | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Week 4 | | | |
| Change from Baseline ≤-10% | XX (XX.X%) | (%X:X%) | (%X:XX) |
| Change from Baseline ≤-5% | (%X:X%) | (%X:XX) XX | (%X:XX) XX |
| Change from Baseline ≥5% | (%X.XX) | (%X:XX) XX | (%X:XX) XX |
| Change from Baseline ≥10% | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Week 8 | | | |
| Change from Baseline ≤-10% | XX (XX.X%) | XX (XX.X%) | (%X:XX) |
| Change from Baseline ≤-5% | (%X.XX) | (%X:XX) XX | (%X:XX) XX |
| Change from Baseline ≥5% | (%X.XX) | (%X:XX) XX | (%X:XX) XX |
| Change from Baseline ≥10% | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Programming note: Continue for Week 9

Note: Percentages are n/Number of subjects in the Safety population within treatment received and overall\*100. Baseline is the last non-missing measurement taken on or before the first application of study drug.
Reference Listing: 16.2.9.4.2



Table 14.3.6.4.3 Shift from Baseline in BMI by Study Visit Safety Population

| | | se | (%XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
|---|---|---|---|
| | | Obese | (%X:X%)<br>XX (XX:X%)<br>XX (XX:X%)<br>XX (XX:X%)<br>XX (XX:X%) |
| | | Overweight | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) |
| | Vehicle<br>(N=XX) | Normal | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) |
| Grade | | Underweight | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) |
| Baseline Grade | | Missing | (%X.XX)<br>(XX)<br>(XX)<br>(XX)<br>(XX)<br>(XX)<br>(XX)<br>(XX) |
| | | Obese | (%X:X%)<br>XX (XX:X%)<br>XX (XX:X%)<br>XX (XX:X%)<br>XX (XX:X%) |
| | 3% | Overweight | (%X:X%)<br>XX (XX:X%)<br>XX (XX:X%)<br>XX (XX:X%)<br>XX (XX:X%) |
| | Roflumilast Foam 0.3% (N=XX) | Normal | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) |
| | Rofl | Missing Underweight | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) |
| | | Missing | XX (XX. X%)<br>XX (XX. X%)<br>XX (XX. X%)<br>XX (XX. X%)<br>XX (XX. X%) |
| | | Post-<br>Baseline<br>Grade [1] | Missing<br>Underweight<br>Normal<br>Overweight<br>Obese |
| | | Study<br>Visit | Week 2 |

Repeat for Overall and Week 4, Week 8, and Week 9

Note: Percentages are n/Number of subjects in the Safety population within treatment received and overall\*100. Baseline is the last non-missing measurement taken on or before the day of first application of study drug. BMI is derived as (weight in kg)/[(height in cm/100)²].
[1] If BMI is below 18.5 then it is categorized as underweight; if BMI ranges between 18.5 – 24.9 then it is categorized as not it is categorized as overweight; if BMI is greater than 30.0 then it is categorized as obese.

Reference Listings: 16.2.9.4.1, 16.2.9.4.2


Sponsor Arcutis, Inc. Protocol Number ARQ-154-203 PCN Number ARCU210100 Statistical Analysis Plan,



Shift from Baseline in Weight by Study Visit – by Weight Loss Intentional/Non-Intentional Safety Population Table 14.3.6.4.4

| Weight Loss: Intentional | | | |
|---|---|---|---|
| Study Visit | Roflumilast Foam 0.3% | Vehicle | Overall |
| Category | (N=XX) | (N=XX) | (N=XX) |
| C /1- /W | | | |
| week z | | | |
| Change from Baseline ≤-10% | (%X:XX) | (%X:X%)<br>XX | (%X:XX)<br>XX |
| Change from Baseline ≤-5% | XX (XX.X%) | (%X:X%) | (%X:X%) |
| Change from Baseline ≥5% | XX (XX X%) | (%X:XX) | (%X:XX) XX |
| Change from Baseline ≥10% | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Week 4 | | | |
| Change from Baseline ≤-10% | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Change from Baseline ≤-5% | (%X:X%) | (%X:X%) XX | (%X:XX) |
| Change from Baseline ≥5% | (%X:X%) | XX (XX.X%) | (%X:XX) XX |
| Change from Baseline ≥10% | (%X:X%) | XX (XX.X%) | XX (XX.X%) |
| Week 8 | | | |
| Change from Baseline ≤-10% | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Change from Baseline ≤-5% | XX (XX X%) | (%X:XX) XX | (%X:XX) XX |
| Change from Baseline ≥5% | XX (XX.X%) | (%X:XX) XX | (%X:XX) XX |
| Change from Baseline ≥10% | (%X:X%) | XX (XX.X%) | (%X:XX) XX |

Programming note: Continue for Week 9 and repeat for Weight Loss: Not Intentional or Missing

Note: Percentages are n/Number of subjects in the Safety population within treatment received and overall\*100. Baseline is the last non-missing measurement taken on or before the first application of study drug.
Reference Listing: 16.2.9.4.2



Table 14.3.6.4.5
Shift from Baseline in BMI by Study Visit - by Weight Loss Intentional/Non-Intentional Safety Population

#### Weight Loss: Intentional

| | | Obese | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) |
|---|---|---|---|
| | | Overweight | (%XXXX)<br>(%XXXXX)<br>(%XXXXXX)<br>(%XXXXXX)<br>(%XXXXXXX)<br>(%XXXXXXX)<br>(%XXXXXXXXXX |
| | Vehicle<br>(N=XX) | Normal | (%XXX)<br>(%XXX)<br>(%XXX)<br>(XXXX)<br>(XXXXX)<br>(XXXXXX)<br>(XXXXXX)<br>(XXXXXX)<br>(XXXXXX)<br>(XXXXXX)<br>(XXXXXX)<br>(XXXXXX)<br>(XXXXXXX)<br>(XXXXXXX)<br>(XXXXXXXX |
| Grade | | dissing Underweight | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) |
| Baseline Grade | | Missing | (%XXX)<br>XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | | Obese | (%X XX)<br>(XX)<br>( |
| | %8 | Overweight | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) |
| | Roflumilast Foam 0.3% (N=XX) | Normal | (%X:X%)<br>XX (XX:X%)<br>XX (XX:X%)<br>XX (XX:X%)<br>XX (XX:X%) |
| | Roflı | Aissing Underweight Normal | (%XXX%)<br>XX (XXXX%)<br>XX (XXXX%)<br>XX (XXXX%)<br>XX (XXXX%) |
| | | Missing | XX (XX. X%)<br>XX (XX. X%)<br>XX (XX. X%)<br>XX (XX. X%)<br>XX (XX. X%) |
| | | Post-<br>Baseline<br>Grade [1] | Missing<br>Underweight<br>Normal<br>Overweight<br>Obese |
| | | Study<br>Visit | Week 2 |

Add Total category for row and column. Repeat for Overall and Week 4, Week 8, and Week 9 and continue for Weight Loss: Not Intentional or Missing

Note: Percentages are n/Number of subjects in the Safety population within treatment received and overall\*100. Baseline is the last non-missing measurement taken on or before the day of first application of study drug. BMI is derived as (weight in kg)/[(height in cm/100)²].
[1] If BMI is below 18.5 then it is categorized as underweight; if BMI ranges between 18.5 – 24.9 then it is categorized as underweight; if BMI ranges between 18.5 – 24.9 then it is categorized as overweight; if BMI is greater than 30.0 then it is categorized as obese.

Reference Listings: 16.2.94.1, 16.2.94.2

Protocol Number ARQ-154-203 PCN Number ARCU210100 Statistical Analysis Plan, Sponsor Arcutis, Inc.



Summary of Columbia-Suicide Severity Rating Scale (C-SSRS) Suicidal Ideation and Suicidal Behavior by Study Visit Safety Population Table 14.3.6.5

| Study Visit<br>C-SSRS Section<br>C-SSRS Item | Roflumilast Foam 0.3% (N=XX) | Vehide<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|
| Screening<br>Suicidal Ideation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Wish to be Dead | XX (XX: X%) | XX (XX.X%) | XX (XX.X%) |
| Non-Specific Active Suicidal Thoughts | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Active Suicidal Ideation with Any Methods | XX (XX.X%) | (%X:XX) | XX (XX.X%) |
| Active Suicidal Ideation with Some Intent | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Active Suicidal Ideation with Specific Plan | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Suicidal Behavior | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Actual Attempt | XX (XX. X%) | (%X:XX) XX | XX (XX.X%) |
| Subject Engaged in Non-Suicidal Self-Injurious Behavior | XX (XX.X%) | (%X:XX) XX | (%X:X%)<br>XX |
| Interrupted Attempt | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Aborted Attempt | XX (XX.X%) | (%X:XX) XX | (%X:X%)<br>XX |
| Preparatory Acts or Behavior | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Repeat for Baseline, Week 4, and Week 8; Add Suicide as a separate row for all visits except Screening.

Abbreviation: C-SSRS = Columbia-Suicide Severity Rating Scale.

Note: Percentages are n/Number of subjects in the Safety population within treatment received and overall\*100. Baseline is the last non-missing measurement taken before the first application of study drug. The number and percent of subjects who experience the event at least once during treatment are summarized. Subjects are counted once for each C-SSRS item answered "Yes" during treatment period. "Baseline/Screening" version will be used for Screening visit and "Since Last Visit" was used for all other visits. Reference Listing: 16.2.9.9


Table 14.3.6.6 Summary of Physical Examination by Study Visit Safety Population

| Study Visit<br>Body System<br>Category | Roflumilast Foam 0.3%<br>(N=XX) | Vehicle<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|
| Screening<br>Skin | | | |
| Nomal | (%X:X%) | XX (XX.X%) | (%X:XX) |
| Abnormal (NCS) | XX (XX.X%) | (%X:X%) XX | (%X:XX) |
| Abnormal (CS) | XX (XX.X%) | XX (XX.X%) | (%X:XX) |
| Missing | (%X:X%) | (%X:X%) | (%X:XX) XX |
| Total | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Lungs | | | |
| Normal | XX (XX.X%) | (%X:X%) | XX (XX.X%) |
| Abnormal (NCS) | XX (XX.X%) | XX (XX.X%) | (%X:XX) |
| Abnormal (CS) | (%X:X%) | (%X:XX) XX | (%X:XX) XX |
| Missing | (%X:X%) XX | (%X:X%) XX | (%X:XX) XX |
| Total | XX (XX.X%) | XX (XX.X%) | (%X:XX) XX |
| Heart | | | |
| Normal | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Abnormal (NCS) | (%X.XX) | (%X:X%) XX | (%X:XX) XX |
| Abnormal (CS) | (%X:X%) | (%X:XX) XX | (%X:XX) XX |
| Missing | XX (XX.X%) | XX (XX.X%) | (%X:XX) |
| Total | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Repeat for Baseline, Week 8

Abbreviations: CS = clinically significant; NCS = not clinically significant.

Note: Percentages are n/Number of subjects in the Safety population within treatment received an overall\*100.

Reference Listing: 16.2.9.5

Sponsor Arcutis, Inc. Protocol Number ARQ-154-203 PCN Number ARCU210100 Statistical Analysis Plan,



Summary of Concomitant Medications by ATC Class Level 4 and Preferred Term Safety Population Table 14.3.6.7

| ATC Class Level 4<br>Preferred Term | Roflumilast Foam 0.3% (N=XX) | Vehicle<br>(N=XX) | Overall<br>(N=XX) |
|---|---|---|---|
| Subjects with at least 1 Concomitant Medication | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| ATC Class 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Lerm 1<br>Preferred Term 2 | XX (XX. X%)<br>XX (XX. X%) | XX (XX.X%)<br>XX (XX.X%) | (%X:X%)<br>XX (XX:X%) |
| Preferred Term 3 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| ATC Class 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 1 | (%X:X%) | (XX.X%) | (XX:X%) |
| Preferred Term 2 | (%X:X%) | (XX.X%) | (%X:XX) XX |
| Preferred Term 3 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Abbreviations: ATC = Anatomic Therapeutic Chemical; PT = preferred term; WHO-DDE = World Health Organization-Drug Dictionary Enhanced.

Note: Percentages are n/Number of subjects in the Safety population within treatment received\*100. Medications were coded using WHO-DDE Global B3 version September 2019. Concomitant medications are all medications that were continuing or starting after first application of study drug. Medications are displayed by alphabetical order of ATC Level 4 classification, then descending frequency of PT within ATC, and then alphabetically by PT. Subjects were counted only once for each ATC and PT. Reference Listing: 16.2.9.7

Programming note: ATC & PT text should be presented as is from dataset.

Table 14.4.1.1 Summary of Pharmacokinetic Concentration Results by Study Visit PK Population

| Study Visit | |
|-------------|-----------------------|
| Time Point | Roflumilast Foam 0.3% |
| Statistic | (N=XX) |
| Baseline | |
| Predose | |
| ב | × |
| Mean (SD) | XX.X (XX.XX) |
| Median | XXX |
| Min, Max | XX, XX |
| Week 4 | |
| Predose | |
| С | × |
| Mean (SD) | XX.X (XX.XX) |
| Median | XXX |
| Min, Max | XX, XX |
| Postdose | |
| u | × |
| Mean (SD) | XX.X (XX.XX) |
| Median | XXX |
| Min, Max | XX, XX |

Programming note: Repeat for Week 8 Predose & Postdose

Note: Subjects are summarized by treatment received. Reference Listing: 16.2.5.6

Statistical Analysis Plan, Sponsor Arcutis, Inc. Protocol Number ARQ-154-203 PCN Number ARCU210100



| ) |
|---|
| i |

| Roflumilast Foam 0.3%<br>(N=XX) | XX XXX<br>XXXXX<br>XX, XXX | XX | XX |
|---|---|---|---|
| Parameter: XXXXXXXX<br>Study Visit<br>Statistic | Baseline<br>n<br>Mean (SD)<br>Median<br>Min, Max | Week 4<br>n<br>Mean (SD)<br>Median<br>Min, Max | Week 8<br>n Mean (SD)<br>Median<br>Min, Max |

Programming note: Continue for all parameters and repeat for Week 8

Note: Subjects are summarized by treatment received. Reference Listing: 16.2.5.6



## 14.3. Planned Listing Shells

Listing 16.2.1.1 Subject Disposition All Subjects

| Date of Last Visit Reason for Early Date of Death/ due to COVID-19 in Extension (Study Day) Termination Cause of Death Disruption Study? | XX Xx | XX Xes | ON XX | | XXXXXX; date of last DDMMMYYYY XX No |
|---|---|---|---|---|---|
| Date of Completion/ Early Termination Date of Last Visi (Study Day) (Study Day) | DDMMMYYYY<br>(XX) | DDMMMYYYY<br>(XX) | DDMMMYYYY<br>(XX) | | DDMMMYYYY DDMMMYYYYY |
| Did Subject<br>Complete<br>Study? | Yes | Yes | Yes | Ongoing | o <sub>N</sub> |
| Randomized<br>Treatment | XXXX | XXXXX | XXXXX | XXXXX | XXXXX |
| Subject<br>ID | XXX | XXX | XXX | ××× | ××× |

Abbreviation: COVID-19 = novel coronavirus disease. Note: Study day is calculated relative to the date of first application of study drug.

Programming Note: If reason for early termination is Other, concatenate the specify text as follows: "Other: XXXXXXXXXX". If reason for early termination is lost to follow-up, concatenate with date of last contact as follows: "Lost to follow-up; date of last contact: DDMMMYYYY".



Listing 16.2.1.2 Subject Visits All Subjects

| Subject ID | Treatment<br>Received | Was Visit<br>Performed? | Visit | Visit Date<br>(Study Day) | If Visit not Performed,<br>COVID-19 Disruption<br>Contributed to Missed Visit |
|---|---|---|---|---|---|
| XXXXX | XXXXXX | Yes | XXXXXX | DDMMMYYYY (XX) | |
| | | Yes | XXXXXX | DDMMMYYYY (XX) | |
| | | Yes | XXXXXXXXX | DDMMMYYYY (XX) | |
| | | o<br>N | XXXXXXX | | Yes |
| XXXXXX | XXXXXX | Yes | XXXXXX | DDMMMYYYY (XX) | |
| | | Yes | XXXXXX | DDMMMYYYY (XX) | |

Abbreviation: COVID-19 = novel coronavirus disease. Note: Study day is calculated relative to the date of first application of study drug.



Inclusion and Exclusion Criteria Listing 16.2.2.1 All Subjects

| | | Subject Screen Failed | | Date/Tim | Date/Time (Study Day) of: | All Inclusion | Any<br>Exclusion |
|---|---|---|---|---|---|---|---|
| Subject ID | Was Subject<br>Rescreened? | due to COVID-19<br>Disruption | Randomized<br>Treatment | Screening | Informed Consent | Criteria Met?<br>[1] | Criteria Met?<br>[2] |
| XXXXX | × | × | XXXXX | DDMMMYYYY<br>(-X) | DDMMMYYYY/hh:mm<br>(-X) | Yes | o<br>Z |
| XXXXXX | × | × | | DDMMMYYYY | DDMMYYYY/hh:mm | No: 06, 10 | <sub>N</sub> |
| XXXXXX | × | × | | DDMMMYYYY | DDMMMYYYY/hh:mm | No: 01 | 9<br>N |
| XXXXXX | XXX | XXX | XXXXX | DDMMMYYYYY<br>(-X) | DDMMMYYYY/hh:mm<br>(-X) | Yes | Yes: 02 |
| XXXXXX | × | × | XXXXX | DDMMMYYYYY<br>(-X) | DDMIMMYYYY<br>(-X) | Yes | o<br>Z |
| XXXXX | × | × | XXXXX | DDMMMYYYY<br>(-X) | DDMMMYYYY (X-) | Yes | N<br>N |

Abbreviation: COVID-19 = novel coronavirus disease.

Note: If a subject is a rescreen, the latest date of screening and informed consent are presented.
[1] 01 = Participants legally competent to sign and give informed consent, 06 = Overall Assessment of Erythema and Overall Assessment of Scaling scores of Moderate ('2') at Baseline; 10 = Subjects are considered reliable and capable of adhering to the Protocol and visit schedule according to the Investigator judgment. [2] 02 = Planned excessive exposure of treated area(s) to either natural or artificial sunlight, tanning bed or other LED. Programming note: If more than 1 inclusion or exclusion criterion number exists, concatenate with a comma as shown above. Decode any relevant criteria in the footnotes as shown in the example. If no criteria are present for a column, remove the [1] and/or [2] from the column header. Time is only collected for informed consent. If time is missing, display as shown in the shell. If subject rescreens, populate the latest date of screening and informed consent.

Statistical Analysis Plan, Sponsor Arcutis, Inc. Protocol Number ARQ-154-203 PCN Number ARCU210100



Listing 16.2.2.2 Protocol Deviations All Subjects

| Subject<br>ID | Treatment<br>Received | Subject Treatment D Received Event Type | Description | COVID-19 Related | COVID-19 Infection |
|---|---|---|---|---|---|
| XXXXX | xxxxx xxxxx | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXX | | |
| XXXXX | XXXXX | XXXXXXXXXX XXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXX | XXXXXX |
| XXXXXX | XXXXX | XXXXXXXXXXX XXXXXX XXXXXX | XXXXX XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | ××××× | ××××× |

Abbreviation: COVID-19 = novel coronavirus disease.

Programming note: the structure of this listing may change depending on the information in the protocol deviations file.



Listing 16.2.3 Analysis Populations All Subjects

| | PK Primary Reason(s) for [6] Exclusion | | | Subject did not receive at least 1 dose of IP. |
|---|---|---|---|---|
| | 4 PK<br>[6] | | | |
| | 12 PRU4<br>[5] | Yes | Yes | 8 |
| | PRU2<br>[4] | Yes | Yes | o<br>N |
| | [3] | | | |
| | mITT ITT [2] | Yes | Yes | Š |
| | Safety<br>[1] | Yes | Yes | o<br>N |
| | Stratification<br>ID | XXXX | XXXX | |
| Randomization | Number | × | ×× | |
| Ra | Date/Time | DDMMMYYY/<br>hh:mm | DDMMMYYY/<br>hh:mm | |
| | Subject Treatment Randomized ID Received Treatment | XXXXX | XXXX | |
| | Treatment<br>Received | XXXXXX | XXXXXX | XXXXX |
| | Subject<br>ID | ×× | ×× | ××× |

Abbreviations: COVID-19 = novel coronavirus disease; ITT = intent-to-treat; IGA = investigator global assessment; IP = investigational product; mITT = modified intent-to-treat; NA = not applicable; WI-NRS = Worst Itch – Numeric Rating Scale. Stratification ID is baseline severity of IGA. If stratification ID = 1 then IGA = Moderate; if 2 then IGA = Severe.

[1] The Safety Population includes all subjects who are enrolled and received at least 1 confirmed dose of IP.

[2] The mITT population includes all subjects with the exception of subjects who missed the week 8 IGA assessment specifically due to COVID-19 disruption.

[3] The ITT population includes all subjects who are randomized.

[4] The PRU2 population is a subset of the ITT population and includes subjects with WI-NRS pruritus score ≥ 2 at Baseline. This population will be used for the analysis of achievement of a 2-point reduction in WI-NRS pruritus score as compared to Baseline.

[5] The PRU4 population is a subset of the ITT population and includes subjects with WI-NRS pruritus score ≥ 4 at Baseline. This population will be used for the analysis of achievement of a 4-point reduction in WI-NRS pruritus score as compared to Baseline.

[6] The PK population will include all subjects receiving the active drug with sufficient plasma concentrations of roflumilast to define a profile, as determined by the pharmacokineticist. This population will be used for analyses of PK parameters.



Listing 16.2.4.1 Demographics and Baseline Characteristics All Subjects

| | | | Child-Bearing<br>Potential? If | Year | Age | | | Was<br>Photography | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject | Treatment | | Yes, Specify | o | (years) | | | Consent | Photography | Height | Weight | BSA |
| | Received | Sex | Contraception | Birth | Ξ | Ethnicity | Race | Obtained? | Consent Date | (cm) | (kg) | (%) |
| XXXXX | XXXXX | ××× | 8<br>8 | *** | × | XXXXXXX | XXXXXX | Yes | DDMMMYYYY | × | × | × |
| XXXXX | XXXXX | XXXXX | N <sub>o</sub> | *** | × | XXXXXXX | XXXXX | Yes | DDMMMYYYY | ×× | × | × |
| XXXXX | XXXXX | ××× | | *** | × | XXXXXX | XXXXX | o<br>N | | ×× | × | × |
| XXXXX | XXXXX | ××× | | *** | × | XXXXXX | XXXX | Yes | DDMMMYYYY | × | × | ×× |
| XXXXX | XXXXX | XXXXX | No | *** | × | XXXXXX | XXXXX | Yes | DDMMMYYYY | × | × | × |
| XXXXX | XXXXX | ×× | Yes: | *** | × | XXXXX | XXXXX | × | DDMMMYYYY | × | × | × |

Abbreviation: BSA = body surface area.

Note: Weight, and BSA are the values at Screening. Height is collected at Baseline Day 0.

[1] Age at Screening.

Programming Note: If subject has multiple races, concatenate them. If child-bearing potential is Yes, concatenate type of contraception with "" as shown in the shell.





| Other Medical History Conditions | Start Date (Study Day)/<br>End Date (Study Day) | DDMMMYYYY $(X)$ / DDMMMYYYY $(X)$ | DDMMMYYYY (X)/ DDMMMYYYY (X)/ DDMMMYYYY (X)/ | DDMMMYYYY (X)/<br>Ongoing |
|---|---|---|---|---|
| Other Medica | System Organ Class/<br>Preferred Term/<br>Verbatim Term | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | ************************************** |
| | Type of History | Topical Corticosteroids: Yes/<br>Topical Antifungals: No/<br>Facial Involvement: Yes | | Topical Corticosteroids: Yes/<br>Topical Antifungals: Yes/<br>Facial Involvement: Yes |
| | Treatment<br>Received | ××××× | | XXXXX |
| | Subject ID | XXXXX | | XXXXX |

Abbreviation: MedDRA = Medical Dictionary for Regulatory Activities.

Note: Study day is calculated relative to the date of first application of study drug. Medical history was coded using MedDRA version 23.0.

Only subjects with medical history recorded are listed.

Programming note: SOC & PT text should be presented as is from the dataset.



Listing 16.2.5.1 Study Drug Application at the Study Site All Subjects

| Kit Number/<br>Can ID | /XXX | *** | ××× | × | XXXX | { | XXXX |
|---|---|---|---|---|---|---|---|
| Reason Pre- and/or<br>Post-Application<br>Can Weight<br>Measurement not<br>Performed | | | | | | | XXXXXXXXXXX |
| Applied<br>Dose<br>(g) | × | ×× | × | | × | ××× | |
| Post-Application<br>Can Weight (g)<br>Measurement | × | XX. | × | | × | × | Not Done |
| Pre-Application<br>Can Weight (g)<br>Measurement | × | ××× | × | | × | × | × |
| Date/Time of<br>Application | DDMMMYYYY/HH:MM | DDMMMYYYY/HH:MM | DDMMMYYYY/HH:MM | | DDMMMYYYY/HH:MM | DDMMMYYYY/HH:MM | DDMMMYYYY/HH:MM |
| Study<br>Visit | XXXXX | XXXXX | XXXXXX | XXXXX | XXXXX | XXXXXX | XXXXX |
| Was Study<br>Drug<br>Application<br>Performed at<br>Study Site? | Yes | | | No: XXXXXX | Yes | | |
| Treatment<br>Received | XXXXXX Yes | | | | XXXXXX Yes | | |
| Subject<br>ID | ××× | | | | XXX | | |

Programming note: For Pre & Post-Application Can Weight Measurement columns, if the weight measurement is not performed, set the value to be "Not Done". If drug not administered, concatenate reason as shown in shell.





Listing 16.2.5.2 Cans All Subjects

| d Return<br>Weight (g) | (x) XXX | XXXX (X) | ON (X) | |
|---|---|---|---|---|
| Date Returned<br>(Study Day) | DDMMMYYYY (X) | DDMMMYYYY (X) | DDMMMYYYY (X) | |
| Dispense Can Returned?<br>Weight (g) Reason if No | Yes | Yes | Yes | No: XXXXX |
| | × | ×× | Q. | |
| Can Dispensed? Date Dispensed<br>Reason if No (Study Day) | DDMMMYYYY (X) | DDMMMYYYY (X) | DDMMMYYYY (X) | |
| Can Dispensed?<br>Reason if No | Yes | Yes | Yes | No: XXXXX |
| Treatment Kit Number/<br>Received Can ID | XXXXX | ×××× | ××××× | XXXX |
| | XXXXXX | | | XXXXX |
| Subject ID | XXXXX | | | XXXX |

Abbreviation: ND = not done. Note: Study day is calculated relative to the date of first application of study drug.

Programming note: within subject, sort by dispense date, return date, kit number and CAN ID.





Listing 16.2.5.3 Diary Dispensation All Subjects

| irned<br>ay) | &&<br>}; | | |
|---|---|---|---|
| Date Returned<br>(Study Day) | DDMMMYYYY(X) $DDMMMYYYY(X)$ | | |
| Reason Diary<br>not Returned | | XXXXXXXXX | XXXXXXXX |
| Diary Returned Reason Diary and Reviewed? not Returned | Yes | N <sub>O</sub> | N <sub>O</sub> |
| Diary<br>Returned<br>Visit | ×××××× | XXXXXX | XXXXX |
| Date Dispensed<br>(Study Day) | DDMMMYYYY (X)<br>DDMMMYYYY (X) | DDMMMYYYY (X) | |
| Diary<br>Dispensed? | Yes | Yes | o<br>N |
| Diary<br>Dispensation<br>Visit | XXXXX | XXXXXX | XXXX |
| Treatment<br>Received | XXXXX | | XXXXXX |
| Subject ID | XXXX | | XXXX |

Note: Study day is calculated relative to the date of first application of study drug.



Listing 16.2.5.4 Compliance (CRF) All Subjects

| Overall Was Subject Retrained if not Check (Study Day) Compliance [1] Compliance [2] Compliant with Medication | | ×× |
|---|---|---|
| Overall<br>Compliance [2] | %<br>X:X | %X:XX |
| Compliance [1] | % % % X X X X X X X X X X X X X X X X X | % |
| Date of Compliance<br>Check (Study Day) | DDMMMYYYY (X)<br>DDMMMYYYY (X)<br>DDMMMYYYY (X) | DDMMMYYYY (X)<br>DDMMMYYYY (X) |
| Subject Compliant with<br>Medication? | *** | *** |
| Study<br>Visit | ×××××<br>××××××<br>××××××××××××××××××××××××× | ×××××<br>××××××<br>××××××××××××××××××××××××× |
| Treatment<br>Received | XXXXX | ××××× |
| Subject ID | ××××× | XXXXX |

Abbreviations: IP = investigational product; CRF = case report form.

Note: Study day is calculated relative to the date of first application of study drug.

[1]This data comes from CRF page, unless otherwise specified.

[2] Overall compliance will be calculated based on number of applications divided by the expected number of IP applications for each subject. Number of expected IP applications is calculated as number of days between first and last application of IP (last treatment date - first treatment date + 1). Number of IP applications is calculated as number of expected IP applications as collected in the CRF.

Programming note: Populate overall compliance only for the first visit.





| Miss | isit Date of Missed Dose COVID-19 (Study Day) Disruption? Reason for Missed Dose | DDMMMYYYY (X) | KXXX DDMMMYYYY (X) No XXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
|---|---|---|---|---|---|
| Study | Visit | XXXXXX | XXXXXX | XXXXX | XXXXXX |
| | Treatment<br>Received | XXXXX | | XXXXXX | XXXXX |
| | Subject ID | XXXXXX | | XXXXXX | XXXXX |

Abbreviation: COVID-19 = novel coronavirus disease. Note: Study day is calculated relative to the date of first application of study drug.

Programming note: Only subjects with missed doses should be presented in this listing.





Listing 16.2.5.6 Pharmacokinetic Blood Collection PK Population

Abbreviations: BLQ = Below the limit of quantification; PK = pharmacokinetic. Note: Study day is calculated relative to the date of first application of study drug.

Statistical Analysis Plan, Sponsor Arcutis, Inc. Protocol Number ARQ-154-203 PCN Number ARCU210100



Listing 16.2.5.7 Pharmacokinetic Calculated Parameters PK Population

| * | Study Visit (h | AUC₀₊<br>h*ng/mL) | AUC <sub>teu</sub><br>(h*ng/mL) | T <sub>max</sub><br>(h) | T <sub>lag</sub><br>(h) | T <sub>last</sub><br>(h) | C <sub>max</sub><br>(ng/mL) | C <sub>min</sub><br>(ng/mL) |
|---|---|---|---|---|---|---|---|---|
| * | | × | × | × | × | × | × | × |
| × | | × | × | × | × | × | × | × |
| × × × × × | | × | × | × | × | × | × | × |
| | | × | × | × | × | × | × | × |

Abbreviation: PK = pharmacokinetic.

Programming note: The above parameters are expected. However the final parameters provided by the pharmacokineticist will be listed and may be different than shown.



Listing 16.2.6.1 Investigator Global Assessment (IGA) All Subjects

| Subject<br>ID | Was<br>Assessment<br>Subject Randomized Completed?<br>ID Treatment Reason if Nc | Was<br>Assessment<br>Completed?<br>Reason if No | If Visit Performed, COVID-19 Disruption Contributed to Delay in Assessment | If Visit not<br>Performed,<br>COVID-19<br>Disruption<br>Contributed to<br>Missed<br>Assessment | Study<br>Visit | Date/Time of<br>Assessment<br>(Study Day) | Result | Result Text Result | Change from<br>Baseline | IGA<br>Success<br>[1] | IGA Success<br>2-grade<br>Improvement<br>[2] |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX | XXXXX | Yes | °N | | XXX | DDMMMYYYY/hh:mm | × | XXXXXX | | | |
| | | Yes | o<br>N | | XXX | (X)<br>DDMMYYYY/hh:mm | × | XXXXXX | × | o<br>N | |
| | | Yes | No | | XXX | DDMMMYYYY/hh:mm | × | XXXXXX | × | No | |
| | | Yes | o<br>N | | ×× | (X)<br>DDMMMYYYY/hh:mm<br>(X) | × | ××××× | × | Yes | |
| ××× | XXXXXX | Yes | °N | | ×× | DDMMMYYYY/hh:mm | × | XXXXXX | | | |
| | | No:<br>XXXXXXXX | | Yes | ×× | ₹ | | | | | |

Abbreviation: COVID-19 = novel coronavirus disease.

Note: Study day is calculated relative to the date of first application of study drug. Baseline is the last non-missing measurement taken on or before the day of first application of study drug. Change from baseline is calculated as Result – Baseline.

[1] IGA success ("Yes") is defined as an IGA score of "Clear" or "Almost Clear" plus a ≥2-grade improvement from baseline at Weeks 2, 4, 8, and 9; "No" otherwise.

[2] IGA success 2-grade improvement ("Yes") is defined as a 2-grade improvement from baseline; "No" otherwise.

Programming note: Concatenate reason not done as shown in the shell.



Listing 16.2.6.2 Overall Assessment of Erythema All Subjects

| Subject<br>ID | Subject Randomized<br>ID Treatment | Was<br>Assessment<br>Completed?<br>Reason if No | If Visit Perfomed, COVID-19 Disruption Contributed to Delay in Assessment | If Visit not<br>Performed,<br>COVID-19<br>Disruption<br>Contributed<br>to Missed<br>Assessment | Study<br>Visit | Date/Time of<br>Assessment<br>(Study Day) | Result | Change<br>from<br>Baseline | Erythema<br>Success<br>(0-1, >=<br>2-grade<br>Improve) [1] | Erythema<br>Success (0-1<br>Score) [2] | Erythema<br>Success<br>(0 Score)<br>[3] |
|---|---|---|---|---|---|---|---|---|---|---|---|
| ×× | XXXX | Yes | o<br>N | | × | DDMMMYYYY/hh:mm (X) | XXXX = X | | | | |
| | | | No | | × | DDMMMYYYY/hh:mm | X = X | × | o<br>N | N <sub>o</sub> | No |
| | | | °N<br>O | | × | DDMMMYYYY/hh:mm | XXXX = X | ×× | Yes | Yes | Yes |
| | | | o <sub>N</sub> | | × | DDMMMYYYY/hh:mm<br>(X) | XXXX = X | × | o<br>N | <u>0</u> | o<br>N |
| XX | XXXXX | Yes | oN | | × | DDMMMYYYY/hh:mm | XXXX = X | × | | | |
| | | No: XXXXXX | | Yes | × | DDMMMYYY/hh:mm<br>(X) | | | | | |

Abbreviation: COVID-19 = novel coronavirus disease.

Note: Study day is calculated relative to the date of first application of study drug. Baseline is the last non-missing measurement taken on or before the day of first application of study drug. Change from baseline is calculated as Result – Baseline.

Programming note: Concatenate reason not done as shown in the shell.

<sup>[1]</sup> Erythema success (0-1, >= 2-grade Improve) ("Yes") is defined as an Erythema score of "0" or "1" PLUS a 2-grade improvement from Baseline at Weeks 2, 4, 8, and 9; "No" otherwise. [2] Erythema success (0-1 Score) ("Yes") is defined as an Erythema score of "0" at Weeks 2, 4, and 8; "No" otherwise. [3] Erythema success (0 Score) ("Yes") is defined as an Erythema score of "0" at Weeks 2, 4, and 8; "No" otherwise.



Listing 16.2.6.3 Overall Assessment of Scaling All Subjects

(Programming note: Same as shell 16.2.6.2; Update any instances of Erythema in the header, body and footnotes to Scaling)



Listing 16.2.6.4 Worst Itch Numerical Rating Scale (WI-NRS) All Subjects

| WI-NRS<br>Success<br>(baseline ≥<br>2)<br>[2] | | Yes | Yes | Yes | | |
|---|---|---|---|---|---|---|
| WI-NRS<br>Success<br>(baseline ≥<br>4) | | Yes | Yes | Yes | | |
| Change<br>from<br>Baseline | | × | × | × | | |
| Result | × | × | × | × | × | |
| Date/Time of<br>Assessment<br>(Study Day) | DDMMYYYYY/hh:mm | DDMMMYYYY/hh:mm | DDMMMYYYY/hh:mm | DDMMMYYYY/hh:mm<br>(X) | DDMMYYYYY/hh:mm | DDMMMYYYYY/hh:mm<br>(X) |
| Study<br>Visit | XX | ×× | ×× | × | ×× | × |
| If Visit not<br>Performed,<br>COVID-19<br>Disruption<br>Contributed<br>to Missed<br>Assessment | | | | | | Yes |
| If Visit Performed, COVID-19 Disruption Contributed to Delay in Assessment/ Telemedicine | o<br>N | No | No | oN | o<br>N | Yes/<br>Yes |
| Was<br>Assessment<br>Completed?<br>Reason if No | Yes | Yes | Yes | Yes | Yes | No: XXXXXX |
| Randomized<br>Treatment | XXXXXX | | | | XXXXX | |
| Subject ID | XXXXXX | | | | XXXXX | |

Abbreviation: COVID-19 = novel coronavirus disease.

Note: Study day is calculated relative to the date of first application of study drug. Subjects rate the intensity of their itch on an 11-point scale ranging from 0 (no itch) to 10 (worst itch imaginable). Higher score indicates greater itch intensity. Baseline is the last non-missing measurement taken before the first application of study drug. Change from

baseline is calculated as Result – Baseline. [1] In subjects with a baseline WI-NRS pruritus score of ≥4, achievement of a ≥4-point improvement from baseline in WI-NRS pruritus score at Weeks 2, 4, and 8. [2] In subjects with a baseline WI-NRS pruritus score of ≥2, achievement of a ≥2-point improvement from baseline in WI-NRS pruritus score at Weeks 2, 4, and 8.

Programming note: Concatenate reason not done as shown in the shell.



Listing 16.2.6.5 All Subjects Scalpdex

| Change<br>from<br>Baseline | |
|---|---|
| Text Result | Never Rarely Sometimes Often All the time Never Rarely Sometimes Often All the time All the time |
| Result | - 0040-004 0 - XXXX |
| Question [1] | DDMMMYYYYY Q1. My scalp condition makes me feel depressed Q2. My scalp itches Q3. My scalp itches Q4. I am ashamed of my scalp condition Q5. I am embarrassed by my scalp condition Q6. I am humiliated by my scalp condition Q7. My scalp condition bleeds Q8. I am annoyed by my scalp condition Q7. My scalp condition Q9. I am bothered by the appearance of my scalp condition Q10. My scalp condition makes me feel self-condition Q1. I am bothered that my scalp condition is incurable Programming note: Continue for all questions. Emotioning Scale [2] Symptoms Scale [3] Functioning Scale [4] |
| Date/Time of<br>Assessment<br>(Study Day) | DDMMMYYYY/ hh:mm (XX) rogramming note |
| Study<br>Visit | ×× |
| COVID-19<br>Disruption<br>Contributed<br>to Missed<br>Assessment | <u>0</u> |
| COVID-19 Disruption Contributed to Delay Assessment/ Telemedicine | <u>o</u> 2 |
| Assessment<br>Completed?<br>Reason if No | se X |
| Randomized<br>Treatment | XXXXXX |
| Subject<br>ID | × |

Abbreviation: COVID-19 = novel coronavirus disease.

Higher score indicates greater itch intensity. Baseline is the last non-missing measurement taken on or before the day of first application of study drug. Change from baseline is calculated as Result - Baseline. Scalpdex is rated on a 1 to 5 scale which will be transformed to 0 to 100 Scale where 1=0; 2=25; 3=50; 4=75; 5=100. This transformed score is used to calculate scale scores. Q refers to Note: Study day is calculated relative to the date of first application of study drug. Subjects rate the intensity of their itch on an 11-point scale ranging from 0 (no itch) to 10 (worst itch imaginable). question number.

i) These questions are based on the "How often during the past 4 weeks do these statements describe you?" prompt. [2] Emotions Scale is calculated as average of (Q2, Q4, Q5, Q6, Q7, Q9, Q10, Q11, Q12, Q14, Q16, Q20, Q20, Q22) after transforming to 0 to 100 scale as mentioned above. Q19 will be reverse scored i.e., 1=100, 2=75; 3=50; 4=25; 5=0.

[3] Symptoms Scale is calculated as average of (Q1, Q3, Q8) after transforming to 0 to 100 scale as mentioned above. [4] Functioning Scale is calculated as average of (Q13, Q15, Q18, Q21, Q23) after transforming to 0 to 100 scale as mentioned above. [5] Total Score is calculated as mean of all 23 questions using the transformed scale. Q18 will be reverse scored as indicated in [2].



Listing 16.2.6.6 Dermatology Life Quality Index (DLQI) All Subjects

| Change<br>from<br>Baseline | | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Text<br>Result | Not at all | Very<br>much | Very<br>much | Verv | much | A lot | o li⊞lo | | Yes | | | Not | relevant | Not | relevant | Very | much | | | |
| Result | 0 | ო | ო | ო | | 7 | - | - | က | | | 0 | | 0 | | က | | | 9 | <u>o</u> |
| Question | 1. Over the last week, how itchy, sore, painful or stinging has your skin been? | <ol> <li>Over the last week, how embarrassed or<br/>self conscious have you been because of<br/>your skin?</li> </ol> | <ol><li>Over the last week, how much has your<br/>skin interfered with you going shopping or</li></ol> | looking after your home or garden? 4. Over the last week, how much has your | skin influenced the clothes you wear? | 5. Over the last week, how much has your | skin affected any social or leisure activities? | skin made it difficult for you to do any sport? | 7. Over the last week, has your skin | prevented you from working or studying? If "No" over the last week how much has your | skin been a problem at work or studying? | 8. Over the last week, how much has your | skin created problems with your partner or any of your close friends or relatives? | 9. Over the last week, how much has your | skin caused any sexual difficulties? | 10. Over the last week, how much of a | problem has the treatment for your skin been, | for example by making your home messy, or | by taking up time :<br>Total Socia [4] | lotal ocore [1] |
| Date/Time of<br>Assessment<br>(Study Day) | DDMMMYYYY/<br>hh:mm (XX) | | | | | | | | | | | | | | | | | | | |
| If Visit not Performed,<br>COVID-19 Disruption<br>Contributed to Missed<br>Assessment | o <sub>N</sub> | | | | | | | | | | | | | | | | | | | |
| If Visit Performed,<br>COVID-19 Disruption<br>Contributed to Delay<br>in Assessment/<br>Telemedicine | N <sub>O</sub> | | | | | | | | | | | | | | | | | | | |
| Assessment<br>Completed?<br>Reason if No | Yes | | | | | | | | | | | | | | | | | | | |
| Study<br>Visit | XX | | | | | | | | | | | | | | | | | | | |
| Randomized<br>Treatment | ××× | | | | | | | | | | | | | | | | | | | |
| Subject<br>ID | ×× | | | | | | | | | | | | | | | | | | | |

Abbreviation: COVID-19 = novel coronavirus disease.

Note: Study day is calculated relative to the date of the first application of study drug.

[1] The total score ranges between 0-30 and calculated as sum of all the 10 questions at each visit. If 1 item is missing, it is scored as 0 for that item. If 2 or more items are missing, the score should not be calculated.







Listing 16.2.6.7 Body Surface Area (BSA) including Scalp All Subjects

| Result | × | × | × | ××× | ××× | ××× | ××× | ××× | %XXX | %XXX |
|---|---|---|---|---|---|---|---|---|---|---|
| Test | Coverage Area (Head) | Coverage Area (Lower Limbs) | Coverage Area (Upper Limbs) | Coverage Area (Trunk) | Area Unaffected (Head) | Area Unaffected (Lower Limbs) | Area Unaffected (Upper Limbs) | Area Unaffected (Trunk) | BSA Result [1] | BSA CRF [2] |
| Date/Time of<br>Assessment<br>(Study Day) | DDMMMYYYY/<br>hh:mm (XX) | | | | | | | | | |
| Study<br>Visit | XXX | | | | | | | | | |
| If Visit not Performed,<br>COVID-19 Disruption<br>Contributed to Missed<br>Assessment | × | | | | | | | | | |
| If Visit Performed, Assessment COVID-19 Disruption Performed? Contributed to Delay Reason if No in Assessment | × | | | | | | | | | |
| | ×× | | | | | | | | | |
| Subject Randomized<br>ID Treatment | XXX | | | | | | | | | |
| Subject<br>ID | XXX | | | | | | | | | |

Abbreviation: COVID-19 = novel coronavirus disease.

Note: Study day is calculated relative to the date of the first application of study drug.

[1] BSA result is calculated as sum of coverage areas of head, lower limbs, upper limbs and trunk. This is derived in the ERT.

[2] BSA captured in the CRF data.



Adverse Events Listing 16.2.7.1 All Subjects

| o Study | | | |
|---|---|---|---|
| AE Lead to<br>D/C? | × | × | × |
| Serious?/ AE Lead to Study<br>Criteria Met D/C? | × | × | XXXXXX |
| Outcome/<br>/ Action Taken/ Serious?/ AE Le<br>Other Action Taken Criteria Met D/C? | /xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | /xxxxxxxx/<br>/xxxxxxxx/ | /xxxxxxxxx/<br>/xxxxxxxxxxx/ |
| CTCAE Toxicity Grade.<br>Relationship | /xxxxxxxxx | ************************************** | /xxxxxxxxx |
| Outcome/ Start Date/Time (Study Day)/ CTCAE Toxicity Grade/ Action Taken/ End Date/Time (Study Day) Relationship Other Action | DDMMMYYYYY/hh:mm (X)/<br>DDMMMYYYYY/ hh:mm (X) | DDMMYYYY/ hh:mm (X)/<br>DDMONYYYY/ hh:mm (X) | DDMONYYYY/ hh:mm (X)/<br>Ongoing |
| System Organ Class/<br>Preferred Term/<br>Verbatim Term | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| TEAE? | × | × | × |
| Subject Treatment<br>ID Received TEAE? | XXXXX XXXX | XXXXX | |
| Subject<br>ID | XXX | XXXX | |

Abbreviations: COVID-19 = novel coronavirus disease; CTCAE = common terminology criteria for adverse events; D/C = discontinue; IP = investigational product; MedDRA = Medical Dictionary for Regulatory Activities; TEAE = Treatment emergent adverse event.

Note: Study day is calculated relative to the date of first application of study drug. AEs were coded using MedDRA version 23.0. All AEs that occur after the date/time of first application of IP will be considered TEAEs.

Programming note: If time missing, display "- -;- -". If Serious? is Yes, concatenate all serious criteria marked as Yes with a semicolon. "Other Action Taken" will be either None, Concomitant Medication, Non-drug Therapy, Hospitalization or Prolongation of Hospitalization, Discontinued Study or Other; if specify text is needed, concatenate "Concomitant Medication:" or "Other:" with the text. If no events meet the criteria for display, present "No events are reported." SOC & PT text should be presented as is from the dataset.




Listing 16.2.8.1.1 Clinical Laboratory Data: Clinical Chemistry All Subjects

| Subject<br>ID | Treatment<br>Received | Parameter (unit) | Study<br>Visit | Date/Time of<br>Assessment<br>(Study Day) | Standard<br>Results | Reference<br>Range<br>[1] | Reference<br>Range<br>Flag | Result<br>Interpretation;<br>Specify CS<br>Finding | Accession | Comments/<br>Reason not Done |
|---|---|---|---|---|---|---|---|---|---|---|
| | xxxxx xxxxx | Alanine | XXXX | DDMMMYYYY/hh:mm | × | XX - XX | High | Normal | XXXXX | |
| | | Ammodansierase (U/L) | ×××× | DDMMMYYYY/hh:mm | × | XX - XX | | Abnormal, | XXX | |
| | | | XXXX | DDMMYYYYY/hh:mm | × | XX – XX | Low | Normal | XXXXX | |
| | | | XXXX | DDMMMYYYY/hh:mm | × | XX - XX | | Normal | XXXXX | |
| | | | XXXX | DDMMMYYYY/hh:mm<br>(XX) | × | XX - XX | | Abnormal, CS;<br>XXXXXXX | XXXX | |
| | | Alkaline | XXXX | DDMMMYYYY/hh:mm | × | XX – XX | Low | XXXXX | XXXXX | |
| | | Pnospnatase (U/L) | XXXX | DDMMYYYYY/hh:mm | × | XX - XX | | XXXXX | XXXX | |
| | | | XXXX<br>XXXX | DDMMMYYYY/hh:mm<br>(XX) | N X | XX - XX | High | XXXXX | XXXX | XXXXXX |

Abbreviations: CS = clinically significant; NCS = not clinically significant; ND = not done.

Note: Study day is calculated relative to the date of first application of study drug. Time is collected in the ACM.

[1] Reference range is used to identify potentially clinically significant laboratory values.





Listing 16.2.8.1.2 Clinical Laboratory Data: Hematology All Subjects

(Same shell as Listing 16.2.8.1.1)

Listing 16.2.8.1.3 Clinical Laboratory Data: Urinalysis All Subjects

(Same shell as Listing 16.2.8.1.1)





| | | Was Prednancy | | | | |
|---|---|---|---|---|---|---|
| | Treatment | Treatment Test Performed? | | | Date/Time Performed | |
| Subject ID | Received | Received Reason if No | Study Visit | Type of Test | (Study Day) | Result |
| XXXX | XXXXX | Yes | XXXXXX | Serum | DDMMMYYYY (XX) | |
| | | | | Urine | DDMMMYYYY/hh:mm (XX) | |
| | | | XXXXXX | Urine | DDMMMYYYY/hh:mm (XX) | XXXXXXXXX |
| XXXXX | XXXXXX | Yes | XXXXXX | Serum | DDMMMYYYY (XX) | XXXXXXXXX |
| | | | | ; | | |
| | | No: XXXXXXXXX | XXXXX | Urine | | |

Note: Study day is calculated relative to the date of first application of study drug.

Programming note: If time missing, display only date.



Listing 16.2.9.1 Investigator Local Tolerability Assessments All Subjects

| Subject<br>ID | Treatment<br>Received | Tolerability<br>Assessment<br>Performed?<br>Reason if No | If Visit<br>Performed,<br>COVID-19<br>Disruption<br>Contributed to<br>Delay in<br>Assessment | If Visit not<br>Performed,<br>COVID-19<br>Disruption<br>Contributed to<br>Missed<br>Assessment | Study Visit | Date/Time of Assessment (Study Day) Dermal Response | Dermal Response | Other Effects |
|---|---|---|---|---|---|---|---|---|
| ××× | XXXXXX | Yes | No | No | XXXXXX | DDMMMYYYY/hh:mm | XXXXXXXX = X | X = XXXXXXXXX |
| | | Yes | No | o <sub>N</sub> | XXXXXX | DDMMMYYYY/hh:mm | XXXXXXXX = X | X = XXXXXXXX |
| | | Yes | o <sub>N</sub> | o <sub>N</sub> | XXXXXX | DDMMMYYYY/hh:mm<br>(XX) | XXXXXXXX = X | XXXXXXXX = X |
| ××× | XXXXXX | Yes | No | o <sub>N</sub> | XXXXXX | DDMMMYYYY/hh:mm | XXXXXXXX = X | XXXXXXXX = X |
| | | Yes | No | o <sub>N</sub> | XXXXXX | DDMMMYYYY/hh:mm | XXXXXXX = X | X = XXXXXXXX |
| | | Yes | o <sub>N</sub> | o <sub>N</sub> | XXXXXX | DDMMMYYYY/hh:mm<br>(XX) | XXXXXXXX = X | XXXXXXXX = X |
| ××× | XXXXXX | Yes | No | o <sub>N</sub> | XXXXXX | DDMMYYYYY/hh:mm | XXXXXXXX = X | XXXXXXXX = X |
| | | Yes | o <sub>N</sub> | o <sub>N</sub> | XXXXXX | DDMMMYYYY/hh:mm | XXXXXXX = X | XXXXXXXX = X |
| | | No: XXXXXXXX | Yes | Yes | XXXXXX | ( <del>\</del> \ <del>\</del> \ | | |

Abbreviations: IP = investigational product; COVID-19 = novel coronavirus disease.

Note: Study day is calculated relative to the date of the first application of study drug. This assessment will be conducted by the investigator prior to the application of IP in the study site.

Programming note: Concatenate reason not done as shown in the shell.



Listing 16.2.9.2 Subject Local Tolerability Assessments All Subjects

| Sensation Following the Application of IP | No sensation | Slight warm, tingling sensation; not | really bouriersonne te Definite warm, tingling sensation that is somewhat bothersome | No sensation | Hot tingling/stinging sensation that has caused definite discomfort | |
|---|---|---|---|---|---|---|
| Grade | 0 = None | 1 = Mild | 2 = Moderate | 0 = None | 3 = Severe | |
| Date/Time of<br>Assessment (Study<br>Day) | DDMMMYYYY/hh:mm | DDMMMYYYY/hh:mm | DDMMMYYYY/hh:mm<br>(XX) | DDMMMYYYY/hh:mm | DDMMMYYYY/hh:mm<br>(XX) | |
| Study<br>Visit | XX | ××× | XXX | × | ××× | XXX |
| If Visit not<br>Performed, COVID-<br>19 Disruption<br>Contributed to<br>Missed Assessment | No<br>N | No | ON | °N | °N | Yes |
| If Visit Performed,<br>COVID-19 Disruption<br>Contributed to Delay<br>in Assessment/<br>Telemedicine | o <sub>N</sub> | No | ON. | O <sub>N</sub> | Yes/<br>Yes | Yes |
| Tolerability<br>Assessment<br>Performed?<br>Reason if No | Yes | Yes | Yes | Yes | Yes | No:<br>XXXXXXX |
| Treatment<br>Received | XXXXXX | | | XXXXX | | |
| Subject<br>ID | ××× | | | XXX | | |

Abbreviations: IP = investigational product; COVID-19 = novel coronavirus disease.

Note: Study day is calculated relative to the date of the first application of study drug. This assessment will be performed at baseline visit 10 to 15 minutes after the application of IP in the study site.

Programming note: Concatenate reason not done as shown in the shell.





Listing 16.2.9.3 Pigmentation Assessment All Subjects

| Result Categorical Result | None | Mild<br>Moderate | Severe |
|---|---|---|---|
| Result | 0 | <del>-</del> ∨ | က |
| Category | Hypopigmentation | Hyperpigmentation<br>Hypopigmentation | Hyperpigmentation |
| Date/Time of<br>Assessment<br>(Study Day) | DDMMMYYYY/hh:mm | DDMMMYYYY/hh:mm | |
| Study | ××× | × | XX |
| If Visit not Performed,<br>COVID-19 Disruption<br>Contributed to Missed<br>Assessment | No | No | Yes |
| If Visit Performed,<br>COVID-19 Disruption<br>Contributed to Delay in<br>Assessment | o <sub>N</sub> | No | Yes |
| Assessment<br>Performed?<br>Reason if No | Yes | Yes | No: XXXXXX |
| Treatment<br>Received | XXXXX | | |
| Subject<br>ID | ××× | | |

Abbreviation: COVID-19 = novel coronavirus disease.

Note: Study day is calculated relative to the date of first application of study drug.

\*\*Programming note: Concatenate reason not done as shown in the shell.



Listing 16.2.9.4.1 Vital Signs All Subjects

| Subject<br>D | Treatment<br>Received | Vital Signs<br>Collected?<br>Reason if No | Study<br>Visit | Date of<br>Assessment<br>(Study Day) | Temp<br>(°C) | Heart<br>Rate<br>(bpm) | Position | Blood Pressure (mmHg) Systolic Diastolic | Blood<br>ure (mmHg)<br>c Diastolic | Height (cm) | BMI<br>(kg/m²) | Abnormal Findings/<br>Clinically Significant/<br>Description of Finding |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | xxxxxx xxxx | Yes | XXXXX | DDMMMYYYY | ×× | × | XXX | × | × | × | × | } |
| | | Yes | ××××× | DDMMMYYYY | × | × | XXXX | × | × | | | ₹ |
| | | No: XXXXXX<br>Yes | XXXX | DDMMMYYYY (X) | × | × | XXXX | × | × | × | × | )<br>)<br>XXX |
| | | | | | | | | | | | | XXXXXX |

Note: Study day is calculated relative to the date of first application of study drug.
[1] BMI is derived as (weight in kg)/[(height in cm/100)²]. Weight is collected at all visits. For visits up to Week 4, baseline day 0 height is used for BMI derivation. Week 8 and Week 9 BMI is derived using Week 8 height.





| Abnormal Findings/<br>Clinically Significant/<br>Description of Finding | | × | XXXXX<br>XXXX |
|---|---|---|---|
| Underlying<br>Reason for<br>Weight Loss | Weight loss<br>was a result of | dieting<br>Other: XXXXX | |
| Weight Loss<br>due to<br>Complications<br>Associated with<br>COVID-19 | No | o<br>Z | |
| Was Weight<br>Loss<br>Intentional? | Yes | Yes | |
| Percent<br>Change in<br>Weight<br>Since<br>Baseline | × | × | |
| Weight<br>(kg) | × | × | |
| Date of<br>Assessment<br>(Study Day) | DDMMMYYYY (X) | DDMMMYYYY (X) | |
| Study<br>Visit | XXXXX | XXXX | ××× |
| Vítal Signs<br>Collected?<br>Reason if No | Yes | Yes | No:<br>XXXXXXX |
| Treatment<br>Received | XXXXXX Yes | | XXXXX |
| Subject<br>ID | XXXXX | | XXXX |

Abbreviation: COVID-19 = novel coronavirus disease. Note: Study day is calculated relative to the date of first application of study drug.

Programming note: If reason for weight loss is "Other", concatenate reason as shown in the shell.



Listing 16.2.9.5 Physical Examination All Subjects

| ficant? | | | | | |
|---|---|---|---|---|---|
| Clinically Significant? | | o<br>Z | | o<br>Z | |
| Abnormal Findings | | XXXXXXX | | XXXXXXX | |
| Result | Normal | Abnormal<br>Normal | Normal | Abnormal<br>Normal | |
| Body System | Skin | Lungs<br>Heart | Skin | Lungs<br>Heart | |
| Date of<br>Assessment<br>(Study Day) | DDMMMYYYY | ( <del>\</del> -) | DDMMMYYYY | ( <del>\</del> -) | |
| Study Visit | XXXXXXX | | XXXXXXX | | XXXXXXX |
| Physical<br>Examination<br>Performed?<br>Reason if No | Yes | | Yes | | No: XXXXXXX |
| Treatment<br>Received | XXXXXXX Yes | | | | |
| Subject ID | XXXXXX | | | | |

Note: Study day is calculated relative to the date of first application of study drug.

Programming note: Concatenate reason not done as shown in the shell.




Listing 16.2.9.6 Medical Photography All Subjects

| Subject ID | Treatment<br>Subject ID Received | Photography<br>Performed? | If Visit Performed,<br>COVID-19 Disruption<br>Contributed to Delay<br>in Assessment | If Visit Performed, If Visit not Performed, COVID-19 Disruption COVID-19 Disruption Contributed to Missed in Assessment Assessment | Study Visit | Date of Assessment<br>(Study Day) |
|---|---|---|---|---|---|---|
| | XXXXX | Yes Yes Yes Yes Yes No: XXXXXXXX | 0 0 0 0 X X X X X X X X X X X X X X X X | No<br>No<br>No<br>Yes | × | DDMMMYYYY (XX) DDMMMYYYY (XX) DDMMMYYYY (XX) DDMMMYYYY (XX) |

Abbreviation: COVID-19 = novel coronavirus disease. Note: Study day is calculated relative to the date of first application of study drug.

Programming note: Concatenate reason not done as shown in the shell.



Listing 16.2.9.7
Prior and Concomitant Medications
All Subjects

| | Subject ID Country Treatment Received | Prior/<br>Concomitant<br>[1] | Indication | ATC Class (Level 4)/<br>Preferred Term/<br>Verbatim Term | Start Date (Study Day)/<br>End Date (Study Day) | Dose (unit) | Route/<br>Frequency |
|---|---|---|---|---|---|---|---|
| XXXXX | | Prior | XXXXXX | /xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | DDMMMYYYY (X)/<br>DDMMMYYYY (X) | (XXX) XXX | /xxxxxxx<br>/xxxxxxx |
| | | Both | XXXXXX | /xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | DDMMMYYYY (X)/<br>Ongoing | (XXX)<br>XXX | )<br>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>>> |
| | | Concomitant | XXXXXX | /xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | DDMMMYYYY $(X)$ / DDMMMYYYY $(X)$ | (XXX) XXX | |

Abbreviations: ATC = anatomic therapeutic chemical; NA = Not applicable; WHO-DDE = World Health Organization-Drug Dictionary Enhanced.

Note: Study day is calculated relative to the date of first application of study drug. Medications were coded using WHO-DDE Global B3 version September 2019.

[1] Prior indicates medication that was started and stopped prior to dosing of study drug. Concomitant indicates medication that started during the treatment period. Both indicates medication that was started prior to dosing of study drug and continued during the treatment period.

Programming note: If Dose unit, Route or Frequency is Other, display other specify text only (ie, do not display "Other: XXXXXX" but just "XXXXXX"). Sort by subject, start date, end date, ATC level 4 & PT. ATC & PT text should be presented as is from the dataset.




Patient Health Questionnaire (PHQ-8) All Subjects Listing 16.2.9.8

| Text Result | Not at all | Several days<br>More than | half the days | Nearly every | day | Not at all | Several days | More than | half the days | Nearly every | day | Moderate<br>depression |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Result | 0 | - 0 | | က | c | 0 | ~ | 2 | | က | | 12 |
| Question [1] | Little interest or pleasure in doing things | <ol> <li>Feeling down, depressed, or hopeless</li> <li>Trouble falling or staving asleep, or</li> </ol> | sleeping too much | 4. Feeling tired or having little energy | | <ol> <li>Poor appetite or overeating</li> </ol> | <ol> <li>Feeling bad about yourself, or that you<br/>are a failure, or have let yourself or your<br/>family down</li> </ol> | 7. Trouble concentrating on things, such | as reading the newspaper or watching television | 8. Moving or speaking so slowly that | other people could have houced. Of the opposite-being so fidgety or restless that you have been moving around a lot more than usual | PHQ8 Total Score [2]<br>Total Score [3] |
| Date/Time of<br>Assessment<br>(Study Day) | DDMMMYYYY/<br>hh:mm (XX) | | | | | | | | | | | |
| Study<br>Visit | ×× | | | | | | | | | | | |
| If Visit not<br>Performed,<br>COVID-19<br>Disruption<br>Contributed to<br>Missed<br>Assessment | N <sub>O</sub> | | | | | | | | | | | |
| If Visit Performed, COVID-19 Disruption Contributed to Delay in Assessment/ Telemedicine | o<br>N | | | | | | | | | | | |
| Assessment<br>Completed?<br>Reason If No | Yes | | | | | | | | | | | |
| Treatment<br>Received | XXXX | | | | | | | | | | | |
| Subject<br>ID | ×× | | | | | | | | | | | |

Abbreviation: COVID-19 = novel coronavirus disease.

## Programming note: Concatenate reason not done as shown in the shell.

Note: Study day is calculated relative to the date of the first application of study drug.

[1] These questions are based on the "Over the last 2 weeks, how often have you been bothered by any of the following problems?" prompt.

[2] Score as collected in the CRF.

[3] The total score is calculated as sum of all the 8 questions. If more than 1 item is missing the total score should not be calculated. If 1 item is missing, the total score is calculated as sum of answered items. If total score ranges between 0-4, it is categorized as None – Minimal depression; 5-9 = Mild depression; 10-14 = Moderate depression; 15-19 = Moderately severe depression; 20-24 = Severe depression.



Listing 16.2.9.9 Columbia-Suicide Severity Rating Scale (C-SSRS) All Subjects

| Result | × | × | | N | | | × | | | × | | × | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | 1 = Less than | once a week | 1 = Fleeting – | few seconds or | minutes | 1 = Easily able to |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Assessment | 1. Wish to be dead | If yes, describe:<br>2. Non-Specific Active Suicidal | Thoughts<br>If was describe: | 3. Active Suicidal Ideation with | Any Methods (not Plan) without | intent to Act<br>If ves. describe: | 4. Active Suicidal Ideation with | Some Intent to Act, without | Specific Plan<br>If ves, describe: | 5. Active Suicidal Ideation with | Specific Plan and Intent If yes, describe: | Most Severe Ideation Type # (1-5) | Description of Ideation | Frequency | | Duration | | | Controllability |
| Category | Suicidal Ideation | | | | | | | | | | | Intensity of Ideation | , | | | | | | |
| If Visit not<br>Performed, COVID-<br>19 Disruption<br>Contributed to<br>Missed<br>Assessment | No | | | | | | | | | | | | | | | | | | |
| If Visit Performed,<br>COVID-19<br>Disruption<br>Contributed to<br>Delay in<br>Assessment/<br>Telemedicine | No | | | | | | | | | | | | | | | | | | |
| Reference<br>Period | Baseline/<br>Screening | ) | | | | | | | | | | | | | | | | | |
| Date/Time of<br>Assessment (Study<br>Day) | DDMMMYYYY/hh:mm<br>(XX) | | | | | | | | | | | | | | | | | | |
| Study Visit | XXXXXX | | | | | | | | | | | | | | | | | | |
| Treatment<br>Received | XXXXXX | | | | | | | | | | | | | | | | | | |
| Subject<br>ID | XXXXX | | | | | | | | | | | | | | | | | | |

Programming note: Reference period will be either Baseline/Screening or Since Last Visit. Display the results following the order of C-SSRS questionnaire for all categories.

control thoughts

Abbreviation: COVID-19 = novel coronavirus disease.

Note: Study day is calculated relative to the date of first application of study drug. Time is collected in the ERT. Assessments that are marked as Not Done are not included in the listing.



## Appendix 1: Premier Research Library of Abbreviations

| Abbreviation | Definition |
|--------------|---------------------------------|
| aCRF | annotated case report form |
| AD | associated documents |
| ADR | adverse drug reactions |
| AE | adverse event |
| AESI | adverse events special interest |
| ANCOVA | analysis of covariance |
| ATC | anatomical therapeutic chemical |
| BLQ | beneath limit of quantification |
| BMI | body mass index |
| BRD | business requirements document |
| BSL | biostatistician lead |



| Abbreviation | Definition |
|--------------|-------------------------------------------------------------|
| CCGs | CRF completion guidelines |
| CD | compact disc |
| CDISC | clinical data interchange standards consortium |
| CEC | central ethics committee |
| CFR | code of federal regulations |
| CI | confidence intervals |
| CIOMS | council for international organizations of medical sciences |
| CIP | clinical investigational plan |
| CM | clinical manager |
| СМН | Cochran Mantel Haenszel |
| CMP | clinical monitoring plan |
| COV | close out visit |
| COVID-19 | Novel coronavirus disease |
| CRA | clinical research associate |



| Abbreviation | Definition |
|--------------|----------------------------------|
| CRF | case report form |
| CRO | contract research organization |
| CS | clinically significant |
| CSM | clinical supply manager |
| CSR | clinical study report |
| CTA | clinical trial administrator |
| CTM | clinical trial manager |
| CTMS | clinical trial management system |
| DB | database |
| DBL | database lock |
| DBP | diastolic blood pressure |
| DCRF | data change request form |
| DDE | drug dispensing error form |
| DEA | drug enforcement administration |



| Abbreviation | Definition |
|--------------|-------------------------------------------|
| DIA | drug information association |
| DIS | data integration specification |
| DLT | dose limiting toxicity |
| DM | data management |
| DMB | data monitoring board |
| DMC | data monitoring committee |
| DML | data management lead |
| DMP | data management plan |
| DNA | deoxyribonucleic acid |
| DOB | date of birth |
| DS | document specialist |
| DSG | drug safety group |
| DSM | drug supply management (drug distributor) |
| DSMB | data safety monitoring board |



| Abbreviation | Definition |
|--------------|------------------------------------------|
| DSP | data safety plan |
| DSUR | development safety update report |
| DTS | data transfer specification |
| DVD | digital video disk |
| EC | ethics committee |
| ECD | edit check and derivation specifications |
| ECG | electrocardiogram |
| eCRF | electronic case report form |
| EDC | electronic data capture |
| EMA | European medicines agency |
| eTMF | electronic trial master file |
| EU | European Union |
| FA | full analysis |
| FDA | food and drug administration |



| Abbreviation | Definition |
|--------------|-------------------------------------------|
| FMP | file management plan |
| FPFV | first patient first visit |
| FPI | first patient in |
| GCP | good clinical practice |
| GMP | good manufacturing practices |
| GPV | global pharmacovigilance |
| HR | heart rate |
| IB | investigator's brochure |
| IC or ICF | informed consent or informed consent form |
| ICH | international council for harmonization |
| ID | identification |
| IDM | independent drug monitoring |
| IEC | independent ethics committee |
| IGA | investigator global assessment |



| Abbreviation | Definition |
|--------------|-----------------------------------------|
| IM | investigator meeting |
| IMV | interim monitoring visit |
| IND | investigational new drug |
| INDSR | investigational new drug safety reports |
| IP | investigational product |
| IRB | institutional review board |
| IRF | inventory release file |
| IRR | infusion related reactions |
| IRT | interactive response technology |
| ISF | investigator site file |
| ITT | intent-to-treat |
| IVRS | interactive voice response system |
| IWRS | interactive web response system |
| IxRS | interactive voice/web response system |



| Abbreviation | Definition |
|--------------|-----------------------------------------------------|
| KPI | key performance indicator |
| LAN | local area network |
| LDM | lead data manager |
| LMS | learning management system |
| ТГОО | lower limit of quantification |
| LPI | last patient in |
| LPLV | last patient last visit |
| LPO | last patient out |
| MAAP | medical affairs and pharmacovigilance teams |
| MAH | marketing authorization holder |
| MedDRA | medical dictionary for regulatory activities |
| MHRA | medicines and healthcare products regulatory agency |
| MM | medical monitor |
| MMP | medical monitoring plan |



| Abbreviation | Definition |
|--------------|---------------------------------------|
| MMRM | mixed effect model repeat measurement |
| MTD | maximum tolerated dose |
| MVR | monitoring visit report |
| Z | number |
| NA | not applicable |
| NCS | non-clinically significant |
| NF | non-functional |
| PD | protocol deviation |
| PDGP | protocol deviation guidance plan |
| PE | physical examination |
| РНО | patient health questionnaire |
| PI | principal investigator |
| PIN | personal identification number |
| PK | pharmacokinetic |




| Abbreviation | Definition |
|--------------|------------------------------------------------|
| PKAP | pharmacokinetic analysis plan |
| PM | project manager |
| PMP | project management plan |
| PP | per-protocol |
| PRIMS | Premier Research information management system |
| PS | project specialist |
| PV | pharmacovigilance |
| PVG | pharmacovigilance group |
| QA | quality assurance |
| QARC | quality assurance, risk and compliance |
| ÓC | quality control |
| Тод | quality of life |
| ROT | record of training |
| RR | respiratory rate or relative rate |



| Abbreviation | Definition |
|------------------------------|------------------------------------------|
| RSM | regional site monitor |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| $\mathrm{SAS}^{\circledast}$ | a software system used for data analysis |
| SBP | systolic blood pressure |
| SC | study coordinator |
| SCR | software change request |
| SD | standard deviation |
| SDS | study design specifications |
| SDTM | study data tabulation model |
| SDV | source data verification |
| SECC | self-evident correction conventions |
| SECP | self-evident correction plan |
| SF | screen failure |



| Abbreviation | Definition |
|--------------|--------------------------------------------------------|
| SFT or SFTP | secure file transfer or secure file transfer plan |
| SIV | site initiation visit |
| SLA | service level agreement |
| SMP | safety management plan |
| SOC | system organ class |
| SOP | standard operating procedure |
| MOS | statement of work |
| SQV | site qualification visit |
| SUA | start-up associate |
| SUSAR | suspected, unexpected, serious adverse (drug) reaction |
| TA | trial assistant |
| TEAE | treatment-emergent adverse event |
| TMF | trial master file |
| TOM | task ownership matrix |



| Abbreviation | Definition |
|--------------|-------------------------------------------|
| UAT | user acceptance testing |
| USA | United States of America |
| UTC | universal coordinated time |
| WAN | wide area network |
| WAR | work at risk |
| WG | working guideline |
| WHO | world health organization |
| WHO-DD | world health organization drug dictionary |
| WI-NRS | worst itch – numeric rating scale |